## Statistical Analysis Plan



| Sponsor | Mayne Pharma |
|---|---|
| Protocol Title: | A Phase 2 Randomized, Multicenter, Double-blind, |
| | Vehicle-controlled, 90-Day, Safety, Efficacy, and |
| | Systemic Exposure Study followed by a 90-Day |
| | Open-label Extension of Trifarotene (CD5789) Cream HE1 |
| | in Adults and Adolescents with Autosomal Recessive |
| | Ichthyosis with Lamellar Scale |
| Protocol Number: | 18-ICH-001 |
| Premier Research PCN: | MAYN7317 |
| Document Version: | Final 2.0 |
| Document Date: | 09-Nov-2021 |

## Approvals

| Role | Signatures | Date (dd-Mmm-yyyy) |
|---|---|---|
| | Print Name: Valerie Smith | |
| | Sign Name: | |
| Biostatistician | | |
| | Print Name: Phoevos Hughes | |
| | Sign Name: | |
| Mayne Pharma<br>Representative | | |
| Representative | | |





## **Document History**

## **Reasons for Version Final 2.0**

The protocol was amended to version 3.0, and this SAP reflects changes in the protocol.

Text was added to inform of the study being terminated by Mayne Pharma.

#### **Summary of Non-Administrative Changes**

- Globally, all references to "Week X" were changed to "Day XX"; e.g., "Week 12" was changed to "Day 90".
- Figures 1 and 2 (Double-blind and Open-label study designs, respectively) were updated according to protocol changes.
- The Schedule of Events was updated, including the addition of coagulation laboratory panel.
- The lower limit for Analysis Visit 1 was updated to be -97.
- Table 8 (Ectropion Scoring) was updated to add a maximum score.
- The derivation of treatment emergent adverse event was updated to match the protocol, with the upper limit of the start of the event being at most 14 days after last application of study drug.





## **Table of Contents**

| Ap | provals | 5 | 1 |
|-----|-----------|--------------------------------------------------|----|
| Do | cument | t History | 2 |
| Ta | ble of C | Contents | 3 |
| Lis | st of Tal | bles | 5 |
| Lis | st of Fig | gures | 5 |
| 1. | Ov | verview | 6 |
| 2. | Stı | ady Objectives and Endpoints | 6 |
| | 2.1. | Study Objectives | 6 |
| | 2.1.1. | Primary Objective | |
| | 2.1.2. | Secondary Objectives | 6 |
| | 2.2. | Study Endpoints | |
| | 2.2.1. | Safety Endpoints | 7 |
| | 2.2.2. | Efficacy Endpoints | 7 |
| | | Pharmacokinetic Variables | |
| 3. | Ov | verall Study Design and Plan | |
| | 3.1. | Overall Design | 8 |
| | 3.2. | Sample Size and Power | |
| | 3.3. | Study Population | |
| | 3.4. | Treatments Administered | |
| | 3.5. | Method of Assigning Subjects to Treatment Groups | |
| | 3.6. | Blinding and Unblinding | |
| | 3.7. | Schedule of Events | |
| 4. | Sta | atistical Analysis and Reporting | |
| | 4.1. | Introduction | |
| | 4.2. | Interim Analysis and Data Monitoring | |
| 5. | | nalysis Populations | |
| 6. | | eneral Issues for Statistical Analysis | |
| | 6.1. | Statistical Definitions and Algorithms | |
| | 6.1.1. | Baseline | |
| | 6.1.2. | Adjustments for Covariates | |
| | 6.1.3. | Multiple Comparisons | |
| | 6.1.4. | Handling of Dropouts or Missing Data | |
| | 6.1.5. | Analysis Visit Windows | |
| | 6.1.6. | Pooling of Sites | |
| | | Derived Variables | |
| | 6.1.8. | Data Adjustments/Handling/Conventions | 22 |





| 7. | Stı | Idy Subjects and Demographics | 24 |
|---|---|---|---|
| | 7.1. | Disposition of Subjects and Withdrawals | 24 |
| | 7.2. | Protocol Violations and Deviations | 24 |
| | 7.3. | Demographics and Other Baseline Characteristics | 24 |
| | 7.4. | Exposure and Compliance | 25 |
| 8. | Ef | ficacy Analysis | 25 |
| | 8.1. | Primary Efficacy Analysis | 25 |
| | 8.1.1. | Investigator's Global Assessment (IGA) | 25 |
| | 8.1.2. | Multiple Imputation | 27 |
| | 8.2. | Secondary Efficacy Analyses | 28 |
| | 8.2.1. | Visual Index for Ichthyosis Severity (VIIS) | 28 |
| | 8.2.2. | Individual Score for Roughness | |
| | 8.2.3. | Palm/Sole Assessment | 31 |
| | 8.2.4. | Quality of life per Dermatology Life Quality Index (DLQI) and Children's DLQI (cDLQI) | 32 |
| | 8.2.5. | Fissures | 33 |
| | 8.3. | Exploratory Efficacy Analyses | 33 |
| | 8.3.1. | Ectropion | 33 |
| | 8.3.2. | Quality of Life per EQ-5D-5L and EQ-5D-Y | 34 |
| 9. | Sa | fety and Tolerability Analysis | 34 |
| | 9.1. | Adverse Events | 35 |
| | 9.1.1. | Adverse Events Leading to Withdrawal | 35 |
| | 9.1.2. | Deaths and Serious Adverse Events | 36 |
| | 9.2. | Clinical Laboratory Evaluations | 36 |
| | 9.3. | Vital Signs | 36 |
| | 9.4. | Electrocardiograms | 36 |
| | 9.5. | Local Tolerability | 37 |
| | 9.6. | Physical Examination. | 37 |
| | 9.7. | Concomitant Medication | 37 |
| | 9.8. | COVID-19 Visit Impact | 37 |
| 10 | Ch | anges from Planned Analysis | 37 |
| 11. | Ot | her Planned Analysis | 38 |
| | 11.1. | Pharmacokinetic Analysis | 38 |
| | 11.2. | Photography | 39 |
| 12 | Re | ferences | 39 |
| 13 | Ta | bles, Listings, and Figures | 39 |
| | 13.1. | Planned Table Descriptions | 40 |
| | 13.2. | Efficacy Data | <b>4</b> ] |





| 13.3. | Safety Data | 44 |
|-------------|-------------------------------------------------------|-----|
| 13.4. | Pharmacokinetic Data | 47 |
| 13.5. | Planned Listing Descriptions | 47 |
| 13.6. | Planned Figure Descriptions | |
| 14. Ta | bles, Listings, and Listing Shells | 50 |
| 14.1. | Standard Layout for all Tables, Listings, and Figures | |
| 14.2. | Planned Table Shells | |
| 14.3. | Planned Listing Shells | |
| | Planned Figure Shells | |
| Appendix | 1: Premier Research Library of Abbreviations | 147 |
| I ist of T | ahlas | |
| List of T | ables | |
| Table 1: S | chedule of Events for Double-blind Period | 12 |
| Table 2: S | chedule of Events for Open-label Extension | 16 |
| Table 3: A | nalysis Visit Windows | 21 |
| Table 4: IO | GA Scoring Definitions | 25 |
| Table 5: V | IIS Scoring Definitions | 28 |
| Table 6: R | oughness Scoring Definitions | 30 |
| Table 7: P | alm/Sole Scoring Definitions | 31 |
| Table 8: E | ctropion Scoring | 33 |
| Table 9: D | Demographic Data Summary Tables and Figures | 41 |
| Table 10: | Efficacy Data | 41 |
| Table 11: | Safety Data | 44 |
| Table 12: | Pharmacokinetic Data | 47 |
| Table 13: | Planned Listings | 47 |
| Table 14: | Planned Figures | 49 |
| List of F | igures | |
| Figure 1: I | Double-blind Study Design | 9 |
| Figure 2: 0 | Open-label Study Design | 10 |
| | Standardized Layout | |
| | Planned Table Shells | |





#### 1. Overview

This statistical analysis plan (SAP) describes the planned analysis and reporting for Mayne Pharma protocol number 18-ICH-001 (A Phase 2 Randomized, Multi-center, Double-blind, Vehicle-controlled, 90-Day, Safety, Efficacy, and Systemic Exposure Study followed by a 90-Day Open-label Extension of Trifarotene (CD5789) Cream HE1 in Adults and Adolescents with Autosomal Recessive Ichthyosis with Lamellar Scale), version 3.0 dated 26-Oct-2020. Reference materials for this statistical plan include the protocol and the accompanying sample data collection documents. Operational aspects related to collection and timing of planned clinical assessments are not repeated in this SAP unless relevant to the planned analysis.

The structure and content of this SAP provides sufficient detail to meet the requirements identified by the Food and Drug Administration (FDA), European Medicines Agency (EMA), and International Conference on Harmonization (ICH) of Technical Requirements for Registration of Pharmaceuticals for Human Use: Guidance on Statistical Principles in Clinical Trials. All work planned and reported for this SAP will follow internationally accepted guidelines, published by the American Statistical Association and the Royal Statistical Society, for statistical practice.

The planned analyses identified in this SAP may be included in clinical study reports (CSRs), regulatory submissions, or future manuscripts. Also, post-hoc exploratory analyses not necessarily identified in this SAP may be performed to further examine study data. Any post-hoc or unplanned, exploratory analysis performed will be clearly identified as such in the final CSR.

Upon sponsor discretion, this study was terminated before the study completed enrollment; however, all planned analyses will still occur. Sixty-five (65) subjects were enrolled in the study before termination. The statistical plan described hereafter is an *a priori* plan. It will be submitted to file prior to any unblinded inferential or descriptive analysis of data pertaining to Mayne Pharma's study 18-ICH-001.

## 2. Study Objectives and Endpoints

#### 2.1. Study Objectives

## 2.1.1. Primary Objective

The primary objective is to compare the safety and efficacy of 2 concentrations of trifarotene cream HE1 versus vehicle in adults and adolescents with moderate to severe autosomal recessive ichthyosis with lamellar scale, also known as lamellar ichthyosis (LI) after 90 days of treatment.

## 2.1.2. Secondary Objectives

The secondary objectives are:

- To assess systemic exposure to trifarotene and its major metabolites after topical application of the investigational product (IP) on up to 90% body surface area (BSA) twice weekly.
- To assess safety for up to 180 days of dosing with open-label trifarotene cream HE1  $200 \mu g/g$ .



## 2.2. Study Endpoints

## 2.2.1. Safety Endpoints

The safety endpoints of this study include the following:

- Reported serious adverse events (SAEs), treatment-emergent AEs (TEAEs), and changes in clinical laboratory tests, vital signs, physical examinations, and 12-lead electrocardiograms (ECGs)
- Local tolerability (Scale: 0-3 [none, mild, moderate, severe], determined by the investigator) for each body area (chest/abdomen, back, legs, arms, and face/neck).

## 2.2.2. Efficacy Endpoints

## 2.2.2.1. Primary Efficacy Endpoint

The primary efficacy endpoint of this study is the proportion of subjects in each treatment group who experience successful resolution of LI where "success" is defined as clear/almost clear on treated areas and at least a 2-grade change from Baseline at Day 90/end-of-treatment (EOT) in the Double-blind Period on the 5-point Investigator Global Assessment (IGA) full body scale.

## 2.2.2.2. Secondary Efficacy Endpoints

The secondary efficacy endpoints of this study include the following:

- The difference in mean scores between the active trifarotene cream HE1 and vehicle groups in the following assessment indices from Baseline through Day 90:
  - o 5-point Visual Index for Ichthyosis Severity (VIIS) for scaling (overall 16 points for scaling, i.e., 0-4 points for 4 body areas: chest/abdomen, back, arms, and legs)
  - o Individual score for roughness (Scale: 0–4) overall
  - o Palm/sole Assessment (Scale: 0–4)
  - Quality of life per Dermatology Life Quality Index (DLQI) and children's DLQI (cDLQI)
- The difference in proportion of subjects with presence of fissures on palms/soles (presence/absence, number of fissures, and pain associated with fissures on a 0-3 scale) at Day 90 between the active trifarotene cream HE1 and vehicle groups

#### 2.2.2.3. Exploratory Efficacy Endpoints

The exploratory efficacy endpoints of this study include the following:

- The difference in mean ectropion (Ectropion Severity Score [ESS] of 0–8) scores between the active trifarotene cream HE1 and vehicle groups from Baseline through Day 90
- The difference in quality of life per EQ-5D-5L and EQ-5D-Y score between the active trifarotene cream HE1 and vehicle groups from Baseline through Day 90

#### 2.2.3. Pharmacokinetic Variables

The pharmacokinetic (PK) endpoints of the study include plasma concentrations of CD5789 and its major metabolites.





## 3. Overall Study Design and Plan

## 3.1. Overall Design

This is a 2-cohort, multicenter study in subjects with moderate to severe LI (i.e., 3–4 on a 5-point Investigator's Global Assessment [IGA] where 0 = clear; 1 = almost clear; 2 = mild; 3 = moderate; 4 = severe). Adults (Cohort A) and adults and adolescents (Cohort B) will be randomized in a double-blind fashion to 1 of 2 doses of trifarotene cream HE1 or vehicle and treated twice weekly for 90 days.

Approximately 15 adults ( $\geq$ 18 years old) will be randomized into the first cohort of subjects (Cohort A) in a 1:1:1 ratio to trifarotene cream HE1 100 µg/g, trifarotene cream HE1 200 µg/g, or vehicle and treated twice weekly for up to 90 days. After the initial 15 subjects complete at least 28 days of treatment, an independent data safety monitoring board (DSMB) will review aggregate safety and tolerability data.

If no safety issues are identified, both adults and adolescents (ages 12 to 17 years, inclusive) will be allowed to enroll in Cohort B. Subjects in Cohort B will be randomized 1:1:1 to trifarotene cream HE1 100  $\mu$ g/g, trifarotene cream HE1 200  $\mu$ g/g, or vehicle and treated twice weekly for up to 90 days in the same manner as subjects in Cohort A. All subjects (Cohort A and Cohort B) who complete the randomized, Double-blind Period of the study will be eligible to enter a 90-day, Open-label Extension (OLE) in which additional PK, safety, and efficacy data will be collected. Subjects in the OLE will receive open-label trifarotene cream HE1 200  $\mu$ g/g twice weekly for up to 90 days. A schematic of each period is provided in Figure 1 and Figure 2.



Figure 1: Double-blind Study Design





Figure 2: Open-label Study Design



The first cohort of 15 adult subjects is a reasonable sample size to assess safety and tolerability before enrolling adolescents. Accounting for a 20% drop-out/nonevaluable rate, a total sample size of 120 subjects randomized in a 1:1:1 ratio to 2 active trifarotene cream HE1 arms and a vehicle cream arm will provide >80% power to detect a difference between each separate trifarotene cream HE1 arm (32 evaluable subjects) and the vehicle cream arm (32 evaluable subjects) 2-sided Fisher's Exact Test assuming a 70% success rate and a 40% success rate, respectively. This study is not powered to detect a difference between the 2 active arms.

## 3.3. Study Population

This study includes adults and adolescents with moderate to severe autosomal recessive ichthyosis with lamellar scale.

#### 3.4. Treatments Administered

For the Double-blind Treatment Period, a fixed dose (determined at Visit 2) of trifarotene cream HE1 100  $\mu$ g/g or 200  $\mu$ g/g or vehicle cream will be applied topically twice weekly on up to 90% body surface area (BSA) of each subject. Trifarotene cream HE1 is a cream containing 100 or 200  $\mu$ g/g (0.01% [w/w] or 0.02% [w/w], respectively) of CD5789. Vehicle contains the same ingredients, without the CD5789. Trifarotene cream HE1 and vehicle will be provided in cream form for topical application and will be packaged in 50-g tubes from which up to 36 g of investigational product (IP) may be dispensed per application, i.e., the maximum dose per





application. Study staff will apply the first dose of study drug to each subject in the clinic on Day 1 after baseline measurements, and will record the amount of study drug applied.

Thereafter, each subject will apply approximately the same amount (up to 36 g) of study drug as for the first dose on up to 90% of BSA twice weekly, sparing the scalp, inguinal, and axillary areas. Subjects will receive an adequate number of tubes to use 1 tube per application and will use a new tube for each treatment day.

For the OLE, all subjects will receive trifarotene cream HE1 200  $\mu$ g/g and apply the same fixed dose in the same manner as in the Double-blind Period for an additional 90 days.

If the treatment causes application site reactions, the frequency of application will be reduced or interrupted only on the area of concern, as indicated herein. During all clinic visits, the investigator will assess local tolerability (Scale: 0-3 [none, mild, moderate, severe]) for stinging/burning, pruritus, erythema) for each body area (chest/abdomen, back, arms, legs, and face/neck), and the following procedures will be followed:

- If a score of 2 (moderate) is recorded on a local tolerability assessment scale (stinging/burning, pruritus, erythema) on any treated area, the study drug will be applied on that area only once weekly, until the score is back to <2. Continue to treat all other areas twice weekly provided the score is <2 on those areas.
- If a score of 3 (severe) is recorded on a local tolerability assessment scale (stinging/burning, pruritus, erythema) on any treated area, the study drug will not be applied on that area until the score is back to <3 (i.e., "drug holiday"). Continue to treat all other areas twice weekly provided the score is <2 on those areas.

## 3.5. Method of Assigning Subjects to Treatment Groups

Subjects will be randomized in a 1:1:1 ratio to trifarotene cream HE1 100  $\mu$ g/g or 200  $\mu$ g/g or vehicle cream in the Double-blind Period.

Subjects who continue into the OLE will receive trifarotene cream HE1 200  $\mu$ g/g and apply the same fixed dose in the same manner as in the Double-blind Period for an additional 90 days.

#### 3.6. Blinding and Unblinding

All subjects, investigators, and study personnel involved in the conduct of the Double-blind Period of the study, including data management, will be blinded to treatment assignment with the exception of a specified unblinded statistician and programmer from Premier Research who will have access to the randomization code.

The primary analysis period is the first 90 days of treatment (i.e., the Double-blind Period). Overall unblinding will take place at the end of the Double-blind Period of the study only after database lock has been achieved. A second analysis will take place for endpoints assessed from Day 90 through the OLE.

#### 3.7. Schedule of Events

A detailed schedule of events for the Double-blind period of the study is provided in Table 1. A detailed schedule of events for the OLE is provided in Table 2.





## **Table 1: Schedule of Events for Double-blind Period**

| | | Double-blind Treatment Period | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | Screening<br>(-97 days to -1 day)<br>Washout up to 90 Days <sup>a</sup> | Baseline<br>(Day 1) | Telephone<br>Visit<br>(Day 7) | Day 14<br>± 5 days | Day 30<br>± 7 days | Telephone<br>Visit<br>(Day 45) | Day 60<br>± 7 days | Day 90 <sup>b,c</sup><br>± 7 days<br>(ET) |
| Visit | 1 | 2 | | 3 <sup>d</sup> | <b>4</b> <sup>d</sup> | | 5 <sup>d</sup> | 6 <sup>d</sup> |
| Written informed consent/assent | X | | | | | | | X <sup>a</sup> |
| Assign screening number | X | | | | | | | |
| Inclusion/exclusion criteria | X | X | | | | | | |
| Demographics | X | | | | | | | |
| Medical history | X | | | | | | | |
| Physical examination | X | X e | | | | | | X e |
| Vital signs (blood pressure and pulse) | X | X | | X | X | | X | X |
| Height, weight, and BMI | X | | | | | | | Xb |
| IGA assessment <sup>f</sup> | X | X | | X | X | | X | X |
| VIISg assessment | X | X | | X | X | | X | X |
| Roughness assessmenth | X | X | | X | X | | X | X |
| Palm/sole assessment | X | X | | X | X | | X | X |
| Palm/sole fissuring assessmenti | X | X | | X | X | | X | X |
| Ectropion score | X | X | | X | X | | X | X |
| Photographs <sup>j</sup> | | X | | | X | | | X |
| Quality of life per Dermatology Life<br>Quality Index (DLQI) | | X | | X | X | | X | X |
| EQ-5D Quality of Life Questionnaire | | X | | X | X | | X | X |
| 12-lead ECG <sup>k</sup> | X | X | | | X | | | X |



| | | | | Double- | blind Treat | ment Period | | |
|---|---|---|---|---|---|---|---|---|
| | Screening<br>(-97 days to -1 day)<br>Washout up to 90 Days <sup>a</sup> | Baseline<br>(Day 1) | Telephone<br>Visit<br>(Day 7) | Day 14<br>± 5 days | Day 30 ± 7 days | Telephone<br>Visit<br>(Day 45) | Day 60 ± 7 days | Day 90 <sup>b,c</sup><br>± 7 days<br>(ET) |
| Visit | 1 | 2 | | 3 <sup>d</sup> | <b>4</b> <sup>d</sup> | | 5 <sup>d</sup> | 6 <sup>d</sup> |
| Clinical laboratory tests (hematology, chemistry, urinalysis) <sup>l</sup> | X | X | | | X | | | X |
| Serology (hepatitis B surface antigen, hepatitis C) | X | | | | | | | |
| Coagulation panel | | X | | | X | | | X |
| Pregnancy test for female subjects (serum at Screening; urine subsequently) <sup>m</sup> | X | X | | | X | | X | X |
| Randomization via IWRS | | X | | | | | | |
| PK blood sample collection <sup>n</sup> | | X | | X | X | | X | X |
| Initial study drug application by clinic staff and measurement <sup>o</sup> | | X | | | | | | |
| Application instructions, advice on emollient and sunscreen use | | X | X | X | X | X | X | X |
| Dispense study drug and diaries <sup>p</sup> | | X | | Xp | Xp | | Xp | $(X)^p$ |
| Concomitant medications | X | X | X | X | X | X | X | X |
| Tolerability assessment | | X | | X | X | | X | X |
| Adverse events (and review diaries) | | X | X | X | X | X | X | X |
| Collect all used/unused study drug <sup>q</sup> | | | | X | X | | X | X |
| Provide information about OLE option | | | | | X | X | X | X |

Abbreviations: BMI = body mass index; DLQI = Dermatology Life Quality Index; ECG = electrocardiogram; ET = early termination; HEENT = head, eyes, ears, nose, throat; ICF = informed consent form; IGA = Investigator's Global Assessment; IWRS = interactive web response system; OLE = open-label extension; PK = pharmacokinetic; WOCBP = women of childbearing potential; VIIS = Visual Index for Ichthyosis Severity





- a. Upon signing informed consent and entering the Screening Period, subjects will stop using physical and medical treatments for LI, including balneotherapy, and begin to washout prohibited topical and systemic treatments with designated washout periods, as applicable. Before asking a subject to enter washout, investigators should confirm the subject meets study eligibility criteria, except for LI severity (Inclusion Criterion #3). Washout may be up to 90 days. After completing any necessary Washout Period, subjects must return to the site within 35 days before the Baseline Visit within the 97-day Screening Period to have their LI severity assessed and study eligibility requirements determined. During washout, subjects may continue their standard ofcare of visible skin (face and scalp) for cosmetic reasons and of extremities (palms/soles) to avoid functional consequences on walking or moving their fingers. In the US/EU, this may include compounded emollients with keratolytics (alpha or beta hydroxyl acids) and/or urea. The investigator should approve and document these standard of care treatments in the electronic case report form (eCRF). If the standard of care treatments of the face and/or palms/soles contain prohibited medications, they must be stopped at the Baseline Visit. Subjects may shower, but not bathe or swim, during the Screening Period.
- b. Day 90 procedures should be conducted for subjects who terminate the study early. If a subject discontinues IP, but continues to attend clinic visits, Day 90 will occur as scheduled. Day 90 will be the first visit of the OLE for subjects who choose to continue. Subjects who decide to continue into the OLE will have the following additional procedures: 1) sign informed consent; 2) will be weighed; 3) will be instructed on study drug application; 4) will be given new diaries, and 5) will be provided with study drug.
- c. A Follow-up telephone call will be made within 14 days after Day 90 to subjects who choose not to continue into the OLE to assess any ongoing adverse events.
- d. Although it is preferable to conduct all necessary study assessments in person (onsite visits), this may not be possible as a result of COVID-19-related travel restrictions. To ensure the safety of subjects, investigators, and site staff, Visits 3-6 and unscheduled visits may be conducted remotely. Screening and baseline visits must be performed onsite only, and must be postponed or scheduled for when onsite visits can be safely conducted.
- e. Limited physical examination to include HEENT, cardiorespiratory, abdomen, range of motion.
- f. IGA: 0 = clear; 1 = almost clear; 2 = mild; 3 = moderate; 4 = severe.
- g. VIIS scale for each body area: chest/abdomen, back, legs, and arms, for a possible overall score = 16.
- h. Roughness (0-4 scale);
- i. Palm/sole fissuring assessment: present/absent/number/pain (0-3 scale).
- j. Photography will be performed at sites with the capability for subjects who sign a photographic ICF. A central reader who will not be an investigator in the study will review the photographs to assess consistency of investigator scoring of LI severity as a quality check.
- k. ECG to be conducted at Screening, Baseline, Day 30, and Day 90 for all subjects. Subjects in the PK substudy will also have postdose ECGs at each serial blood draw on Day 1 and Day 30.
- 1. Subjects must be fasting (i.e., at least 8 hours) for clinical laboratory tests, but not for PK blood draws.
- m. Note: Subjects who are premenstrual at Screening but begin menses during the course of the study should follow the pregnancy testing schedule for WOCBP correlating to the visit menses began.
- n. Samples for PK will be drawn from all subjects at Baseline and at each clinic visit. At selected sites among subjects who consent to participate in the PK substudy, samples will be taken predose and at 1, 2, 4, 8, 12, and 24 hours postdose on Day 1. On Day 30, IP will be applied in the clinic for PK substudy subjects, and PK samples will be taken predose and at 1, 2, 4, 8, 12, and 24 hours postdose. Trough levels will be drawn when the subjects are in the clinic for other study visits (i.e., Day 14, Day 60, and Day 90). Visits for PK must occur at least 24 hours after the last application of the IP to avoid contamination of the blood samples with any IP that may have remained in the skin after the last application.
- o. Study staff will apply initial dose of study drug in the clinic after Baseline measurements, and the amount of study drug used will be measured (i.e., 36-g tube will be measured before and after application to determine amount used).
- p. Study drug provided in 50-g tubes (maximum single application is 36 g). Measure study drug kits (tubes and box, but not leaflets) before dispensing; subjects must record days/times of study drug application in the diaries and any areas of skin not treated, e.g., due to local reactions. Dispense enough additional study drug until next visit (except at Day 90, unless subject consents to continue into OLE).

AD-ST-33.05 Effective date: 22-Jan-2018





q. Confirm study drug compliance by weighing the studykits (tubes and boxes, but not leaflets) and reviewing diary.

AD-ST-33.05 Effective date: 22-Jan-2018





**Table 2: Schedule of Events for Open-label Extension** 

| | | 0 | pen-label Tr | Follow-up | | | |
|---|---|---|---|---|---|---|---|
| | Telephone<br>Visit<br>(Day 97) <sup>a</sup> | Day 104<br>± 5 days | Day 120<br>± 7 days | Telephone<br>Visit<br>(Day 134) | Day 150<br>± 7 days | Day 180<br>± 7<br>days/ET | Day 194 or 14 days after End of<br>Open-label Treatment |
| Visit | | 7ª | 8 <sup>a</sup> | | 9ª | 10 <sup>a</sup> | 11 <sup>a</sup> |
| Informed consent <sup>b</sup> | | | | | | | |
| Physical examination <sup>c</sup> | | | | | | X | X |
| Vital signs (blood pressure and pulse) | | | X | X | X | X | X |
| Record IGA <sup>d</sup> | | X | X | | X | X | X |
| VIIS <sup>e</sup> assessment | | X | X | | X | X | X |
| Roughness assessment <sup>f</sup> | | X | X | | X | X | X |
| Palm/sole assessment | | X | X | | X | X | X |
| Palm/sole fissuring assessment | | X | X | | X | X | X |
| Ectropion score | | X | X | | X | X | X |
| Clinical laboratory tests<br>(hematology, chemistry,<br>urinalysis) <sup>g</sup> | | | X | | | X | |
| Pregnancy test for female subjects (urine) <sup>h</sup> | | | X | | X | X | X |
| Coagulation panel | | | X | | | X | |
| 12-lead ECG | | | X | | | X | |
| PK blood sample collection <sup>i</sup> | | | X | | | X | |
| Application instructions, advice on emollient and sunscreen use <sup>j</sup> | X | X | X | X | | | |
| Dispense study drug and diaries <sup>k</sup> | | X | X | | X | | |
| Concomitant medications | X | X | X | X | X | X | X |



| | | 0 | pen-label Tr | eatment Perio | od <sup>a</sup> | | Follow-up |
|---|---|---|---|---|---|---|---|
| | Telephone<br>Visit<br>(Day 97) <sup>a</sup> | Day 104<br>± 5 days | Day 120<br>± 7 days | Telephone<br>Visit<br>(Day 134) | Day 150<br>± 7 days | Day 180<br>± 7<br>days/ET | Day 194 or 14 days after End of<br>Open-label Treatment |
| Visit | | 7ª | <b>8</b> <sup>a</sup> | | 9a | 10 <sup>a</sup> | 11ª |
| Tolerability assessment | | X | X | | X | X | |
| Adverse events (and review diaries) | X | X | X | X | X | X | X |
| Collect all used/unused study drug <sup>1</sup> | | X | X | | X | X | |

Abbreviations: ECG = electrocardiogram; ET = early termination; HEENT = head, eyes, ears, nose, throat; ICF = informed consent form; IGA = Investigator's Global Assessment; PK = pharmacokinetic; OLE = open-label extension; VIIS = Visual Index for Ichthyosis Severity; WOCBP = women of childbearing potential

- a. Although it is preferable to conduct all necessary study assessments in person (on -site visits), this may not be possible as a result of COVID-19-related travel restrictions. To ensure the safety of subjects, investigators, and site staff, Visits 7-11 and unscheduled visits may be conducted remotely.
- b. Subjects will sign the OLE ICF at the Double-blind Day 90 Visit. All efficacy assessments, safety/tolerability assessments, including clinical laboratory testing and PK from Day 90 will be carried over for the OLE and will not be repeated.
- c. Limited physical examination to include HEENT, cardiorespiratory, abdomen, range of motion.
- d. IGA: 0 = clear; 1 = almost clear; 2 = mild; 3 = moderate; 4 = severe
- e. VIIS scale for each body area: chest/abdomen, back, legs, and arms, for a possible overall score = 16.
- f. Roughness (0-4 scale); fissuring assessment on palms/soles: present/absent/number/pain (0-3 scale).
- g. Subjects must be fasting (at least 8 hours) for clinical chemistry testing, but not for PK only blood draws.
- h. Subjects who are premenstrual at Screening but begin menses during the course of the study should follow the pregnancy testing schedule for WOCBP correlating to the visit menses began.
- i. Samples for PK will be drawn from all subjects at Day 120 and Day 180. Visits for PK must occur at least 24 hours after the last application of the IP to avoid contamination of the blood samples with any IP that may have remained in the skin after the last application.
- j. Subjects must record days/times of study drug application in the diaries and any areas of skin not treated (e.g., due to local reactions).
- k. All subjects in the OLE will receive trifarotene 200 μg/g. Study drug provided in 50-g tubes (maximum single application is 36 g). Measure study drug tubes before dispensing. Dispense enough additional study drug until the next visit (except at Day 180).
- 1. Confirm study drug compliance by weighing the study kits (tubes and boxes, but not leaflets) dispensed and returned and reviewing diary.





## 4. Statistical Analysis and Reporting

#### 4.1. Introduction

Data processing, tabulation of descriptive statistics, calculation of inferential statistics, and graphical representations will be performed primarily using SAS (release 9.4 or higher). If the use of other software is warranted, the final statistical methodology report will detail what software was used for what purposes.

Continuous (quantitative) variable summaries will include the number of subjects (n) with nonmissing values, mean, standard deviation (SD), standard error (SE), median, minimum, and maximum.

Categorical (qualitative) variable summaries will include the frequency and percentage of subjects who are in the particular category or each possible value. In general, the denominator for the percentage calculation will be based upon the total number of subjects in the study population for the treatment groups, unless otherwise specified. The denominator for by-visit displays will be the number of subjects in the relevant study population with nonmissing data at each study visit.

The minimum and maximum will be reported with the same degree of precision (i.e., the same number of decimal places) as the observed data. Measures of location (mean and median) will be reported to 1 degree of precision more than the observed data and measures of spread (SD, SE) will be reported to 2 degrees of precision more than the observed data.

Percentages will be presented to 1 decimal place, unless otherwise specified and with the following exceptions: a percentage of 0% will not be displayed (i.e., only the count of 0 will be displayed), and a percentage of 100% will be displayed with 0 decimal places.

Unless otherwise indicated, all statistical tests will be conducted at the 0.05 significance level using 2-tailed tests, and P values will be reported. Corresponding 95% confidence intervals (CIs) will be presented for statistical tests. A P value of  $\leq$ 0.10 but >0.05 will be considered evidence of a trend.

## 4.2. Interim Analysis and Data Monitoring

The DSMB will meet after 15 subjects in Cohort A have completed at least 28 days of double-blind treatment to review aggregate safety and tolerability data (including PK concentration data, PK parameters, and ECG results). The safety data will be unblinded. At that time, the DSMB will decide whether Cohort B (adults and subjects aged 12–17) may begin enrolling, or if additional adult safety data are required before allowing subjects aged 12 – 17 to participate in the study. The DSMB will meet again after 60 subjects have enrolled in the study. The sponsor may request additional reviews, e.g., should any other findings/issues pertaining to safety emerge requiring DSMB review. Details of the DSMB operation will be developed in conjunction with the members of the DSMB before the first meeting and will be modified as required. The unblinded DSMB outputs will not be seen by anyone except the DSMB and the performing statistician.





The primary analysis period is the first 90 days of treatment (i.e., the Double-blind Period). Overall unblinding will take place at the end of the Double-blind Period of the study only after database lock has been achieved. The data will be cleaned and frozen and an unblinded analysis of the data will be performed. The data will be considered final at this point and no changes to these data will be permitted following unblinding with the exception of outcomes and end dates of ongoing AEs and concomitant mediations. A second analysis will take place for endpoints assessed from Day 90 through the OLE.

The protocol assumes a 20% dropout/non-evaluable rate. This rate will be continuously monitored throughout the COVID-19 pandemic. In the event that this rate dramatically increases, a blinded sample size reestimation may be performed to ensure statistical power for the primary endpoint is maintained using the assumptions in Section 3.2.

## 5. Analysis Populations

The following 5 analysis populations are planned for the Double-blind Period of this study:

- Safety: all subjects who are randomized to treatment and receive at least 1 application of study drug in the Double-blind Period. This population will be the primary population for analyses of safety. Subjects will be analyzed by actual treatment received.
- Intent-to-treat (ITT): all randomized subjects. This population will be used as the primary population for the analysis of efficacy for the Double-blind Period of the study. Subjects will be analyzed by randomized treatment.
- Modified intent-to-treat (mITT): all subjects in the Safety population with at least 1 postbaseline assessment of efficacy in the Double-blind Period. Subjects will be analyzed by randomized treatment.
- **Per-protocol (PP)**: subjects in the mITT population who met all inclusion criteria and no exclusion criteria, were compliant with study drug application, and who had no significant protocol deviations. Subjects will be analyzed by actual treatment received.
- **Pharmacokinetic (PK)**: all subjects in the Safety population who have at least 1 plasma sample with quantifiable concentration. This population will be used to summarize all PK endpoints. Subjects will be analyzed by actual treatment received.

The following analysis populations are planned for the OLE of this study:

- **OLE Safety:** all subjects who complete the 90-day Double-blind Treatment Period and receive at least 1 application of study drug in the OLE.
- **OLE ITT:** all subjects who complete the 90-day Double-blind Treatment Period and sign the OLE informed consent.
- **OLE mITT:** all subjects in the OLE Safety population with at least 1 assessment of efficacy after Visit 6.
- OLE PP: all subjects in the OLE mITT population who met all inclusion criteria and no exclusion criteria, were compliant with study drug application from baseline through EOT, and who had no significant protocol deviations throughout the study.

Since all subjects in the OLE are to receive trifarotene cream HE1 200  $\mu$ g/g, analyses will be by actual treatment received.





Inclusion in the analysis populations will be determined prior to database lock. Deviations related to COVID-19 will also be evaluated in determining PP population eligibility.

## 6. General Issues for Statistical Analysis

## 6.1. Statistical Definitions and Algorithms

#### 6.1.1. Baseline

The last nonmissing assessment recorded prior to the first dose of treatment in the Double-blind Period will be used as the baseline observation for all calculations of change from baseline, including those in the OLE.

## **6.1.2.** Adjustments for Covariates

If there is a statistical difference among treatment groups with respect to baseline characteristics, that variable may be added to the statistical models as a blocking factor or covariate to determine the effect on treatment. Age group and baseline score are planned for inclusion in statistical models, unless otherwise indicated. Age group will be categorized as adolescents (ages 12 to 17 years, inclusive) and adults ( $\geq$ 18 years).

## **6.1.3.** Multiple Comparisons

No adjustments will be made for multiple comparisons. All *P* values for the secondary and exploratory endpoints will be provided in the summary tables for informational purposes only.

## 6.1.4. Handling of Dropouts or Missing Data

All possible efforts will be made to ensure that subjects stay in the study and all data are collected as scheduled. Withdrawn subjects will not be replaced. If a substantial number of subjects are withdrawn from the study, the sponsor will evaluate the need for developing replacement criteria. Randomized subjects withdrawn from the study may not reenter.

Missing endpoint values in this study may result from subjects discontinuing from the study prematurely or missing intermediate assessments while remaining on study. To assess the effect of missing data on the primary efficacy analysis, a sensitivity analysis will be performed using multiple imputation (MI) for the Double-blind Period only. Multiple imputations will be used to replace missing IGA outcomes using multiple draws from the posterior predictive distribution estimated from the vehicle treatment. The IGA scores will be imputed and then categorized as treatment success.

Sensitivity analyses to investigate robustness to missing data will be performed for the primary endpoint as described in Section 8.1.2.

Missing safety data and data for secondary endpoints will not be imputed.





## **6.1.5.** Analysis Visit Windows

Visits will be analyzed as scheduled. Unscheduled and/or repeated measurements will only be included if a scheduled measurement is not available and the unscheduled/repeated measurement falls within the analysis visit windows as described in Table 3. The windows follow the Schedule of Events in Table 1 and Table 2. Unscheduled/repeated measurements will be listed.

**Table 3: Analysis Visit Windows** 

| Visit | Target Start Day | Lower Limit | Upper Limit |
|-------|------------------|-------------|-------------|
| 1 | | -97 | -1 |
| 2 | 1 | 1 | 1 |
| 3 | 14 | 9 | 19 |
| 4 | 30 | 23 | 37 |
| 5 | 60 | 53 | 67 |
| 6 | 90 | 83 | 97 |
| 7 | 104 | 99 | 109 |
| 8 | 120 | 113 | 127 |
| 9 | 150 | 143 | 157 |
| 10 | 180 | 173 | 187 |
| 11 | 194 | 194 | 194 |

Visit windows may be extended (as reasonable) so as to accommodate delays for assessments due to the COVID-19 pandemic.

## 6.1.6. Pooling of Sites

Not applicable. Site will be omitted from statistical models as the anticipated number of subjects per site is small, treatment is self-administered, and the sites are using standardized procedures for all assessments. If the distribution of enrollments at sites is such that one or few are enrolling a majority of subjects, an ad hoc analysis by site may be performed.

#### 6.1.7. Derived Variables

- IGA average score = in protocol version 1.0, IGA was assessed by body area (chest/abdomen, back, arms, and legs). Under protocol version 2.0, this was changed to a global (overall) assessment. For comparability, the average of the body area IGA results will be taken to yield one score for subjects enrolled under protocol version 1.0. Scores will range from 0 to 4. Higher scores indicate worse disease.
- VIIS total score = sum of the individual body area scaling scores, with a range of 0 to 16. Each individual item is scored on a scale of 0-4, where 0 = normal skin; no perceptible scale or smoothening and 4 = confluent, primarily large, thick scales. Higher scores indicate worse scaling.
- Ectropion total score = sum of the 8 individual item scores (lateral apposition, medial apposition, scleral show, conjunctival show, excess tear film, redness of the eye, round canthus, punctum lacrimale), with a range of 0 to 8. Each individual item is scored 0



(nonaffected/no/invisible), 0.5 (≤1 mm/emerging), or 1 (affected/yes/visible). Higher scores indicates worse ectropion.

- DLQI total score = sum of the 10 individual item scores, with a range of 0 to 30. Higher scores indicate poorer quality of life.
- CDLQI total score = sum of the 10 individual item scores, with a range of 0 to 30. Higher scores indicate poorer quality of life.
- Number of doses taken = total number of tubes returned total number of tubes returned unused
- Number of weeks on study = (last day on study treatment start date + 1) / 7
- Number of expected doses = 2 \* number of weeks on study
- Total weight used = total weight of tubes dispensed (grams) total weight of tubes returned (grams)
- Initial application amount used = tube weight before drug application (grams) tube weight after drug application (grams), as collected on the initial study drug application CRF
- Compliance by tube weight = total weight used / total weight of tubes dispensed \*100%
- Compliance by number of doses = number of doses taken / number of expected doses \* 100%
- Change from baseline = value at current time point value at baseline.
- TEAE = An AE is defined as treatment emergent if the onset or worsening is at the time of or following the start of the first application of study drug (trifarotene or vehicle) through the Follow-up Visit or Early Termination Visit, whichever occurs first..

#### 6.1.8. Data Adjustments/Handling/Conventions

All collected data will be presented in listings. Data not subject to analysis according to this plan will not appear in any tables or graphs but will be included only in the data listings.

All P values will be displayed in 4 decimals and rounded using standard scientific notation (e.g., 0.XXXX). If a P value less than 0.0001 occurs it will be shown in tables as <0.0001.

Adverse events will be coded using the MedDRA version 21.1 thesaurus. Concomitant mediations will be coded using the WHO-DD version September 2018.

A treatment-related AE is any AE with a relationship to the study drug of possibly related and related.





If partial AE or medication dates occur, the convention for replacing missing dates for the purpose of statistical analysis is as follows:

## For partial AE and medication start dates:

- If the year is unknown, then do not impute the date but assign a missing value.
- If the year is known, but the month or month and day is unknown, then:
  - o If the year matches the year of first dose date and the end date (if present) is after first dose date, then impute as the month and day of the first dose date.
  - o Otherwise, assign 01 January.
- If the year and month are known, but the day is unknown, then:
  - o If the month and year match the month and year of the first dose date, then impute as the day of the first dose date.
  - o Otherwise, assign 01.

## For partial AE and medication end dates:

- If the year is unknown, then do not impute the date but assign as missing value.
- If the year is known, but the month or month and day is unknown, then:
  - o If the year matches the year of the last date of the study (date of last contact if subject lost to follow-up; date of completion or early termination otherwise), then impute as the month and day of the last date of the study.
  - o Otherwise, assign 31 December.
- If the year and month are known, but the day is unknown, then:
  - o If the month and year match the month and year of the last date of the study, then impute as the day of the last date of the study.
  - Otherwise, assign the last day of the month.

## If partial times occur, the convention is as follows:

- if the missing time occurs on the day of the first dose and both the hour and minute are missing then the time assigned is the time of the first dose, otherwise if both the hour and minute are missing and the date is not the date of first dose the time assigned is 12:00;
- if the date is the same as the date of the first dose and



- o only hour is missing the hour assigned is 12 or the hour of first dose, whichever is later;
- o only the minute is missing the minute assigned is 30 or the minute of first dose, whichever is later;
- Otherwise if the date is not the same as the date of first dose, the hour assigned is 12 if the hour is missing and the minute assigned is 30 if the minute is missing.

## 7. Study Subjects and Demographics

## 7.1. Disposition of Subjects and Withdrawals

Disposition will include tabulations of the number of subjects randomized into each treatment group, the number of subjects completing Day 90 of the study, the number of subjects withdrawing early from the Double-blind Period, tabulated reasons for withdrawal from the Double-blind Period, and number of subjects in each analysis population. This analysis will be conducted on the ITT population.

Additionally, the number of subjects entering the OLE, completing the study through OLE follow up (Day 194), withdrawing early from the OLE, and tabulated reasons for withdrawal from the OLE will be presented for the OLE ITT population.

If a subject discontinues due to COVID-19, those reasons will also be presented.

#### 7.2. Protocol Violations and Deviations

Major protocol violations, including those due to the impact of COVID-19, as determined by a Sponsor blinded review of the data prior to database lock and unblinding of the study, may result in the removal of a subject's data from the PP population.

All protocol violations will be presented in a data listing, with a flag to indicate if a violation was considered major and resulted in the exclusion of the subject from the PP population.

#### 7.3. Demographics and Other Baseline Characteristics

Summary statistics for age, gender, race, ethnicity, height, weight, BMI, and baseline IGA score will be presented by treatment group. See Section 6.1.1 for definition of baseline.

These analyses will be conducted for the ITT and OLE ITT populations.

The number and percent of subjects reporting various medical histories, grouped by MedDRA system organ class (SOC) and preferred term (PT), will be tabulated by treatment group. This analysis will be conducted for the Safety population.

Prior medications will be summarized by treatment group, by the number and percentage of subjects taking each medication, classified using WHO-DDE ATC Class Level 4 and preferred term (ATC Class Level 5) and will be presented by treatment group and overall. This analysis will be conducted for the Safety population. Prior medications are defined in Section 9.7.





## 7.4. Exposure and Compliance

Compliance by tube weight and compliance by number of doses will be summarized by treatment group using descriptive statistics. The total weight of tubes dispensed and returned, as well as total number of tubes dispensed, returned, and returned unused will also be summarized. This analysis will be conducted for the Safety population and for the OLE Safety population.

A subject is compliant with study product if he or she takes at least 80%-120% of the scheduled doses as assessed by number of doses taken reported, supplemented by tube weight and diary entries. The number and percentage of subjects who were compliant will be tabulated by treatment group for the Double-blind Period and overall for the OLE. Derivations of compliance are defined in Section 6.1.7.

All initial study drug application, drug accountability (dispensed and returned), and subject diary data collected will be listed. Changes in treatment administration or treatment dispensation due to COVID-19 including start and end dates of change, method of alternative administration/dispensation, dosing interruptions, and relevant changes to compliance expectations (weights or tube counts) will be documented from the COVID-19 visit impact log.

## 8. Efficacy Analysis

All efficacy endpoints will be summarized using the ITT population. The primary analysis will be repeated in the mITT and PP populations.

Summaries of efficacy variables in the OLE will be provided using the OLE ITT. Primary IGA summaries will also be provided for the OLE mITT and OLE PP populations. For continuous efficacy analyses using MMRM, only formal comparisons of change from baseline will be performed in the OLE. No other formal inferential analyses will be conducted for efficacy variables in the OLE.

All efficacy data, regardless of population, will be presented in data listings.

If alternative methods are used for capturing efficacy assessments (i.e., in person not on site at the subject's home, remotely with visual aid, or remotely via telephone), additional sensitivity or subgroup analyses may be performed to assess the potential impact to efficacy analyses. These will be delineated as ad hoc analyses in the CSR.

## 8.1. Primary Efficacy Analysis

## 8.1.1. Investigator's Global Assessment (IGA)

The 5-point IGA is a measure of disease severity and meets the need for a clinically meaningful measure of success for ichthyosis studies. Each level of severity will consider both the severity of scaling and the severity of roughness. The investigator will rate the subject's condition using the 5-point scale (0-4), excluding the following areas: knees, elbows, neck, palms, soles, axillae, groin, and scalp, where higher scores represent more severe disease. The IGA is collected at all clinic visits. The scoring is as follows below in Table 4.

#### **Table 4: IGA Scoring Definitions**





| Score | Definition |
|---|---|
| 0 | Clear: No scaling and no roughness |
| 1 | Almost clear: Occasional fine scales; hardly palpable roughness (mostly smooth) |
| 2 | Mild: Small and fine scales predominate; no more than a few large scales; mild roughness on palpation |
| 3 | Moderate: Some large scales that may be thick; coarse roughness on palpation |
| 4 | Severe: Confluent, primarily large (>1cm) thick scales with plate-like hyperkeratosis |

The primary efficacy endpoint is the proportion of subjects in each treatment group who experience successful resolution of LI where "success" is defined as clear/almost clear overall and at least a 2-grade change from Baseline at Day 90/EOT in the Double-blind Period on the 5-point IGA scale. The number and percentage of subjects with treatment success will be summarized by treatment group. The primary efficacy endpoint will be analyzed using a logistic regression model with treatment, baseline IGA score, and age group as factors. The odds ratios and 95% CIs for the odds ratios will be presented. The difference in proportions between the active trifarotene cream HEI groups and vehicle cream group, 95% CIs for the differences, and *P* values for the differences in treatment will also be presented.

The potential for heterogeneity of treatment effects will be assessed by testing treatment-by-factor interactions. The logistic regression model for the primary analyses will be expanded to include the treatment-by-age group interaction. In the event of quasi or complete separation, the logistic regression model will use Firth's penalized maximum likelihood estimation.

The same logistic regression model will be used to analyze the proportion of subjects with at least a 50% reduction in IGA score from baseline as a secondary analysis.

The change from baseline IGA score will be analyzed using a mixed model for repeated measures (MMRM). The MMRM model will include change from baseline in IGA score as the dependent variable, treatment, study visit, treatment-by-visit interaction, and age group as fixed effects, subject as a random effect, and baseline IGA score as a covariate. All post-baseline study visits will be included in the model; however, the primary comparison will be between the active trifarotene cream HE1 groups and vehicle at Day 90. An unstructured covariance matrix will be used to model the within-subject errors. The Kenward-Roger approximation will be used to estimate degrees of freedom. In case of convergence issues, other covariance structures will be explored including autoregressive (AR(1)), compound symmetry (CS), and variance components (VC) with each model fit to find the covariance structure with the best fit. The fit statistics will be compared for all covariance structures; the structure with the smallest Akaike information criterion will be retained as the preferred model and noted in the resulting table. For the OLE period, the model will not include treatment or treatment-by-visit interaction since all subjects receive the same treatment in the OLE.

The least squares (LS) mean change from baseline will be presented along with the associated 95% CI within each treatment group. The overall *P* value of the model will be presented to test





the null hypothesis that the change from baseline to subsequent study visit is 0 with a 2-sided alternative considering a difference in either direction.

In comparing treatments (active trifarotene cream HE1 groups minus vehicle), LS mean differences in change from baseline will be presented along with associated 95% CIs and *P* values. The null hypothesis that the difference in change from baseline in active trifarotene cream HE1 groups minus control vehicle is 0 with a 2-sided alternative considering a difference in either direction. Even if a difference from vehicle is observed, as described above, successful treatment is defined as clear/almost clear overall (IGA scores of 0 or 1) and at least a 2-grade change from baseline.

The observed value and change from baseline in IGA score will also be summarized descriptively by study visit and treatment group using descriptive statistics in addition to the above noted models for the Double-blind Period and OLE. Categorical IGA scores will also be presented.

## 8.1.2. Multiple Imputation

Multiple imputation (MI) of the primary endpoint will be performed as an analysis of sensitivity to missing data in the Double-blind Period only. Following database lock, thorough assessment on the extent of missing data due to COVID-19 will be carried out specifically as pertains to the primary and secondary endpoints. This will inform decisions around reasonability of imputing missing data for secondary endpoints in the Double-blind Period as well. The final determination will be documented in the CSR.

MI assumes that the statistical behavior of drug- and control-treated subjects after discontinuing study drug becomes that of the vehicle group. Multiple-imputations will be used to replace missing IGA outcomes using multiple draws from the posterior predictive distribution estimated from the vehicle treatment group. IGA scores will be imputed and then categorized as treatment success according to Section 8.1.1 above. A placebo-based pattern mixture model (PMM) will be utilized following the steps outlined in Ratitch B and O'Kelly, M.J. (2011)<sup>4</sup>.

Data are processed sequentially by repeatedly calling SAS® PROC MI to impute missing outcomes at study visit t = 1, ..., T. The following procedure is followed:

- *Initialization (Step 1)*. Set t = 0 (baseline study visit).
- Iteration (Step 2). Set t = t + 1. Create a dataset combined records from drug- and vehicle-treated subjects with columns for covariates X and outcomes at study visits 1, ..., t with outcomes for all subjects set to missing at study visit t and set to observed or imputed values at study visits 1, ..., t-1.
- *Imputation (Step 3)*. Run placebo-based pattern mixture model in SAS® PROC MI on this data to impute missing values for study visit *t* using previous outcomes for study visit 1 to t-1 and baseline covariates.
  - Replace imputed data for all subjects at study visit t with their observed values, whenever available. If t < T then go to Step 2, otherwise proceed to Step 4.
  - Repeat steps 1-3, m times with different seed values to create m imputed complete datasets. In this analysis, m will be assigned 50.



• Analysis (Step 4). For each completed dataset use the model as it would have been applied had the data been complete for the continuous outcome. The final inference on treatment difference is conducted from the multiple datasets, as implemented in SAS® PROC MI ANALYZE.

The steps for this approach are detailed below:

1. Transpose data horizontally by study visit and impute all non-monotone (intermittent) missing data using the Markov Chain Monte Carlo (MCMC) method of PROC MI. Note that this imputation will sample data within each treatment group. SAS pseudo code is provided below.

```
PROC MI DATA=example seed = 6654 NIMPUTE = 20 OUT = outdata1;
    BY <treatment>;
    MCMC chain=multiple impute=monotone;
    VAR <treatment> <baseline score> <visitX score> .. <visit6 score>;
RUN;
```

2. Using the imputed datasets from Step #1 that are now monotone missing (no intermittent missing data), a single call to PROC MI (including the MNAR statement) will be utilized to impute the monotone missing data. Within the call to PROC MI, one timepoint is imputed at a time. When imputing at time-point *t*, the imputation step will include all vehicle subjects, but only those from the active arms that have a value missing at time-point *t*. Subjects with non-missing data that are on active arms will not contribute to the estimation for this step.

Repeat the above step for all timepoints t. Thus, the data for timepoint t+1 uses the data imputed from previous timepoints.

SAS pseudo code is provided below. SAS accomplishes this iterative process in one step.

```
PROC MI DATA=example seed = 2617 NIMPUTE = 1 OUT = outdata1;
    BY _imputation_;
    CLASS <treatment>;
    MONOTONE REG ( / details);
    MNAR MODEL (<v1 score> .. <v6 score> /
        modelobs=(treatment=("vehicle"));
    VAR <baseline score> <v1 score> .. <vX score>..<v6 score> ;
RUN;
```

3. Pass the output from Step 2 into the model by the imputation variable (coalesce into one from each step above). When all missing data are imputed, PROC MIANALYZE will be used to combine the parameters from the analyses for inference.

## 8.2. Secondary Efficacy Analyses

## 8.2.1. Visual Index for Ichthyosis Severity (VIIS)

The investigator will rate the subject's condition using the 5-point VIIS for each body area (chest/abdomen, back, legs, and arms) and an overall score at all clinic visits. The scoring is as follows in Table 5.

## **Table 5: VIIS Scoring Definitions**



| Score | Definition |
|---|---|
| 0 | Normal skin; no perceptible scale, or smoothening |
| 1 | Areas of normal skin intermixed with areas showing smoothening (diminished fine skin markings; shininess; waxiness) or small scales (visible separated/fractured stratum corneum) |
| 2 | Confluent smoothening (diminished fine skin markings; shininess; waxiness) or small scales (visible separated/fractured stratum corneum) |
| 3 | Confluent scales (visibly separated/fractured stratum corneum) including some large (>1cm), thick scales |
| 4 | Confluent, primarily large, thick scales |

The change from baseline VIIS score will be analyzed using an MMRM. The MMRM model will include change from baseline in VIIS score as the dependent variable, treatment, study visit, treatment-by-visit interaction, and age group as fixed effects, subject as a random effect, and baseline VIIS score as a covariate. All post-baseline study visits will be included in the model; however, the primary comparison will be between the active trifarotene cream HE1 groups and vehicle at Day 90. An unstructured covariance matrix will be used to model the within-subject errors. The Kenward-Roger approximation will be used to estimate degrees of freedom. In case of convergence issues, other covariance structures will be explored including AR(1), CS, and VC with each model fit to find the covariance structure with the best fit. The fit statistics will be compared for all covariance structures; the structure with the smallest Akaike information criterion will be retained as the preferred model and noted in the resulting table. For the OLE period, the model will not include treatment or treatment-by-visit interaction since all subjects receive the same treatment in the OLE.

The LS mean change from baseline will be presented along with the associated 95% CI within each treatment group. The overall *P* value of the model will be presented to test the null hypothesis that the change from baseline to subsequent study visit is 0 with a 2-sided alternative considering a difference in either direction.

In comparing treatments (active trifarotene cream HE1 groups minus vehicle), LS mean differences in change from baseline will be presented along with associated 95% CIs and *P* values. The null hypothesis that the difference in change from baseline in active trifarotene cream HE1 groups minus control vehicle is 0 with a 2-sided alternative considering a difference in either direction.

The observed value and change from baseline in VIIS score will also be summarized descriptively by study visit and treatment group using descriptive statistics in addition to the above noted model for the Double-blind Period and OLE.





## 8.2.2. Individual Score for Roughness

The amount of roughness of the skin overall will be measured on a 5-point scale at all clinic visits. The scoring is as follows in Table 6.

**Table 6: Roughness Scoring Definitions** 

| Score | Definition |
|-------|---------------------------------------------------------------|
| 0 | Clear: Smooth skin |
| 1 | Almost clear: Hardly palpable roughness |
| 2 | Mild: Mild roughness on palpation (fine sand paper-like) |
| 3 | Moderate: Moderate, coarse roughness (coarse sand paper-like) |
| 4 | Severe: Very coarse skin (broken cornflakes-like) |

The change from baseline individual score for roughness will be analyzed using an MMRM. The MMRM model will include change from baseline in individual score for roughness as the dependent variable, treatment, study visit, treatment-by-visit interaction, and age group as fixed effects, subject as a random effect, and baseline individual score for roughness as a covariate. All post-baseline study visits will be included in the model; however, the primary comparison will be between the active trifarotene cream HE1 groups and vehicle at Day 90. An unstructured covariance matrix will be used to model the within-subject errors. The Kenward-Roger approximation will be used to estimate degrees of freedom. In case of convergence issues, other covariance structures will be explored including AR(1), CS, and VC with each model fit to find the covariance structure with the best fit. The fit statistics will be compared for all covariance structures; the structure with the smallest Akaike information criterion will be retained as the preferred model and noted in the resulting table. For the OLE period, the model will not include treatment or treatment-by-visit interaction since all subjects receive the same treatment in the OLE.

The LS mean change from baseline will be presented along with the associated 95% CI within each treatment group. The overall *P* value of the model will be presented to test the null hypothesis that the change from baseline to subsequent study visit is 0 with a 2-sided alternative considering a difference in either direction.

In comparing treatments (active trifarotene cream HE1 groups minus vehicle), LS mean differences in change from baseline will be presented along with associated 95% CIs and *P* values. The null hypothesis that the difference in change from baseline in active trifarotene cream HE1 groups minus control vehicle is 0 with a 2-sided alternative considering a difference in either direction.

The observed value and change from baseline in individual score for roughness will also be summarized descriptively by study visit and treatment group using descriptive statistics in addition to the above noted model for the Double-blind Period and OLE.





Additionally, the proportion of subjects who experience a 2-grade change from baseline to Day 90 in individual score for roughness will be summarized by treatment group and analyzed using a logistic regression model with treatment, baseline individual score for roughness, and age group as factors. The odds ratios and 95% CIs for the odds ratios will be presented. The difference in proportions between the active trifarotene cream HE1 groups and vehicle cream group, 95% CIs for the differences, and *P* values for the differences in treatment will also be presented.

The potential for heterogeneity of treatment effects will be assessed by testing treatment-by-factor interactions. The logistic regression model for the analysis will be expanded to include the treatment-by-age group interaction. In the event of quasi or complete separation, the logistic regression model will use Firth's penalized maximum likelihood estimation.

#### 8.2.3. Palm/Sole Assessment

Thickening of the skin on the palms and soles will be measured on a 5-point scale at all clinic visits. The scoring is as follows in Table 7.

**Table 7: Palm/Sole Scoring Definitions** 

| Score | Definition |
|---|---|
| 0 | Clear: No thickening, no roughness, no fissure |
| 1 | Almost clear: Only slight thickening, minimal to no roughness, no fissures |
| 2 | Mild: Some thickening, mild roughness on palpation, few fissures may be present |
| 3 | Moderate: Substantial and diffuse thickening, coarse roughness on palpation may be present, fissures may be present |
| 4 | Severe: Very thickened and rough skin, numerous fissures |

The change from baseline palm/sole assessment score will be analyzed using an MMRM. The MMRM model will include change from baseline in palm/sole assessment score as the dependent variable, treatment, study visit, treatment-by-visit interaction, and age group as fixed effects, subject as a random effect, and baseline palm/sole assessment score as a covariate. All post-baseline study visits will be included in the model; however, the primary comparison will be between the active trifarotene cream HE1 groups and vehicle at Day 90. An unstructured covariance matrix will be used to model the within-subject errors. The Kenward-Roger approximation will be used to estimate degrees of freedom. In case of convergence issues, other covariance structures will be explored including AR(1), CS, and VC with each model fit to find the covariance structure with the best fit. The fit statistics will be compared for all covariance structures; the structure with the smallest Akaike information criterion will be retained as the preferred model and noted in the resulting table. For the OLE period, the model will not include treatment or treatment-by-visit interaction since all subjects receive the same treatment in the OLE.





The LS mean change from baseline will be presented along with the associated 95% CI within each treatment group. The overall *P* value of the model will be presented to test the null hypothesis that the change from baseline to subsequent study visit is 0 with a 2-sided alternative considering a difference in either direction.

In comparing treatments (active trifarotene cream HE1 groups minus vehicle), LS mean differences in change from baseline will be presented along with associated 95% CIs and P values. The null hypothesis that the difference in change from baseline in active trifarotene cream HE1 groups minus control vehicle is 0 with a 2-sided alternative considering a difference in either direction.

The observed value and change from baseline in palm/sole assessment score will also be summarized descriptively by study visit and treatment group using descriptive statistics in addition to the above noted model for the Double-blind Period and OLE.

Additionally, the proportion of subjects who experience a 2-grade change from baseline to Day 90 in palm/sole assessment score will be summarized by treatment group and analyzed using a logistic regression model with treatment, baseline palm/sole assessment score, and age group as factors. The odds ratios and 95% CIs for the odds ratios will be presented. The difference in proportions between the active trifarotene cream HE1 groups and vehicle cream group, 95% CIs for the differences, and *P* values for the differences in treatment will also be presented.

The potential for heterogeneity of treatment effects will be assessed by testing treatment-by-factor interactions. The logistic regression model for the analysis will be expanded to include the treatment-by-age group interaction. In the event of quasi or complete separation, the logistic regression model will use Firth's penalized maximum likelihood estimation.

# 8.2.4. Quality of life per Dermatology Life Quality Index (DLQI) and Children's DLQI (cDLQI)

The DLQI is a dermatology-specific Quality of Life instrument for subjects aged 17 years and older. The cDLQI is for subjects aged 12 to 16 years. It is a 10-question validated questionnaire with 6 domains: symptoms and feelings, daily activities, leisure, work and school, personal relationships, and treatment. Higher scores indicate poorer quality of life. The investigator will use his or her judgment of the maturity of the subject to decide which version of the questionnaire to use; the same version will be used for the subject throughout the study.

The change from baseline DLQI/cDLQI score will be analyzed using an MMRM. The MMRM model will include change from baseline in DLQI/cDLQI score as the dependent variable, treatment, study visit, and treatment-by-visit interactionas fixed effects, subject as a random effect, and baseline DLQI/cDLQI score as a covariate. All post-baseline study visits will be included in the model; however, the primary comparison will be between the active trifarotene cream HE1 groups and vehicle at Day 90. An unstructured covariance matrix will be used to model the within-subject errors. The Kenward-Roger approximation will be used to estimate degrees of freedom. In case of convergence issues, other covariance structures will be explored including AR(1), CS, and VC with each model fit to find the covariance structure with the best fit. The fit statistics will be compared for all covariance structures; the structure with the smallest Akaike information criterion will be retained as the preferred model and noted in the resulting table.





The LS mean change from baseline will be presented along with the associated 95% CI within each treatment group. The overall *P* value of the model will be presented to test the null hypothesis that the change from baseline to subsequent study visit is 0 with a 2-sided alternative considering a difference in either direction.

In comparing treatments (active trifarotene cream HE1 groups minus vehicle), LS mean differences in change from baseline will be presented along with associated 95% CIs and *P* values. The null hypothesis that the difference in change from baseline in active trifarotene cream HE1 groups minus control vehicle is 0 with a 2-sided alternative considering a difference in either direction.

The observed value and change from baseline in DLQI/cDLQI score will also be summarized descriptively by study visit and treatment group using descriptive statistics in addition to the above noted model for the Double-blind Period.

#### **8.2.5.** Fissures

Fissuring will be assessed by recording the presence or absence of fissures, the number of fissures present, and the pain associated with each fissure. A fissure is a longitudinal and deep crack that separates the stratum corneum and may penetrate down to the dermis, causing pain and sometimes bleeding. The subject will assess pain associated with fissures as ranging from 0-3 (none, mild, moderate, severe).

The number and proportion of subjects with fissures present on palms or soles along with 95% CIs will be summarized by treatment group and study visit. A 2-sided Pearson's Chi-Square Test, or Fisher's Exact Test, as appropriate, will be performed at the 5% significance level to determine whether there is a significant difference between treatment groups. The null hypothesis that there is no difference in proportion of subjects with fissures present between active trifarotene cream HE1 and vehicle, with a 2-sided alternative considering a difference in either direction. The difference in proportions between active trifarotene cream HE1 and vehicle (active trifarotene cream HE1 minus vehicle), 95% CIs for the differences, and *P* values for the differences in treatment will also be presented.

The number of fissures and fissure pain level will be summarized descriptively by body area and treatment group.

## 8.3. Exploratory Efficacy Analyses

#### 8.3.1. Ectropion

The Ectropion Severity Score (ESS), has a maximum score of 8 points. A higher score indicates a worse ectropion. The score takes the severity of ectropion in terms of lateral and medial apposition, scleral show, conjunctival show, and roundness of the eye into account and gives an indication of the functional aspects involved in ectropion by scoring redness, excess tear film, and the position of the lacrimal punctum. The scoring is as follows in Table 8.

**Table 8: Ectropion Scoring** 

| Points per Item |
|-----------------|



| | 0 | 0.5 | 1 |
|--------------------|-------------|----------|----------|
| Lateral apposition | Nonaffected | - | Affected |
| Medial apposition | Nonaffected | - | Affected |
| Sceral show | No | ≤ 1 mm | > 1mm |
| Conjunctival show | No | - | Yes |
| Excess tear film | No | - | Yes |
| Redness of the eye | No | - | Yes |
| Round canthus | No | - | Yes |
| Punctum lacrimale | Invisible | Emerging | Visible |
| Maximum score | | | 8 points |

The observed value and change from baseline in ectropion score will be summarized descriptively by study visit and treatment group using descriptive statistics for the Double-blind Period and OLE.

## 8.3.2. Quality of Life per EQ-5D-5L and EQ-5D-Y

The EQ-5D is a measure of health related quality of life. The EQ-5D consists of a descriptive system and the EQ visual analog scale (VAS). The EQ-5D-5L is intended for use in adult subjects, while the EQ-5D-Y is to be used for children and adolescents. The investigator will use his or her judgment of the maturity of the subject to decide which version of the EQ-5D to use; the same version will be used for the subject throughout the study. The descriptive system comprises 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The EQ VAS records the subject's self-rated health on a vertical 0-100 VAS. This can be used as a quantitative measure of health outcome that reflects the subject's own judgement.

The observed value and change from baseline in EQ-5D-5L/EQ-5D-Y score will be summarized descriptively by study visit and treatment group using descriptive statistics for the Double-blind Period and OLE.

## 9. Safety and Tolerability Analysis

Safety variables include treatment-emergent AEs, clinical laboratory values, vital signs, ECG readings, local tolerability assessments, and physical examination results. No formal inferential analyses will be conducted for safety variables in either period.





Safety analyses through Day 90 of the Double-blind Period will be conducted using data from the Safety population and safety analyses in the OLE will be conducted using the OLE Safety population.

#### 9.1. Adverse Events

All AEs, TEAEs, and SAEs will be coded using the MedDRA dictionary Version 21.1.

Treatment-emergent AEs are defined as:

- AEs with onset at the time of or following the start of treatment with study drug through 14 days after the last application of study drug, or
- AEs starting prior to the start of treatment but increasing in severity or relationship at the time of, or following, the start of treatment with study drug through the last application of study drug.

The causal relationship of the AE to the study drug is determined by the investigator as Not Related, Unlikely Related, Possibly Related, and Related. These will be mapped to Unrelated (Not Related or Unlikely Related) and Related (Possibly Related, or Related).

Adverse event severity grades are reported as mild, moderate, or severe.

Summaries of incidence rates (frequencies and percentages) of individual TEAEs will be presented by SOC, PT, and treatment group for the Double-blind Period and OLE. Such summaries will be displayed for all TEAEs, TEAEs by maximum severity, and TEAEs by relationship.

Each subject will be counted only once within each summation level (SOC and PT). If a subject experiences more than 1 TEAE within each summation level, the TEAE with the strongest relationship or the maximum severity, as appropriate, will be included in the summaries of relationship and severity. If a particular event is missing the severity and/or relationship, then the strongest possible severity or relationship will be assumed for analysis (severity = severe, relationship = related).

Incidences will be presented by descending frequency of SOC and PT within SOC, and then alphabetically within PT where the incidence is the same; this is based on overall subjects then alphabetically in case of a tie.

Missing and partially missing AE start and/or stop dates and times will be imputed, for the purpose of statistical analysis, according to the specifications described in Section 6.1.8.

In the AE data listings, all AEs will be displayed. AEs that are treatment emergent will be flagged.

#### 9.1.1. Adverse Events Leading to Withdrawal

A summary of incidence rates (frequencies and percentages) of TEAEs leading to withdrawal of study drug, by treatment group, SOC, and PT will be prepared for both the Double-blind Period and OLE.





A data listing of AEs leading to withdrawal of study drug during each period will also be provided, displaying details of the event(s) captured on the CRF.

#### 9.1.2. Deaths and Serious Adverse Events

Any deaths that occur during the study will be listed.

Serious adverse events will be listed and also tabulated by SOC and PT and presented by treatment group for the Double-blind Period and overall for the OLE.

## 9.2. Clinical Laboratory Evaluations

Laboratory tests (clinical chemistry, hematology, coagulation, and quantitative urinalysis) will be performed at Screening, Baseline, Day 30, Day 90, Day 120, and Day 180. Results will be summarized descriptively by treatment group and study visit as both observed values and change from baseline values for the Double-blind Period and OLE. See Section 6.1.1 for the definition of baseline. Number and percentage of subjects with abnormal qualitative urinalysis results will be provided by treatment group and study visit.

The number of subjects with clinical laboratory values below, within, or above normal ranges, by study visit will be tabulated (shift tables) for each clinical laboratory parameter by treatment group.

Laboratory values will be displayed in the data listings and those that are outside the normal range will be flagged and presented along with corresponding normal ranges (if available). A separate listing of abnormal laboratory values will be provided. All study visits within a parameter for a subject will be presented if at least 1 study visit within that parameter has an abnormal result.

Serology results and pregnancy test results will be listed separately.

## 9.3. Vital Signs

Vital signs will be collected at Screening, Baseline, Day 14, Day 30, Day 60, Day 90, Day 120, Day 150, Day 180, and Day 194. Descriptive summaries of actual values and changes from baseline will be calculated for systolic blood pressure (mmHg), diastolic blood pressure (mmHg), and pulse (bpm).

The number of subjects with vital sign values below, within, or above normal ranges, by study visit will be tabulated (shift tables) for each parameter by treatment group.

These summaries will be presented by study visit and treatment group. See Section 6.1.1 for the definition of baseline.

## 9.4. Electrocardiograms

12-Lead ECGs will be collected at Screening, Baseline, Day 30, Day 90, Day 120, and Day 180. For subjects in the PK substudy, additional ECGs will be performed postdose during serial blood sampling on Day 1 and Day 30. Descriptive summaries will be presented for heart rate (bpm),




PR interval (ms), QRS interval (ms), uncorrected QT interval (ms), QTcF (ms). These summaries will be presented by study visit and treatment group.

The number and percentage of subjects with normal and abnormal ECG results will be summarized by treatment group and study visit.

## 9.5. Local Tolerability

During all clinic visits, the investigator will assess local tolerability (Scale: 0-3 [none, mild, moderate, severe]) for each treated body area (chest/abdomen, back, arms, legs, and face/neck).

Descriptive summaries of the investigator's assessment of erythema, stinging/burning, and pruritus will be presented by body area, period, treatment group, and study visit.

## 9.6. Physical Examination

Physical examinations will be performed at Screening, Baseline, Day 90, Day 180, and Day 194. The number and percentage of subjects with normal and abnormal findings in the complete physical examination will be displayed for each treatment group in each period.

#### 9.7. Concomitant Medication

Prior and concomitant medications, coded using World Health Organization-Drug Dictionary Enhanced (WHO-DDE) (September 2018), will be summarized descriptively by Anatomical Therapeutic Chemical (ATC) classification Level 4 and PT (i.e., ATC classification Level 5), if applicable, using counts and percentages for the Safety Population.

Prior medications and concomitant medications will be presented separately. The assignment of medications as prior and/or concomitant will be done as follows:

- **Prior medications:** Medications that started before the first dose of study drug will be considered prior medications whether or not they were stopped before dose.
- Concomitant medications: Any medications continuing or starting after the first dose of study drug through the end of study will be considered to be concomitant.

If a medication starts prior to the first dose and continues after the first dose it will be considered both prior and concomitant. Prior and concomitant medications will also be listed. Prior and concomitant medications will be summarized descriptively by treatment using counts and percentages.

### 9.8. COVID-19 Visit Impact

A listing of the COVID-19 visit impact log will be presented which will display which (if any) study visits were impacted by the pandemic. The listing will display if the visit was performed and if the visit type was adjusted as well as the reason(s) for adjustment.

### 10. Changes from Planned Analysis

Age was added as a factor for MMRM analyses because the study is enrolling both adults and





adolescents.

## 11. Other Planned Analysis

### 11.1. Pharmacokinetic Analysis

The pharmacokinetic characterization of drug concentrations for each dose to be profiled will use noncompartmental analysis (NCA).

Samples for PK will be drawn from all subjects at Baseline and at each clinic visit for trough values. Subjects who provide written informed consent to participate in the optional PK substudy will provide blood samples for PK analysis predose on Day 1 and at 1, 2, 4, 8, 12, and 24 hours postdose on Day 1 and Day 30.

The PK parameter estimates will be completed using WinNonlin (Pharsight Corporation) software using the actual elapsed times from dose administration to sample collection (i.e., not nominal time).

Standard PK parameters assessed will include measures of the extent of absorption using estimates of the Area under the plasma concentration-time curve from time 0 to the time of the last quantifiable plasma concentration (AUC<sub>0-t</sub>), Area under the plasma concentration-time curve from time 0 to infinity (if data permits) (AUC<sub>0-inf</sub>) and rate-of-absorption using the maximum serum concentration ( $C_{max}$ ), the time of  $C_{max}$  ( $T_{max}$ ), apparent first order terminal elimination half-life ( $t_{1/2}$ ), apparent terminal phase rate constant ( $\lambda_z$ ) (if data permits).

For noncompartmental analysis, plasma concentrations will be listed and summarized at each time point using descriptive statistics. Descriptive statistics reported will include the arithmetic mean, SD, CV%, geometric mean, minimum, maximum, and median. Only the range and the median will be reported for  $T_{max}$ , as this is a categorical parameter. The PK parameters will also be summarized by treatment using descriptive statistics.

Individual plasma concentration plots and mean data graphs will be produced using both linear and semi-logarithmic scales. Mean data graphs will show plasma concentration profiles by treatment group. Pharmacokinetic plasma parameter estimates and summaries will be completed for the subjects in the PK population.





## 11.2. Photography

Photography collection dates will be listed.

### 12. References

- 1. US Federal Register. (1998) International Conference on Harmonization; Guidance on Statistical Principles for Clinical Trials. Department of Health and Human Services: Food and Drug Administration [Docket No. 97D-0174]. Federal Register Volume 63, Number 179, pages 49583-49598. September 16, 1998.
- 2. ASA. (2016) Ethical Guidelines for Statistical Practice. Prepared by the Committee on Professional Ethics, April 2016. http://www.amstat.org/about/ethicalguidelines.cfm
- 3. RSS. (2014) The Royal Statistical Society: Code of Conduct, 2014. http://www.rss.org.uk/Images/PDF/join-us/RSS-Code-of-Conduct-2014.pdf.
- 4. Ratitich, B. and O'Kelly, M.J. (2011). Implementation of Pattern-Mixture Models Using Standard SAS / STAT Procedures.

### 13. Tables, Listings, and Figures

All listings, tables, and figures will have a header showing the sponsor company name and protocol and a footer showing the version of SAS, the file name and path, and the source of the data (CRF page or listing number).

The following reporting conventions will be adopted for the presentation of study data. These conventions will enhance the review process and help to standardize the presentation with common notations.

### **General Reporting Conventions**

- All tables and data listings will be developed in landscape orientation.
- Specialized text styles, such as bolding, italics, borders, shading, and superscripted and subscripted text will not be used in tables, figures, and data listings unless they add significant value to the table, figure, or data listing.
- Only standard keyboard characters should be used in tables and data listings. Special characters, such as nonprintable control characters, printer-specific characters, or font specific characters, will not be used on a table, figure, or data listing.
- All titles will be centered on a page. All footnotes will be left justified and at the bottom of a page.
- Missing values for both numeric and character variables will be presented as blanks in a table or data listing. A value of zero may be used if appropriate to identify when the frequency of a variable is not observed.
- All date values will be presented as ddmmmyyyy (e.g., 29AUG2011) format.
- If applicable, all observed time values will be presented by using a 24-hour clock HH:MM:SS format (e.g., 01:35:45 or 11:26). Seconds should only be reported if they were measured as part of the study.
- Adverse events with missing MedDRA coding will have their system organ class and/or





preferred term presented as "Not Coded" in the tables. The "Not Coded" frequencies will be sorted to the end of the tables. This will only be applicable for any deliveries sent before database lock (e.g., for dry runs on blinded data).

• Programming notes may be inserted into the shells, these notes will not appear in the final output.

### **Population Summary Conventions**

- Population sizes may be presented for each classification factor as totals in the column header as (N=xxx), where appropriate.
- All population summaries for categorical variables will include all categories that were planned and for which the subjects may have had a response. Percentages corresponding to null categories (cells) will be suppressed; however, counts and percentages of missing values may be needed.
- All population summaries for continuous variables will include: N, mean, SD, median, minimum, and maximum. Other summaries (e.g., number missing, 95% CIs) may be used as appropriate. The precision of the maximum and minimum will match the maximum precision in the data. The mean and median will have 1 additional decimal place. The SD will have 2 additional decimal places.
- All percentages are rounded (where, for example, 0.05% is rounded up to 0.1%) and reported to a single decimal point (xx.x%).
- A percentage of 0% will not be displayed (i.e., only the count of 0 will be displayed), and a percentage of 100% will be displayed with 0 decimal places.
- All *P* values will be displayed in four decimals and rounded using standard scientific notation (e.g., 0.XXXX). If a *P* value less than 0.0001 occurs it will be shown in tables as <0.0001.

### 13.1. Planned Table Descriptions

The following are planned summary tables for protocol number 18-ICH-001. The table numbers and page numbers are place holders only and will be determined when the tables are produced.



# **Table 9: Demographic Data Summary Tables and Figures**

| Number | Population | Title | Unique/Non-unique |
|---|---|---|---|
| Table 14.1.1.1 | ITT | Summary of Subject Disposition | Unique |
| Table 14.1.1.2 | OLE ITT | Summary of Subject Disposition | Non-unique |
| Table 14.1.2.1 | ITT | Demographics and Baseline Characteristics | Unique |
| Table 14.1.2.2 | OLE ITT | Demographics and Baseline Characteristics | Non-unique |
| Table 14.1.3 | Safety | Summary of Medical Histories by System Organ Class and Preferred Term | Unique |
| Table 14.1.4 | Safety | Summary of Prior Medications by ATC Class Level 4 and Preferred Term | Unique |
| Table 14.1.5.1 | Safety | Summary of Drug Accountability (Drug Returned and Dispensed) | Unique |
| Table 14.1.5.2 | OLE<br>Safety | Summary of Drug Accountability (Drug Returned and Dispensed) | Non-unique |
| Table 14.1.5.3 | Safety | Summary of Treatment Exposure and Compliance | Unique |
| Table 14.1.5.4 | OLE<br>Safety | Summary of Treatment Exposure and Compliance | Non-unique |

# 13.2. Efficacy Data

# **Table 10: Efficacy Data**

| Number | Population | Title | Unique/Non-unique |
|---|---|---|---|
| 14.2.1.1.1 | ITT | Primary Analysis: Logistic Regression Analysis of Successful<br>Resolution of LI | Unique |
| 14.2.1.1.2 | OLE ITT | Proportion of Subjects with Successful Resolution of LI in the OLE | Unique |
| 14.2.1.2.1 | mITT | Primary Analysis, Sensitivity: Logistic Regression Analysis of<br>Successful Resolution of LI | Non-unique |
| 14.2.1.2.2 | OLE mITT | Proportion of Subjects with Successful Resolution of LI in the OLE | Non-unique |
| 14.2.1.3.1 | PP | Primary Analysis, Sensitivity: Logistic Regression Analysis of<br>Successful Resolution of LI | Non-unique |



| Number | Population | Title | Unique/Non-unique |
|---|---|---|---|
| 14.2.1.3.2 | OLE PP | Proportion of Subjects with Successful Resolution of LI in the OLE | Non-unique |
| 14.2.1.4 | ITT | Primary Analysis, Sensitivity: Logistic Regression Analysis of<br>Successful Resolution of LI Using Multiple Imputation | Non-unique |
| 14.2.1.5.1 | ITT | Logistic Regression Analysis of 50% Reduction in IGA score from Baseline | Non-unique |
| 14.2.1.5.2 | OLE ITT | Proportion of Subjects with a 50% Reduction in IGA score from Baseline | Non-unique |
| 14.2.1.6.1 | ITT | MMRM Analysis of Change from Baseline in IGA Score | Unique |
| 14.2.1.6.2 | OLE ITT | MMRM Analysis of Change from Baseline in IGA Score | Non-unique |
| 14.2.1.7.1 | ITT | Categorical IGA Scores | Unique |
| 14.2.1.7.2 | OLE ITT | Categorical IGA Scores | Non-unique |
| 14.2.2.1 | ITT | Secondary Analysis: MMRM Analysis of Change from Baseline in VIIS Score | Non-unique |
| 14.2.2.2 | OLE ITT | MMRM Analysis of Change from Baseline in VIIS Score | Non-unique |
| 14.2.3.1 | ITT | Secondary Analysis: MMRM Analysis of Change from Baseline in Individual Score for Roughness | Non-unique |
| 14.2.3.2 | OLE ITT | MMRM Analysis of Change from Baseline in Individual Score for Roughness | Non-unique |
| 14.2.3.3 | ITT | Logistic Regression Analysis of 2-grade Change in Individual<br>Score for Roughness from Baseline | Non-unique |
| 14.2.4.1 | ITT | Secondary Analysis: MMRM Analysis of Change from Baseline in Palm/Sole Assessment | Non-unique |
| 14.2.4.2 | OLE ITT | MMRM Analysis of Change from Baseline in Palm/Sole<br>Assessment | Non-unique |
| 14.2.4.3 | ITT | Logistic Regression Analysis of 2-grade Change in Palm/Sole<br>Assessment from Baseline | Non-unique |
| 14.2.5.1 | ITT | Secondary Analysis: MMRM Analysis of Change from Baseline in Dermatology Life Quality Index | Non-unique |
| 14.2.5.2 | ITT | Secondary Analysis: MMRM Analysis of Change from Baseline in Children's Dermatology Life Quality Index | Non-unique |
| 14.2.6.1.1 | ITT | Secondary Analysis: Presence of Fissures on Palms or Soles | Unique |
| 14.2.6.1.2 | OLE ITT | Presence of Fissures on Palms or Soles | Unique |
| 14.2.6.2.1 | ITT | Secondary Analysis: Summary of Number of Fissures and Fissure Pain Level | Unique |
| 14.2.6.2.2 | OLE | Summary of Number of Fissures and Fissure Pain Level | Non-unique |





| Number | Population | Title | Unique/Non-unique |
|---|---|---|---|
| 14.2.7.1 | ITT | Exploratory Analysis: Summary of Change from Baseline in Ectropion Score | Unique |
| 14.2.7.2 | OLEITT | Summary of Change from Baseline in Ectropion Score | Non-unique |
| 14.2.8.1 | ITT | Exploratory Analysis: Change from Baseline in EQ-5D-5L | Non-unique |
| 14.2.8.2 | ITT | Exploratory Analysis: Change from Baseline in EQ-5D-Y | Non-unique |



# 13.3. Safety Data

**Table 11: Safety Data** 

| | | Title | Unique/Non-unique |
|---|---|---|---|
| 14.3.1.1.1 | Safety | Overall Summary of Treatment Emergent Adverse Events during the Double-blind Period | Unique |
| 14.3.1.1.2 | OLE<br>Safety | Overall Summary of Treatment Emergent Adverse Events during the OLE | Non-unique |
| 14.3.1.2.1 | Safety | Incidence of Treatment Emergent Adverse Events during the Double-blind Period by System Organ Class and Preferred Term | Unique |
| 14.3.1.2.2 | OLE<br>Safety | Incidence of Treatment Emergent Adverse Events during the OLE Period by System Organ Class and Preferred Term | Non-unique |
| 14.3.1.3.1 | Safety | Incidence of Treatment Emergent Adverse Events during the Double-blind Period by System Organ Class, Preferred Term, and Maximum Severity | Unique |
| 14.3.1.3.2 | OLE<br>Safety | Incidence of Treatment Emergent Adverse Events during the OLE by System Organ Class, Preferred Term, and Maximum Severity | Non-unique |
| 14.3.1.4.1 | Safety | Incidence of Treatment Emergent Adverse Events during the Double-blind Period by System Organ Class, Preferred Term, and Relationship to Study Drug | Unique |
| 14.3.1.4.2 | OLE<br>Safety | Incidence of Treatment Emergent Adverse Events during the OLE by System Organ Class, Preferred Term, and Relationship to Study Drug | Non-unique |
| 14.3.2.1.1 | Safety | Incidence of Adverse Events Leading to Withdrawal during the Double-blind Period by SOC, PT, and Treatment | Non-unique |
| 14.3.2.1.2 | OLE<br>Safety | Incidence of Adverse Events Leading to Withdrawal during the OLE Period by SOC, PT, and Treatment | Non-unique |
| 14.3.2.2.1 | Safety | Incidence of Serious Adverse Events during the Double-blind<br>Period by SOC, PT, and Treatment | Non-unique |
| 14.3.2.2.2 | OLE<br>Safety | Incidence of Serious Adverse Events during the OLE by SOC, PT, and Treatment | Non-unique |
| 14.3.3.1.1 | Safety | Listing of Adverse Events Leading to Withdrawal during the Double-blind Period | Unique |
| 14.3.3.1.2 | OLE<br>Safety | Listing of Adverse Events Leading to Withdrawal during the Double-blind Period | Non-unique |
| 14.3.3.2.1 | Safety | Listing of Serious Adverse Events during the Double-blind<br>Period | Non-unique |
| 14.3.3.2.2 | Safety | Listing of Serious Adverse Events during the OLE | Non-unique |
| 14.3.3.3.1 | Safety | Listing of Deaths during the Double-blind Period | Non-unique |



| Number | umber Population Title | | Unique/Non-unique |
|---|---|---|---|
| 14.3.3.3.2 | Safety | Listing of Deaths during the OLE | Non-unique |
| 14.3.4.1 | Safety | Listing of Abnormal Laboratory Data | Unique |
| 14.3.5.1.1.1 | Safety | Laboratory Data: Change from Baseline in Clinical Chemistry<br>Parameters by Study Visit | Unique |
| 14.3.5.1.1.2 | OLE<br>Safety | Laboratory Data: Change from Baseline in Clinical Chemistry<br>Parameters by Study Visit | Non-unique |
| 14.3.5.1.2.1 | Safety | Laboratory Data: Shift from Baseline in Clinical Chemistry<br>Parameters by Study Visit | Unique |
| 14.3.5.1.2.2 | OLE<br>Safety | Laboratory Data: Shift from Baseline in Clinical Chemistry<br>Parameters by Study Visit | Non-unique |
| 14.3.5.2.1.1 | Safety | Laboratory Data: Change from Baseline in Hematology<br>Parameters by Study Visit | Non-unique |
| 14.3.5.2.1.2 | OLE<br>Safety | Laboratory Data: Change from Baseline in Hematology<br>Parameters by Study Visit | Non-unique |
| 14.3.5.2.2.1 | Safety | Laboratory Data: Shift from Baseline in Hematology<br>Parameters by Study Visit | Non-unique |
| 14.3.5.2.2.2 | OLE<br>Safety | Laboratory Data: Shift from Baseline in Hematology<br>Parameters by Study Visit | Non-unique |
| 14.3.5.3.1.1 | Safety | Laboratory Data: Change from Baseline in Coagulation<br>Parameters by Study Visit | Non-unique |
| 14.3.5.3.1.2 | OLE<br>Safety | Laboratory Data: Change from Baseline in Coagulation<br>Parameters by Study Visit | Non-unique |
| 14.3.5.3.2.1 | Safety | Laboratory Data: Shift from Baseline in Coagulation<br>Parameters by Study Visit | Non-unique |
| 14.3.5.3.2.2 | OLE<br>Safety | Laboratory Data: Shift from Baseline in Coagulation<br>Parameters by Study Visit | Non-unique |
| 14.3.5.4.1.1 | Safety | Laboratory Data: Change from Baseline in Quantitative<br>Urinalysis Parameters by Study Visit | Non-unique |
| 14.3.5.4.1.2 | OLE<br>Safety | Laboratory Data: Change from Baseline in Quantitative<br>Urinalysis Parameters by Study Visit | Non-unique |
| 14.3.5.4.2.1 | Safety | Laboratory Data: Shift from Baseline in Quantitative<br>Urinalysis Parameters by Study Visit | Non-unique |
| 14.3.5.4.2.2 | OLE<br>Safety | Laboratory Data: Shift from Baseline in Quantitative<br>Urinalysis Parameters by Study Visit | Non-unique |
| 14.3.5.4.3.1 | Safety | Laboratory Data: Summary of Qualitative Urinalysis<br>Parameters by Study Visit | Unique |



| Number | Tumber Population Title | | Unique/Non-unique |
|---|---|---|---|
| 14.3.5.4.3.2 | OLE<br>Safety | Laboratory Data: Summary of Qualitative Urinalysis<br>Parameters by Study Visit | Non-unique |
| 14.3.6.1.1 | Safety | Summary of Vital Signs by Study Visit | Non-unique |
| 14.3.6.1.2 | OLE<br>Safety | Summary of Vital Signs by Study Visit | Non-unique |
| 14.3.6.2.1 | Safety | Summary of 12-Lead Electrocardiogram by Study Visit | Non-unique |
| 14.3.6.2.2 | OLE<br>Safety | Summary of 12-Lead Electrocardiogram by Study Visit | Non-unique |
| 14.3.6.2.3 | Safety | Summary of 12-Lead Electrocardiogram Interpretation by Study Visit | Unique |
| 14.3.6.2.4 | OLE<br>Safety | Summary of 12-Lead Electrocardiogram Interpretation by Study Visit | Unique |
| 14.3.6.3.1 | Safety | Summary of Local Tolerability Assessments by Study Visit | Unique |
| 14.3.6.3.2 | OLE<br>Safety | Summary of Local Tolerability Assessments by Study Visit | Non-unique |
| 14.3.6.4.1 | Safety | Summary of Physical Examination Results by Study Visit | Unique |
| 14.3.6.4.2 | OLE<br>Safety | Summary of Physical Examination Results by Study Visit | Non-unique |
| 14.3.6.5.1 | Safety | Summary of Concomitant Medications by ATC Class Level 4 and Preferred Term | Non-unique |
| 14.3.6.5.2 | OLE<br>Safety | Summary of Concomitant Medications by ATC Class Level 4 and Preferred Term | Non-unique |



#### 13.4. Pharmacokinetic Data

Table 12: Pharmacokinetic Data

| Number | Population | Title | Unique/Non-unique |
|---|---|---|---|
| 14.4.1.1 | Safety | Summary of Pharmacokinetic Concentrations by Study Visit | Unique |
| 14.4.1.2 | Safety | Summary of Pharmacokinetic Parameters | Unique |

## 13.5. Planned Listing Descriptions

The following are planned data and patient/subject data listings for protocol number 18-ICH-001.

In general, 1 listing will be produced per CRF domain. All listings will be sorted by treatment, site, and subject number. All calculated variables will be included in the listings.

In all listings a blank line will be placed between each subject. Within a data listing, if an item appears line after line (e.g., repetition of subject number), then only the first occurrence will be displayed.

In data listings, the information for 1 subject will be kept on 1 page if at all possible, rather than splitting a subject's information across pages.

**Table 13: Planned Listings** 

| Number | Population | Title | Unique/Non-unique | Provide at Topline? |
|---|---|---|---|---|
| 16.2.1 | All Subjects | Subject Disposition | Unique | |
| 16.2.2.1 | All Subjects | Inclusion and Exclusion Criteria | Unique | |
| 16.2.2.2 | All Subjects | Screen Failures | Unique | |
| 16.2.2.3 | All Subjects | Protocol Deviations | Unique | |
| 16.2.3 | All Subjects | Analysis Populations | Unique | |
| 16.2.4.1 | All Subjects | Subject Demographics | Unique | |
| 16.2.4.2 | All Subjects | Informed Consent and Reconsent | Unique | |
| 16.2.4.3 | All Subjects | Medical History | Unique | |
| 16.2.5.1 | All Subjects | Initial Study Drug Application | Unique | |
| 16.2.5.2 | All Subjects | Drug Accountability (Dispensed and Returned) | Unique | |
| 16.2.5.3 | All Subjects | Subject Diary | Unique | |
| 16.2.5.4.1 | All Subjects | Pharmacokinetic Sample Collection | Unique | |
| 16.2.5.4.2 | All Subjects | Pharmacokinetic Sample Collection (Substudy) | Unique | |
| 16.2.5.4.3 | PK | Pharmacokinetic Concentrations | Unique | |



| Number | Population | Title | Unique/Non-unique | Provide at Topline? |
|---|---|---|---|---|
| 16.2.5.4.4 | All Subjects | Pharmacokinetic Calculated<br>Parameters | Unique | |
| 16.2.6.1 | All Subjects | Investigator's Global Assessment (IGA) | Unique | |
| 16.2.6.2 | All Subjects | Visual Index for Ichthyosis (VIIS) | Non-unique | |
| 16.2.6.3 | All Subjects | Roughness Assessment | Non-unique | |
| 16.2.6.4 | All Subjects | Palm/Sole Assessment | Non-unique | |
| 16.2.6.5.1 | All Subjects | Quality of Life per Dermatology<br>Life Quality Index (DLQI) | Non-unique | |
| 16.2.6.5.1 | All Subjects | Quality of Life per Children's<br>Dermatology Life Quality Index<br>(DLQI) | Non-unique | |
| 16.2.6.6 | All Subjects | Fissuring Assessment | Unique | |
| 16.2.6.7 | All Subjects | Ectropion Score | Non-unique | |
| 16.2.6.8 | All Subjects | EQ-5D | Non-unique | |
| 16.2.7.1 | All Subjects | Adverse Events | Unique | |
| 16.2.8.1 | All Subjects | Laboratory Data: Clinical Chemistry | Unique | |
| 16.2.8.2 | All Subjects | Laboratory Data: Hematology | Non-unique | |
| 16.2.8.3 | All Subjects | Laboratory Data: Coagulation | Non-unique | |
| 16.2.8.4 | All Subjects | Laboratory Data: Urinalysis | Non-unique | |
| 16.2.8.5 | All Subjects | Laboratory Data: Serology | Non-unique | |
| 16.2.8.6 | All Subjects | Laboratory Data: Pregnancy Tests | Non-unique | |
| 16.2.9.1 | All Subjects | Vital Signs | Non-unique | |
| 16.2.9.2 | All Subjects | 12-Lead Electrocardiogram | Non-unique | |
| 16.2.9.3 | All Subjects | Local Tolerability Assessments | Unique | |
| 16.2.9.4 | All Subjects | Physical Examination | Unique | |
| 16.2.9.5 | All Subjects | Prior and Concomitant Medications | Unique | |
| 16.2.9.6 | All Subjects | Photography | Unique | |
| 16.2.9.7 | All Subjects | Trial Continuation | Unique | |
| 16.2.9.8 | All Subjects | Telephone Contact | Unique | |
| 16.2.9.9 | All Subjects | COVID-19 Visit Impact Log | Unique | |

# 13.6. Planned Figure Descriptions

Not applicable.





# **Table 14: Planned Figures**

Not Applicable.





## 14. Tables, Listings, and Listing Shells

# 14.1. Standard Layout for all Tables, Listings, and Figures

The following standard layout will be applied to all tables, listings, and figures in support of this study. Note that programming notes may be added if appropriate after each TLF shell.





# Figure 3: Standardized Layout

| Mayne Pharma | Page xx of xx |
|---|---|
| Protocol: 18-ICH-001 | <version></version> |
| < Table, Listing, Figure > xx.x.x | |
| <title figure="" listing="" of="" or="" table="">&lt;/td&gt;&lt;td&gt;&lt;/td&gt;&lt;/tr&gt;&lt;tr&gt;&lt;td&gt;&lt;Study Population and if applicable subgroup Description&gt;&lt;/td&gt;&lt;td&gt;&lt;/td&gt;&lt;/tr&gt;&lt;tr&gt;&lt;td&gt;&lt;/td&gt;&lt;td&gt;&lt;/td&gt;&lt;/tr&gt;&lt;tr&gt;&lt;td&gt;Body of Table, Listing or Figure&lt;/td&gt;&lt;td&gt;&lt;/td&gt;&lt;/tr&gt;&lt;tr&gt;&lt;td&gt;&lt;/td&gt;&lt;td&gt;&lt;/td&gt;&lt;/tr&gt;&lt;tr&gt;&lt;td&gt;&lt;Note: If directly Applicable&gt;&lt;/td&gt;&lt;td&gt;&lt;/td&gt;&lt;/tr&gt;&lt;tr&gt;&lt;td&gt;Footnote 1 &lt; if applicable &gt; Recommendation is to keep footnotes to a minimum&lt;/td&gt;&lt;td&gt;&lt;/td&gt;&lt;/tr&gt;&lt;tr&gt;&lt;td&gt;Footnote 2 &lt; if applicable &gt;&lt;/td&gt;&lt;td&gt;&lt;/td&gt;&lt;/tr&gt;&lt;tr&gt;&lt;td&gt;Footnote n &lt; if applicable&gt;&lt;/td&gt;&lt;td&gt;&lt;/td&gt;&lt;/tr&gt;&lt;tr&gt;&lt;td&gt;&lt;pre&gt;&lt;pgm path&gt;\&lt;pgm name.sas&gt;&lt;/pre&gt;&lt;/td&gt;&lt;td&gt;&lt;/td&gt;&lt;/tr&gt;&lt;tr&gt;&lt;td&gt;Executed on DDMONYYYY at hh:mm on data from DDMONYYYY; SAS Version 9.X&lt;/td&gt;&lt;td&gt;&lt;/td&gt;&lt;/tr&gt;&lt;/tbody&gt;&lt;/table&gt;</title> | |





## 14.2. Planned Table Shells

See Figure 4 below.





**Figure 4: Planned Table Shells** 

#### Table 14.1.1.1 Summary of Subject Disposition ITT Population

| Category | Trifarotene cream HE1<br>100 ug/g<br>(N=XXX) | Trifarotene cream HE1<br>200 ug/g<br>(N=XXX) | Vehicle<br>(N=XXX) | Overall<br>(N=XXX) |
|---|---|---|---|---|
| ITT Population | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Safety Population | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| mITT Population | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| PP Population | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| PK Population | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Completed Continuing | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Completed not Continuing to OLE | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Ongoing in Double-blind Study | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Early Discontinuation of Medication | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

Abbreviations: ITT = intent-to-treat; mITT = modified intent-to-treat; OLE = open label extension; PK = pharmacokinetic; PP = per protocol.

Note: Percentages are n/Number of subjects in the ITT Population within randomized treatment group and overall\*100. The ITT population includes all randomized subjects. The Safety population includes all subjects who are randomized to treatment and receive at least 1 application of study drug in the Double-blind Period. The mITT population includes all subjects in the Safety population with at least 1 postbaseline assessment of efficacy in the Double-blind period. The PP population includes all subjects in the mITT population who met all inclusion criteria and no exclusion criteria, were compliant with study drug application, and who had no significant protocol deviations. The PK population includes all subjects in the Safety population who have at least 1 plasma sample with quantifiable concentration. Completed continuing represents subjects who completed study visits and Double-blind treatment period (Day 90) and are continuing to OLE. Completed not continuing represents subjects who completed study visits and Double-blind treatment period (Day 90) but are not continuing to OLE. Early discontinuation of medication represent subjects who did not complete treatment but are not withdrawn from study (i.e., still in follow-up). Early termination from study represents subjects who did not complete study visits or complete the Double-blind treatment period.

SOURCE: Listing 16.2.1





# Table 14.1.1.1 (cont.) Summary of Subject Disposition ITT Population

| | Trifarotene cream HE1 | Trifarotene cream HE1 | | |
|---|---|---|---|---|
| | 100 ug/g | 200 ug/g | Vehicle | Overall |
| Category | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) |
| Early Termination from Study | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Reason for Early Termnation: | , | , | , | , , |
| Adverse Event | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Intercurrent Illness | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Death | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Lack of Efficacy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Lost to Follow-up | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Non-compliance with Study Procedures | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Administrative Reasons | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Physician Decision | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Pregnancy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Protocol Violation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Subject Meets an Exclusion Criteria | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Withdrawal by Subject | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Subject Withdrew Consent | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Terminated by Sponsor | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Other | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Blind Broken | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

Abbreviations: ITT = intent-to-treat; mITT = modified intent-to-treat; OLE = open label extension; PK = pharmacokinetic; PP = per protocol.

Note: Percentages are n/Number of subjects in the ITT Population within randomized treatment group and overall\*100. The ITT population includes all randomized subjects. The Safety population includes all subjects who are randomized to treatment and receive at least 1 application of study drug in the Double-blind Period. The mITT population includes all subjects in the Safety population with at least 1 postbaseline assessment of efficacy in the Double-blind period. The PP population includes all subjects in the mITT population who met all inclusion criteria and no exclusion criteria, were compliant with study drug application, and who had no significant protocol deviations. The PK population includes all subjects in the Safety population who have at least 1 plasma sample with quantifiable concentration. Completed continuing represents subjects who completed study visits and Double-blind treatment period (Day 90) and are continuing to OLE. Completed not continuing represents subjects who completed study visits and Double-blind treatment period (Day 90) but are not continuing to OLE. Early discontinuation of medication represent subjects who did not complete treatment but are not withdrawn from study (i.e., still in follow-up). Early termination from study represents subjects who did not complete study visits or complete the Double-blind treatment period.

SOURCE: Listing 16.2.1

**Programming note:** Only include the Ongoing in Double-blind Study row when the overall n>0 for that row (i.e. dry runs).





#### Table 14.1.1.2 Summary of Subject Disposition OLE ITT Population

| | Trifarotene cream HE1 |
|--------------------------------------|-----------------------|
| | 200 ug/g |
| Category | (N=XXX) |
| OLE ITT Population | XX (XX.X%) |
| OLE Safety Population | XX (XX.X%) |
| OLE mITT Population | XX (XX.X%) |
| OLE PP Population | XX (XX.X%) |
| Completed | XX (XX.X%) |
| Ongoing in OLE Study | XX (XX.X%) |
| Early Discontinuation of Medication | XX (XX.X%) |
| Early Termination from Study | XX (XX.X%) |
| Reason for Early Termnation: | , |
| Adverse Event | XX (XX.X%) |
| Intercurrent Illness | XX (XX.X%) |
| Death | XX (XX.X%) |
| Lack of Efficacy | XX (XX.X%) |
| Lost to Follow-up | XX (XX.X%) |
| Non-compliance with Study Procedures | XX (XX.X%) |
| Administrative Reasons | XX (XX.X%) |
| Physician Decision | XX (XX.X%) |
| Pregnancy | XX (XX.X%) |
| Protocol Violation | XX (XX.X%) |
| Subject Meets an Exclusion Criteria | XX (XX.X%) |
| Withdrawal by Subject | XX (XX.X%) |
| Subject Withdrew Consent | XX (XX.X%) |
| Study Terminated by Sponsor | XX (XX.X%) |
| Other | XX (XX.X%) |

Abbreviations: EOT = end of treatment; ITT = intent-to-treat; mITT = modified intent-to-treat; OLE = open label extension; PP = per protocol.

Note: Percentages are n/Number of subjects in the OLE ITT Population within treatment group and overall\*100. All subjects received Trifarotene cream HE1 200 ug/g in the OLE. The OLE ITT population includes all subjects who complete the 90-day Double-blind treatment Period and sign the OLE informed consent. The OLE Safety population includes all subjects who complete the 90-day Double-blind treatment Period and receive at least 1 application of study drug in the OLE. The OLE mITT population includes all subjects in the Safety population with at least 1 assessment of efficacy in after Visit 6 (Day 90). The OLE PP population includes all subjects in the OLE mITT population who met all inclusion criteria and no exclusion criteria, were compliant with study drug application from baseline through EOT, and who had no significant protocol deviations throughout the study. Completed continuing represents subjects who completed study visits and OLE treatment period. Early discontinuation of medication represent subjects who did not complete treatment but are not withdrawn from study (i.e., still in follow-up). Early termination from study represents subjects who did not complete the OLE treatment period.

SOURCE: Listing 16.2.1

AD-ST-33.05 Effective date: 22-Jan-2018





Table 14.1.2.1 Summary of Demographics and Baseline Characteristics ITT Population

| | Trifarotene cream HE1 | Trifarotene cream HE1 | | |
|---|---|---|---|---|
| Variable | 100 ug/g | 200 ug/g | Vehicle | Overall |
| Statistic or Category | (N=XX) | (N=XX) | (N=XX) | (N=XX) |
| Age (years) | | | | |
| n | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX | XX, XX |
| | | • | · | • |
| Sex | | | | |
| Male | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Female | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Child-bearing Age? [1] | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Ethnicity [2] | | | | |
| Hispanic or Latino | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Not Hispanic or Latino | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Not Applicable | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| •• | , | , | , | , |
| Race [2] | | | | |
| American-Indian or Alaska Native | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Asian | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Black or African-American | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Native Hawaiian or Other Pacific Islander | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| White | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| More than One Race | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Race not Provided | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

Abbreviations: IGA = Investigator's Global Assessment; SD = standard deviation.

Note: Percentages are n/Number of subjects in the ITT Population within randomized treatment group and overall\*100.

SOURCE: Listings 16.2.4.1, 16.2.6.1

<sup>[1]</sup> Only captured for female subjects; percentages are based on the number of female subjects in the Safety Population.

<sup>[2]</sup> Not captured in France.





# Table 14.1.2.1(cont.) Summary of Demographics and Baseline Characteristics ITT Population

| Variable<br>Statistic or Category | Trifarotene cream HE1<br>100 ug/g<br>(N=XX) | Trifarotene cream HE1<br>200 ug/g<br>(N=XX) | Vehicle<br>(N=XX) | Overall<br>(N=XX) |
|---|---|---|---|---|
| Height (cm) | | | | |
| n | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX | XX, XX |
| Weight (kg) | | | | |
| n n | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | xx.x | xx.x | xx.x | xx.x |
| Min, Max | XX, XX | XX, XX | XX, XX | XX, XX |
| Body Mass Index (kg/m²) | | | | |
| n ( ) | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | xx.x | xx.x | xx.x | xx.x |
| Min, Max | XX, XX | XX, XX | XX, XX | XX, XX |
| GA Score | | | | |
| n | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | xx.x | xx.x | xx.x | xx.x |
| Min, Max | XX, XX | XX, XX | XX, XX | XX, XX |

Abbreviations: IGA = Investigator's Global Assessment; SD = standard deviation.

Note: Percentages are n/Number of subjects in the ITT Population within randomized treatment group and overall\*100.

SOURCE: Listings 16.2.4.1, 16.2.6.1

<sup>[1]</sup> Only captured for female subjects; percentages are based on the number of female subjects in the Safety Population.

<sup>[2]</sup> Not captured in France.





# Table 14.1.2.2 Summary of Demographics and Baseline Characteristics OLE ITT Population

#### Same shell as Table 14.1.2.1

Programming note: Only include one column for Trifarotene cream HE1 200 ug/g.

Update Note: to read "Percentages are n/Number of subjects in the OLE ITT Population within treatment group and overall\*100. All subjects received Trifarotene cream HE1 200 ug/g in the OLE."

Add OLE = open label extension to Abbreviations.





Table 14.1.3 Summary of Medical Histories by System Organ Class and Preferred Term Safety Population

| System Organ Class<br>Preferred Term | Trifarotene cream HE1<br>100 ug/g<br>(N=XX) | Trifarotene cream HE1<br>200 ug/g<br>(N=XX) | Vehicle<br>(N=XX) | Overall<br>(N=XX) |
|---|---|---|---|---|
| Subjects with at least 1 Recorded Medical History | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| System Organ Class 1 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Preferred Term 1 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Preferred Term 2 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Preferred Term 3 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| System Organ Class 2 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Preferred Term 1 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Preferred Term 2 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Preferred Term 3 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

Abbreviation: MedDRA = Medical Dictionary for Regulatory Activities; PT = preferred term; SOC = system organ class.

Note: Percentages are n/Number of subjects in the Safety population within actual treatment group and overall\*100. Medical histories are coded using MedDRA version 21.1. Subjects were counted once for each system organ class (SOC) and once for each preferred term (PT). Medical history terms are displayed by descending frequency of SOC, then PT within SOC, and then alphabetically by PT.

SOURCE: Listing 16.2.4.3

Programming note: SOC & PT text should be in title case in table, as shown in the shell.





Table 14.1.4 Summary of Prior Medications by ATC Class Level 4 and Preferred Term Safety Population

| ATC Class Level 4<br>Preferred Term (ATC Class Level 5) | Trifarotene cream HE1<br>100 ug/g<br>(N=XX) | Trifarotene cream HE1<br>200 ug/g<br>(N=XX) | Vehicle<br>(N=XX) | Overall<br>(N=XX) |
|---|---|---|---|---|
| Subjects with at least 1 Prior Medication | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| ATC Class 1 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Preferred Term 1 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Preferred Term 2 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Preferred Term 3 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| ATC Class 2 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Preferred Term 1 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Preferred Term 2 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Preferred Term 3 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

Abbreviations: ATC = Anatomic Therapeutic Chemical; PT = preferred term; WHO-DDE = World Health Organization-Drug Dictionary Enhanced.

Note: Percentages are n/Number of subjects in the Safety population within actual treatment group and overall\*100. Medications were coded using WHO-DDE version March 2019.

Prior medications are all medications that were started before the first dose of study drug. Medications are displayed by descending frequency of ATC Level 4 classification, by PT within ATC, and then alphabetically by PT, based on the overall column. Subjects were counted only once for each ATC and PT.

SOURCE: Listing 16.2.9.5

Programming note: ATC & PT text should be in title case in table, as shown in the shell.





#### Table 14.1.5.1 Summary of Drug Accountability (Drug Returned and Dispensed) Safety Population

| Visit | Trifarotene cream HE1 | Trifarotene cream HE1 | | |
|---|---|---|---|---|
| Parameter | 100 ug/g | 200 ug/g | Vehicle | Overall |
| Statistic | (N=XX) | (N=XX) | (N=XX) | (N=XX) |
| Baseline [1] | | | | |
| Total Weight of Tubes Dispensed (g) | | | | |
| n | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | xx.x | xx.x | xx.x | XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX | XX, XX |
| Day 14 | | | | |
| Total Weight of Tubes Dispensed (g) | | | | |
| n | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | xx.x | xx.x | xx.x |
| Min, Max | XX, XX | XX, XX | XX, XX | XX, XX |
| Total Number of Tubes Returned | | | | |
| n | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | xx.x | xx.x | xx.x | xx.x |
| Min, Max | XX, XX | XX, XX | XX, XX | XX, XX |

Abbreviation: OLE = open label extension. SD = standard deviation.

Note: Subjects are summarized by actual treatment group. Subjects were randomized to either Trifarotene cream HE1 100 ug/g, Trifarotene cream HE1 200 ug/g, or vehicle in the Double-blind period. All subjects received Trifarotene cream HE1 200 ug/g in the OLE.

[1] Baseline is defined as the last non-missing assessment recorded prior to the first dose of treatment in the Double-blind Period.

SOURCE: Listings 16.2.5.1, 16.2.5.2, 16.2.5.3





# Table 14.1.5.1 (cont.) Summary of Drug Accountability (Drug Returned and Dispensed) Safety Population

| Visit | Trifarotene cream HE1 | Trifarotene cream HE1 | | |
|---|---|---|---|---|
| Parameter | 100 ug/g | 200 ug/g | Vehicle | Overall |
| Statistic | (N=XX) | (N=XX) | (N=XX) | (N=XX) |
| Day 14 | | | | |
| Total Number of Tubes Returned Unused | | | | |
| n | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX | XX, XX |
| Total Weight of Tubes Returned (g) | | | | |
| n | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | xx.x | xx.x | xx.x | XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX | XX, XX |

Abbreviation: OLE = open label extension. SD = standard deviation.

Note: Subjects are summarized by actual treatment group. Subjects were randomized to either Trifarotene cream HE1 100 ug/g, Trifarotene cream HE1 200 ug/g, or vehicle in the Double-blind period. All subjects received Trifarotene cream HE1 200 ug/g in the OLE.

SOURCE: Listings 16.2.5.1, 16.2.5.2, 16.2.5.3

Programming note: Continue for Day 30, Day 60, and Day 90.





#### Table 14.1.5.2 Summary of Drug Accountability (Drug Returned and Dispensed) OLE Safety Population

#### Same shell as Table 14.1.5.1

Programming note: Only include one column for Trifarotene cream HE1 200 ug/g.

Continue for Day 104, Day 120, Day 150 and Day 180.

Update Note: to read "Note: Subjects are summarized by treatment group. All subjects received Trifarotene cream HE1 200 ug/g in the OLE."

AD-ST-33.05 Effective date: 22-Jan-2018





# Table 14.1.5.3 Summary of Treatment Exposure and Compliance Safety Population

| Variable<br>Statistic or Category | Trifarotene cream HE1<br>100 ug/g<br>(N=XX) | Trifarotene cream HE1<br>200 ug/g<br>(N=XX) | Vehicle<br>(N=XX) | Overall<br>(N=XX) |
|---|---|---|---|---|
| Statistic of Category | (N-XX) | (14->>>) | (N-XX) | (14-7/ |
| Compliance by Tube Weight (%) [1] | | | | |
| n | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | XX.X | XX.X |
| | XX. XX | | XX, XX | XX, XX |
| Min, Max | *** | XX, XX | ***, *** | <b>^^</b> , <b>^^</b> |
| Compliant | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| lot Compliant | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Compliance by Number of Doses (%) [2] | | | | |
| n | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | xx.x | xx.x | xx.x | xx.x |
| Min, Max | XX, XX | XX, XX | XX, XX | XX, XX |
| Timi, Ties | 704,704 | 701,701 | 701,701 | 701, 701 |
| Compliant | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Not Compliant | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

Abbreviation: SD = standard deviation.

Note: Percentages are n/Number of subjects in the Safety population within actual treatment group and overall\*100. A subject is compliant with study product if he or she takes at least 80%-120% of the scheduled doses as assessed by diary entries, supplemented by tube weight.

SOURCE: Listings 16.2.5.1, 16.2.5.2, 16.2.5.3

<sup>[1]</sup> Compliance by tube weight = total weight used / total weight of tubes dispensed \*100%, where total weight used = total weight of tubes dispensed (grams) – total weight of tubes returned (grams)

<sup>[2]</sup> Compliance by number of doses = number of doses taken / number of expected doses \* 100%, where number of doses taken = total number of tubes dispensed – total number of tubes returned – total number of tubes returned – total number of tubes returned unused, number of expected doses = 2 \* number of weeks on study, and number of weeks on study = (last day on study – treatment start date + 1) / 7





# Table 14.1.5.4 Summary of Treatment Exposure and Compliance OLE Safety Population

#### Same shell as Table 14.1.5.3

Programming note: Only include one column for Trifarotene cream HE1 200 ug/g.

Update Note: to read "Note: Percentages are n/Number of subjects in the OLE Safety population within treatment group and overall\*100. All subjects received Trifarotene cream HE1 200 ug/g in the OLE."

Add OLE = open label extension to Abbreviations.

AD-ST-33.05 Effective date: 22-Jan-2018





Table 14.2.1.1.1

Primary Analysis: Logistic Regression Analysis of Successful Resolution of LI
ITT Population

| Study Visit<br>Statistic | Trifarotene cream HE1<br>100 ug/g<br>(N = XX) | Trifarotene cream HE1<br>200 ug/g<br>(N = XX) | Overall Trifarotene<br>cream HE1<br>(N = XX) | Vehicle<br>(N = XX) |
|---|---|---|---|---|
| Day 90 | | | | |
| n [1] | XX | XX | XX | XX |
| Successful Resolution [2] | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Odds Ratio (Trifarotene cream HE1 vs Vehicle) | X.XX | X.XX | X.XX | |
| 95% CI for Odds Ratio | (X.XX, X.XX) | (X.XX, X.XX) | (X.XX, X.XX) | |
| P value [3] | X.XXX | X.XXX | X.XXX | |
| Difference in Proportion (Trifarotene cream HE1 vs Vehicle) | X.XX | X.XX | X.XX | |
| 95% CI for Proportion Difference | (X.XX, X.XX) | (X.XX, X.XX) | (X.XX, X.XX) | |
| P value [3] | ` x.xxx ´ | ` x.xxx ´ | ` x.xxx | |

Abbreviation: CI = confidence interval; EOT = end of treatment; IGA = Investigator's Global Assessment; ITT = intent to treat; LI = Lamellar Ichthyosis; OR = odds ratio. Note: Percentages are n/Number of subjects in the ITT population within randomized treatment group\*100. The 5-point (0 - 4) IGA is a measure of disease severity which considers both scaling and roughness. Higher IGA scores represent more severe disease.

[1] Number of subjects with an IGA assessment at each visit.

[2] Number of subjects with successful resolution of LI at a visit. Successful resolution is defined as clear/almost clear overall (IGA of 0 or 1, respectively) and at least a 2grade change from Baseline on the

5-point (0 - 4) IGA scale. Baseline is defined as the last non-missing assessment recorded prior to the first dose of treatment in the Double-blind Period.

[3] Estimates for odds ratio, 95% CI for odds ratio, and P value are from a logistic regression model with treatment, baseline IGA score, and age group as factors. The odds ratio is the estimate of the odds of having successful resolution of LI for subjects treated with Trifarotene cream HE1 relative to that for subjects treated with vehicle. Age group is defined as adolescents (ages 12 to 17 years, inclusive) and adults ≥18 years.

SOURCE: Listing 16.2.6.1

Programming note: If Firth's penalized maximum likelihood is used, add 'Firth's penalized maximum likelihood estimation is used.' to end of 'Note:' footnote. If the treatment-by-age interaction is significant, include it in the logistic regression model and update footnote [3] to include this factor. After Day 90, repeat table for Days 14, 30, and 60.





# Table 14.2.1.1.2 Proportion of Subjects with Successful Resolution of LI in the OLE OLE ITT Population

| Study Visit<br>Statistic | Trifarotene cream HE1<br>200 ug/g<br>(N = XX) |
|---|---|
| Day 104<br>n [1]<br>Successful Resolution [2] | XX<br>XX (XX.X%) |
| Day 120<br>n [1]<br>Successful Resolution [2] | XX<br>XX (XX.X%) |
| Day 150<br>n [1]<br>Successful Resolution [2] | XX<br>XX (XX.X%) |
| Day 180<br>n [1]<br>Successful Resolution [2] | XX<br>XX (XX.X%) |
| Day 194<br>n [1]<br>Successful Resolution [2] | XX<br>XX (XX.X%) |

Abbreviation: CI = confidence interval; EOT = end of treatment; IGA = Investigator's Global Assessment; ITT = intent to treat; LI = Lamellar Ichthyosis; OLE = open label extension. Note: Percentages are n/Number of subjects in the OLE ITT population within treatment group\*100. All subjects received Trifarotene cream HE1 200 ug/g in the OLE. The 5-point (0 - 4) IGA is a measure of disease severity which considers both scaling and roughness. Higher IGA scores represent more severe disease.

[1] Number of subjects with an IGA assessment at each visit.

[2] Number of subjects with successful resolution of LI at a visit. Successful resolution is defined as clear/almost clear overall (IGA of 0 or 1, respectively) and at least a 2-grade change from Baseline on the 5-point (0 - 4) IGA scale. Baseline is defined as the last non-missing assessment recorded prior to the first dose of treatment in the Double-blind Period.

SOURCE: Listing 16.2.6.1





# Table 14.2.1.2.1 Primary Analysis, Sensitivity: Logistic Regression Analysis of Successful Resolution of LI mITT Population

#### Same shell as Table 14.2.1.1.1

**Programming note:** Update Abbreviations to remove ITT and include mITT = modified intent-to-treat.

Update Note: to read "Note: Percentages are n/Number of subjects in the mITT population within randomized treatment group\*100."

Table 14.2.1.2.2
Proportion of Subjects with Successful Resolution of LI in the OLE
OLE mITT Population

#### Same shell as Table 14.2.1.1.2

Programming note: Update Abbreviations to remove ITT and include mITT = modified intent-to-treat and OLE = open label extension.

Update Note: to read "Note: Percentages are n/Number of subjects in the OLE mITT population within treatment group\*100. All subjects received Trifarotene cream HE1 200 ug/g in the OLE."

Table 14.2.1.3.1

Primary Analysis, Sensitivity: Logistic Regression Analysis of Successful Resolution of LI
PP Population

#### Same shell as Table 14.2.1.1.1

**Programming note:** Update Abbreviations to remove ITT and include PP = per protocol.

Update Note: to read "Note: Percentages are n/Number of subjects in the PP population within actual treatment group\*100."

Table 14.2.1.3.2
Proportion of Subjects with Successful Resolution of LI in the OLE OLE PP Population

#### Same shell as Table 14.2.1.1.2

Programming note: Update Abbreviations to remove ITT and include OLE = open label extension and PP = per protocol.

Update Note: to read "Note: Percentages are n/Number of subjects in the OLE PP population within treatment group\*100. All subjects received Trifarotene cream HE1 200 ug/g in the OLE."

AD-ST-33.05 Effective date: 22-Jan-2018





Table 14.2.1.4
Primary Analysis, Sensitivity: Logistic Regression Analysis of Successful Resolution of LI Using Multiple Imputation
ITT Population

#### Same shell as Table 14.2.1.1.1

Programming note: Update footnote [3] to read "Estimates for odds ratio, 95% CI for odds ratio, and P value are from a logistic regression model with treatment, baseline IGA score, and age group as factors. The odds ratio is the estimate of the odds of having successful resolution of LI for subjects treated with Trifarotene cream HE1 relative to that for subjects treated with vehicle. Missing values were considered MNAR and imputed using MI with a placebo-based pattern mixture model and then categorized as treatment success. Age group is defined as adolescents (ages 12 to 17 years, inclusive) and adults ≥18 years."

Table 14.2.1.5.1
Logistic Regression Analysis of 50% Reduction in IGA score from Baseline
ITT Population

#### Same shell as Table 14.2.1.1.1

Programming note: Update "Successful Resolution [2]" row text to read "50% Reduction from Baseline [2]".

Update footnote [2] to read "Number of subjects with a 50% reduction in IGA score from baseline at a visit. Baseline is defined as the last non-missing assessment recorded prior to the first dose of treatment in the Double-blind Period. Higher IGA scores represent more severe disease."

Update [3] to read "Estimates for odds ratio, 95% CI for odds ratio, and P value are from a logistic regression model with treatment, baseline IGA score, and age group as factors. The odds ratio is the estimate of the odds of having a 50% reduction in IGA score from baseline for subjects treated with Trifarotene cream HE1 relative to that for subjects treated with vehicle. Age group is defined as adolescents (ages 12 to 17 years, inclusive) and adults ≥18 years."

Table 14.2.1.5.2
Proportion of Subjects with a 50% Reduction in IGA score from Baseline
OLE ITT Population

#### Same shell as Table 14.2.1.1.2

Programming note: Update "Successful Resolution [2]" row text to read "50% Reduction from Baseline [2]".

Update Note: to read "Note: Percentages are n/Number of subjects in the OLE ITT population within treatment group\*100. All subjects received Trifarotene cream HE1 200 ug/g in the

Update footnote [2] to read "Number of subjects with a 50% reduction in IGA score from baseline at a visit. Baseline is defined as the last non-missing assessment recorded prior to the first dose of treatment in the Double-blind Period. Higher IGA scores represent more severe disease."

AD-ST-33.05 Effective date: 22-Jan-2018





#### Table 14.2.1.6.1 MMRM Analysis of Change from Baseline in IGA Score **ITT Population**

| Study Visit | 100 | tene cream HE1 Trifarotene cream H<br>100 ug/g 200 ug/g<br>(N=XXX) (N=XXX) | | ug/g |
|---|---|---|---|---|
| Statistic [1] | Observed | CFB | Observed | CFB |
| Baseline [2] | | | | |
| n | XXX | | XXX | |
| Mean (SD) | XX.XX (XX.XXX) | | XX.XX (XX.XXX) | |
| Median | XX.XX | | xx.xx | |
| Min, Max | XX.X, XX.X | | XX.X, XX.X | |
| Day 14 | | | | |
| n | XXX | XXX | XXX | XXX |
| Mean (SD) | XX.XX (XX.XXX) | XX.XX (XX.XXX) | XX.XX (XX.XXX) | XX.XX (XX.XXX) |
| Median | XX.XX | XX.XX | XX.XX | XX.XX |
| Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| LS Mean (SE) CFB | | X.XX (X.XXX) | | X.XX (X.XXX) |
| 95% CI for LS Mean CFB | | (X.XX, X.XX) | | (X.XX, X.XX) |
| P value for CFB = 0 | | ` X.XXXX | | ` X.XXXX |
| Comparison vs. Vehicle | | | | |
| Difference in LS Mean (SE) | | X.XX (X.XXX) | | X.XX (X.XXX) |
| 95% CI for Difference in LS Mean | | (X.XX, X.XX) | | (X.XX, X.XX) |
| P value for Difference | | `x.xxxx ´ | | ` X.XXXX |

Abbreviations: CFB = change from baseline; CI = confidence interval; IGA = Investigator's Global Assessment; ITT = intent to treat; LS = least-squares; MMRM = mixed model for repeated measures; SD = standard deviation; SE = standard error.

Note: Subjects are summarized by randomized treatment group. The 5-point (0 - 4) IGA is a measure of disease severity which considers both scaling and roughness. Higher IGA scores represent more severe disease.

[1] LS mean CFB, LS mean differences (Trifarotene cream HE1 - vehicle), 95% Cls, and P values were obtained from a mixed model for repeated measures (MMRM) with change from baseline in IGA score as the repeated dependent variable, fixed effect terms for baseline IGA score, treatment, study visit, treatment-by-study visit interaction, and age group as independent variables. An unstructured covariance matrix was used to model the within-subject correlation. Age group is defined as adolescents (ages 12 to 17 years, inclusive) and adults ≥18 years.

[2] Baseline is defined as the last non-missing assessment recorded prior to the first dose of treatment in the Double-blind Period.

SOURCE: Listing 16.2.6.1

Programming note: If the unstructured covariance structure does not converge, use other structures as outlined in the SAP section 8.1 and update the footnote accordingly. Include Days 30, 60, and 90 as well. Rows will be the same as what is displayed for Day 14. Repeat Table for Overall Trifarotene cream HE1 and Vehicle columns. Vehicle column will not have Comparison vs. Vehicle row cells populated.





#### Table 14.2.1.6.2 MMRM Analysis of Change from Baseline in IGA Score OLE ITT Population

**Programming note:** Update Note: to read "Subjects are summarized by treatment group. All subjects received Trifarotene cream HE1 200 ug/g in the OLE."

Only include one set of columns for Trifarotene cream HE1 200 ug/g.

Do not include Comparison vs. Vehicle rows.

Baseline [2], Days 104, 120, 150, 180, and 194 will be displayed.

Update footnote [1] to read "LS mean CFB, 95% CIs, and P values were obtained from a mixed model for repeated measures (MMRM) with change from baseline in IGA score as the repeated dependent variable, fixed effect terms for baseline IGA score, study visit, and age group as independent variables. An unstructured covariance matrix was used to model the within-subject correlation. Age group is defined as adolescents (ages 12 to 17 years, inclusive) and adults ≥18 years."





#### Table 14.2.7.1.1 Categorical IGA Scores ITT Population

| Study Visit<br>Category | Trifarotene<br>cream HE1<br>100 ug/g<br>(N=XX) | Trifarotene<br>cream HE1<br>200 ug/g<br>(N=XX) | Overall<br>Trifarotene<br>cream HE1<br>(N=XX) | Vehicle<br>(N=XXX) |
|---|---|---|---|---|
| Baseline [1] | | | | |
| 0 = Clear | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 1 = Almost clear | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 2 = Mild | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 3 = Moderate | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 4 = Severe | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Day 14 | | | | |
| 0 = Clear | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 1 = Almost clear | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 2 = Mild | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 3 = Moderate | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 4 = Severe | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Day 90 | | | | |
| 0 = Clear | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 1 = Almost clear | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 2 = Mild | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 3 = Moderate | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 4 = Severe | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

Abbreviations: IGA = Investigator's Global Assessment; ITT = intent to treat;

Note: Percentages are n/Number of subjects in the ITT population within randomized treatment group\*100. The 5-point (0 - 4) IGA is a measure of disease severity which considers both scaling and roughness. Higher IGA scores represent more severe disease.

[1] Baseline is defined as the last non-missing assessment recorded prior to the first dose of treatment in the Double-blind Period.

SOURCE: Listing 16.2.6.1




Table 14.2.1.7.2 Categorical IGA Scores OLE ITT Population

Programming note: Update Note: to read "Percentages are n/Number of subjects in the OLE ITT population within treatment group\*100. All subjects received Trifarotene cream HE1 200 ug/g in the OLE."

Only include one set of columns for Trifarotene cream HE1 200 ug/g.

Baseline [2], Days 104, 120, 150, 180, and 194 will be displayed.

Add OLE = open label extension to Abbreviations.

Table 14.2.2.1
Secondary Analysis: MMRM Analysis of Change from Baseline in VIIS Score ITT Population

## Same shell as Table 14.2.1.6.1

**Programming note:** Update Note: to read "Note: Subjects are summarized by randomized treatment group. The VIIS is scored on a 5-point (0 - 4) scale by body area (chest/abdomen, back, legs, and arms). Higher VIIS scores represent worse scaling."

Update [1] to read "LS mean CFB, LS mean differences (Trifarotene cream HE1 - vehicle), 95% CIs, and P values were obtained from a mixed model for repeated measures (MMRM) with change from baseline in VIIS score as the repeated dependent variable, fixed effect terms for baseline VIIS score, treatment, study visit, treatment-by-study visit interaction, and age group as independent variables. An unstructured covariance matrix was used to model the within-subject correlation. Age group is defined as adolescents (ages 12 to 17 years, inclusive) and adults ≥18 years."

Remove IGA and add VIIS= Visual Index for Ichthyosis Severity to Abbreviations.

Update SOURCE: to Listing 16.2.6.2

Table 14.2.2.2

MMRM Analysis of Change from Baseline in VIIS Score
OLE ITT Population

#### Same shell as Table 14.2.2.1

Update Note: to read "Subjects are summarized by treatment group. All subjects received Trifarotene cream HE1 200 ug/g in the OLE."

Only include one set of columns for Trifarotene cream HE1 200 ug/g.

Do not include Comparison vs. Vehicle rows.

Baseline [2], Davs 104, 120, 150, 180, and 194 will be displayed.

Update footnote [1] to read "LS mean CFB, 95% CIs, and P values were obtained from a mixed model for repeated measures (MMRM) with change from baseline in IGA score as the repeated dependent variable, fixed effect terms for baseline IGA score, study visit, and age group as independent variables. An unstructured covariance matrix was used to model the within-subject correlation. Age group is defined as adolescents (ages 12 to 17 years, inclusive) and adults ≥18 years."

Update SOURCE: to Listing 16.2.6.2





## Table 14.2.3.1

Secondary Analysis: MMRM Analysis of Change from Baseline in Individual Score for Roughness ITT Population

#### Same shell as Table 14.2.1.6.1

**Programming note:** Update Note: to read "Note: Subjects are summarized by randomized treatment group. The individual score for roughness measures the amount of roughness of the skin overall and is scored on a 5-point (0 - 4) scale. Higher scores indicate more severe roughness."

Update footnote [1] to read "LS mean CFB, LS mean differences (Trifarotene cream HE1 - vehicle), 95% CIs, and P values were obtained from a mixed model for repeated measures (MMRM) with change from baseline in individual score for roughness as the repeated dependent variable, fixed effect terms for baseline individual score for roughness, treatment, study visit, treatment-by-study visit interaction, and age group as independent variables. An unstructured covariance matrix was used to model the within-subject correlation.
[2] Baseline is defined as the last non-missing assessment recorded prior to the first dose of treatment in the Double-blind Period. Age group is defined as adolescents (ages 12 to 17 years, inclusive) and adults ≥18 years."

Update SOURCE: to Listing 16.2.6.3

# Table 14.2.3.2 MMRM Analysis of Change from Baseline in Individual Score for Roughness OLE ITT Population

#### Same shell as Table 14.2.1.6.1

Update Note: to read "Subjects are summarized by treatment group. All subjects received Trifarotene cream HE1 200 ug/g in the OLE. The individual score for roughness measures the amount of roughness of the skin overall and is scored on a 5-point (0 - 4) scale. Higher scores indicate more severe roughness."

Only include one set of columns for Trifarotene cream HE1 200 ug/g.

Do not include Comparison vs. Vehicle rows.

Baseline [2], Days 104, 120, 150, 180, and 194 will be displayed.

Update footnote [1] to read "LS mean CFB, 95% CIs, and P values were obtained from a mixed model for repeated measures (MMRM) with change from baseline in individual score for roughness as the repeated dependent variable, fixed effect terms for baseline individual score for roughness, study visit, and age group as independent variables. An unstructured covariance matrix was used to model the within-subject correlation. Age group is defined as adolescents (ages 12 to 17 years, inclusive) and adults ≥18 years."

Update SOURCE: to Listing 16.2.6.3

### Table 14.2.3.3

Logistic Regression Analysis of 2-grade Change in Individual Score for Roughness from Baseline ITT Population

## Same shell as Table 14.2.1.1.1

Programming note: Update "Successful Resolution [2]" row text to read "2-grade Change from Baseline [2]".

Update Note: to read "Note: Percentages are n/Number of subjects in the ITT population within randomized treatment group\*100. The individual score for roughness measures the amount of roughness of the skin overall and is scored on a 5-point (0 - 4) scale. Higher scores indicate more severe roughness."

Update footnote [2] to read "Number of subjects with a 2-grade change in individual score for roughness from baseline at a visit. Baseline is defined as the last non-missing assessment recorded prior to the first dose of treatment in the Double-blind Period. Higher scores indicate more severe roughness."

Update [3] to read "Estimates for odds ratio, 95% CI for odds ratio, and P value are from a logistic regression model with treatment, baseline individual score for roughness, and age group as factors. The odds ratio is the estimate of the odds of having a 2-grade change in individual score for roughness from baseline for subjects treated with Trifarotene cream HE1 relative to that for subjects treated with vehicle. Age group is defined as adolescents (ages 12 to 17 years, inclusive) and adults ≥18 years."

Update SOURCE: to Listing 16.2.6.3





# Table 14.2.4.1 Secondary Analysis: MMRM Analysis of Change from Baseline in Palm/Sole Assessment ITT Population

### Same shell as Table 14.2.1.6.1

**Programming note:** Update Note: to read "Note: Subjects are summarized by randomized treatment group. Thickening of the skin on the palms and soles will be measured on a 5-point (0 - 4) scale. Higher scores indicate more severe thickening."

Update footnote [1] to read "LS mean CFB, LS mean differences (Trifarotene cream HE1 - vehicle), 95% CIs, and P values were obtained from a mixed model for repeated measures (MMRM) with change from baseline in palm/sole assessment score as the repeated dependent variable, fixed effect terms for baseline palm/sole assessment score, treatment, study visit, treatment-by-study visit interaction, and age group as independent variables. An unstructured covariance matrix was used to model the within-subject correlation.

[2] Baseline is defined as the last non-missing assessment recorded prior to the first dose of treatment in the Double-blind Period. Age group is defined as adolescents (ages 12 to 17

years, inclusive) and adults ≥18 years."

Update SOURCE: to Listing 16.2.6.4

Table 14.2.4.2

MMRM Analysis of Change from Baseline in Palm/Sole Assessment
OLE ITT Population

## Same shell as Table 14.2.1.6.1

Update Note: to read "Subjects are summarized by treatment group. All subjects received Trifarotene cream HE1 200 ug/g in the OLE. Thickening of the skin on the palms and soles will be measured on a 5-point (0 - 4) scale. Higher scores indicate more severe thickening."

Only include one set of columns for Trifarotene cream HE1 200 ug/g.

Do not include Comparison vs. Vehicle rows.

Baseline [2], Days 104, 120, 150, 180, and 194 will be displayed.

Update footnote [1] to read "LS mean CFB, 95% CIs, and P values were obtained from a mixed model for repeated measures (MMRM) with change from baseline in palm/sole assessment score as the repeated dependent variable, fixed effect terms for baseline palm/sole assessment score, study visit, and age group as independent variables. An unstructured covariance matrix was used to model the within-subject correlation. Age group is defined as adolescents (ages 12 to 17 years, inclusive) and adults ≥18 years."

Update SOURCE: to Listing 16.2.6.4





# Table 14.2.4.3 Logistic Regression Analysis of 2-grade Change in Palm/Sole Assessment from Baseline ITT Population

### Same shell as Table 14.2.1.1.1

Programming note: Update "Successful Resolution [2]" row text to read "2-grade Change from Baseline [2]".

Update Note: to read "Note: Percentages are n/Number of subjects in the ITT population within randomized treatment group\*100. Thickening of the skin on the palms and soles will be measured on a 5-point (0 - 4) scale. Higher scores indicate more severe thickening."

Update footnote [2] to read "Number of subjects with a 2-grade change in palm/sole assessment score from baseline at a visit. Baseline is defined as the last non-missing assessment recorded prior to the first dose of treatment in the Double-blind Period. Higher scores indicate more severe roughness."

Update [3] to read "Estimates for odds ratio, 95% CI for odds ratio, and P value are from a logistic regression model with treatment, baseline palm/sole assessment score, and age group as factors. The odds ratio is the estimate of the odds of having a 2-grade change in palm/sole assessment score from baseline for subjects treated with Trifarotene cream HE1 relative to that for subjects treated with vehicle. Age group is defined as adolescents (ages 12 to 17 years, inclusive) and adults ≥18 years."

Update SOURCE: to Listing 16.2.6.4





Table 14.2.5.1
Secondary Analysis: MMRM Analysis of Change from Baseline in Dermatology Life Quality Index ITT Population

#### Same shell as Table 14.2.1.6.1

**Programming note:** Update Note: to read "Note: Subjects are summarized by randomized treatment group. DLQI total score is derived as the sum of the 10 individual item scores, with a range of 0 to 30. Higher scores indicate poorer quality of life."

Update footnote [1] to read "LS mean CFB, LS mean differences (Trifarotene cream HE1 - vehicle), 95% CIs, and P values were obtained from a mixed model for repeated measures (MMRM) with change from baseline in DLQI score as the repeated dependent variable, fixed effect terms for baseline DLQI score, treatment, study visit, and treatment-by-study visit interaction as independent variables. An unstructured covariance matrix was used to model the within-subject correlation.

[2] Baseline is defined as the last non-missing assessment recorded prior to the first dose of treatment in the Double-blind Period."

Update SOURCE: to Listing 16.2.6.5.1

Table 14.2.5.2
Secondary Analysis: MMRM Analysis of Change from Baseline in Children's Dermatology Life Quality Index ITT Population

#### Same shell as Table 14.2.1.6.1

**Programming note:** Update Note: to read "Note: Subjects are summarized by randomized treatment group. cDLQI total score is derived as the sum of the 10 individual item scores, with a range of 0 to 30. Higher scores indicate poorer quality of life."

Update footnote [1] to read "LS mean CFB, LS mean differences (Trifarotene cream HE1 - vehicle), 95% CIs, and P values were obtained from a mixed model for repeated measures (MMRM) with change from baseline in cDLQI score as the repeated dependent variable, fixed effect terms for baseline cDLQI score, treatment, study visit, and treatment-by-study visit interaction as independent variables. An unstructured covariance matrix was used to model the within-subject correlation.

[2] Baseline is defined as the last non-missing assessment recorded prior to the first dose of treatment in the Double-blind Period."

Update SOURCE: to Listing 16.2.6.5.2





# Table 14.2.6.1.1 Secondary Analysis: Presence of Fissures on Palms or Soles ITT Population

| Study Visit Category/Statistic [1] | Trifarotene<br>cream HE1<br>100 ug/g<br>(N=XX) | Trifarotene<br>cream HE1<br>200 ug/g<br>(N=XX) | Overall<br>Trifarotene<br>cream HE1<br>(N=XX) | Vehicle<br>(N=XXX) |
|---|---|---|---|---|
| Baseline [2] | | | | |
| Fissures Present | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| No Fissures Present | xx (xx.x%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Day 14 | | | | |
| Fissures Present | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| No Fissures Present | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Comparison vs. Vehicle | | | | |
| Difference in Percentage of Fissures Present | XX.X | XX.X | XX.X | |
| 95% CI for Difference in Percentage of Fissures Present | (XX.X, XX.X) | (XX.X, XX.X) | (XX.X, XX.X) | |
| P value for Difference | X.XXXX | X.XXXX | X.XXXX | |
| Day 90 | | | | |
| Fissures Present | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| No Fissures Present | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Comparison vs. Vehicle | | | | |
| Difference in Percentage of Fissures Present | XX.X | XX.X | XX.X | |
| 95% CI for Difference in Percentage of Fissures Present | (XX.X, XX.X) | (XX.X, XX.X) | (XX.X, XX.X) | |
| P value for Difference | X.XXXX | X.XXXX | X.XXXX | |

Abbreviations: CI = confidence interval; ITT = intent-to-treat.

Note: Percentages are n/Number of subjects in the ITT population within randomized treatment group\*100.

SOURCE: Listing 16.2.6.6

Programming Note: If cell counts are <5, use Fisher's Exact Test and update footnote [1] accordingly. Include all study visits (Days 14, 30, and 60).

<sup>[1]</sup> P value from 2-sided Pearson's Chi-Square test. Difference is calculated Trifarotene cream HE1 - vehicle.

<sup>[2]</sup> Baseline is defined as the last non-missing assessment recorded prior to the first dose of treatment in the Double-blind Period.





# Table 14.2.6.1.2 Presence of Fissures on Palms or Soles OLE ITT Population

| Trifarotene cream HE1<br>200 ug/g |
|-----------------------------------|
| XX (XX.X%)<br>XX (XX.X%) |
| XX (XX.X%)<br>XX (XX.X%) |
| XX (XX.X%)<br>XX (XX.X%) |
| XX (XX.X%)<br>XX (XX.X%) |
| XX (XX.X%)<br>XX (XX.X%) |
| XX (XX.X%)<br>XX (XX.X%) |

Abbreviations: CI = confidence interval; ITT = intent-to-treat; OLE = open label extension.

Note: Percentages are n/Number of subjects in the OLE ITT population within treatment group\*100. All subjects received Trifarotene cream HE1 200 ug/g in the OLE.

[1] Baseline is defined as the last non-missing assessment recorded prior to the first dose of treatment in the Double-blind Period.

SOURCE: Listing 16.2.6.6





# Table 14.2.6.2.1 Secondary Analysis: Summary of Number of Fissures and Fissure Pain Level ITT Population

Body Area: Palms

| Study Visit Category/Statistic | Trifarotene<br>cream HE1<br>100 ug/g<br>(N=XX) | Trifarotene<br>cream HE1<br>200 ug/g<br>(N=XX) | Overall<br>Trifarotene<br>cream HE1<br>(N=XX) | Vehicle<br>(N=XXX) |
|---|---|---|---|---|
| outogo. y/ otunono | (1770) | (11701) | (11.701) | (11 70 0 1) |
| Baseline [1] | | | | |
| Number of Fissures | | | | |
| n | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX | XX, XX |
| Fissure Pain Level | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| None | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Mild | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Moderate | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Severe | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Day 90 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Number of Fissures | , | , | , | , |
| n | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX | XX, XX |
| Fissure Pain Level | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| None | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Mild | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Moderate | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Severe | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

Abbreviations: CI = confidence interval; ITT = intent-to-treat.

Note: Percentages are n/Number of subjects in the ITT population within randomized treatment group\*100.

[1] Baseline is defined as the last non-missing assessment recorded prior to the first dose of treatment in the Double-blind Period.

SOURCE: Listing 16.2.6.6

Programming note: Repeat for Body Area: Soles. Include all study visits (Days 14, 30, and 60).





# Table 14.2.6.2.2 Summary of Number of Fissures and Fissure Pain Level OLE ITT Population

## Same shell as Table 14.2.6.2.1

Programming note: Only include one set of columns for Trifarotene cream HE1 200 ug/g.

Update Note: to read "Note: Percentages are n/Number of subjects in the OLE ITT population within treatment group\*100. All subjects received Trifarotene cream HE1 200 ug/g in the OLE."

Baseline [2], Days 104, 120, 150, 180, and 194 will be displayed.

Add OLE = open label extension to Abbreviations.





Table 14.2.7.1
Exploratory Analysis: Summary of Change from Baseline in Ectropion Score ITT Population

| Study Visit | 100 ເ | Trifarotene cream HE1<br>100 ug/g<br>(N=XXX) | | |
|---|---|---|---|---|
| Statistic | Observed | CFB | Observed | CFB |
| Baseline [1] | | | | |
| n | XXX | | XXX | |
| Mean (SD) | XX.XX (XX.XXX) | | XX.XX (XX.XXX) | |
| Median | XX.XX | | XX.XX | |
| Min, Max | XX.X, XX.X | | XX.X, XX.X | |
| Day 14 | | | | |
| n | XXX | XXX | XXX | XXX |
| Mean (SD) | XX.XX (XX.XXX) | XX.XX (XX.XXX) | XX.XX (XX.XXX) | XX.XX (XX.XXX) |
| Median | XX.XX | XX.XX | XX.XX | XX.XX |
| Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Day 90 | | | | |
| n | XXX | XXX | XXX | XXX |
| Mean (SD) | XX.XX (XX.XXX) | XX.XX (XX.XXX) | XX.XX (XX.XXX) | XX.XX (XX.XXX) |
| Median | XX.XX | XX.XX | XX.XX | XX.XX |
| Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |

Abbreviations: CFB = change from baseline; ITT = intent to treat; SD = standard deviation.

Note: Subjects are summarized by randomized treatment group. Ectropion total score is derived as the sum of the 8 individual item scores (lateral apposition, medial apposition, scleral show, conjunctival show, excess tear film, redness of the eye, round canthus, punctum lacrimale), with a range of 0 to 8. Each individual item is scored 0 (nonaffected/no/invisible), 0.5 (≤ 1 mm/emerging), or 1 (affected/yes/visible). Higher scores indicates worse ectropion.

[1] Baseline is defined as the last non-missing assessment recorded prior to the first dose of treatment in the Double-blind Period.

SOURCE: Listing 16.2.6.7

Programming note: Include Days 30, and 60 as well. Repeat Table for Overall Trifarotene cream HE1 and Vehicle columns.





# Table 14.2.7.2 Summary of from Baseline in Ectropion Score OLE ITT Population

# Same shell as 14.2.7.1

Programming note: Only include one set of columns for Trifarotene cream HE1 200 ug/g.

Update Note: to read "Note: Percentages are n/Number of subjects in the OLE ITT population within treatment group\*100. All subjects received Trifarotene cream HE1 200 ug/g in the OLE."

Baseline [2], Days 104, 120, 150, 180, and 194 will be displayed.

Add OLE = open label extension to Abbreviations.





Table 14.2.8.1
Exploratory Analysis: Change from Baseline in EQ-5D-5L ITT Population

## Same Shell as Table 14.2.7.1

| | Trifarotene c | ream HF1 | Trifarotene o | ream HF1 |
|---|---|---|---|---|
| | 100 ug | ····· · · <del>-</del> · | 200 u | |
| Study Visit | (N=X) | | (N=X | 0 0 |
| Statistic | Observed | CFB | Observed | CFB |
| | The EQ-5D-5L is intended for use in adult subjects. The EQ VAS records the subject's self-rated healt SOURCE: to Listin | h on a vertical 0-100 VAS. A | | |
| | Table 14.2.<br>Exploratory Analysis: Change fro<br>ITT Populat | om Baseline in EQ-5D-Y | | |
| | Same Shell as Tab | ole 14.2.7.1 | | |
| Programming Note: Headers will be as fo | lows. Repeat for the following Parameters: Taking C<br>or Unhappy, Number Subjec | | Activities, Having Pain or Discon | nfort, Feeling Worried, Sad |
| Parameter: Mobility | | | | |
| | Trifarotene ci | | Trifarotene o | |
| | 100 u | 100 ug/g<br>(N=XXX) | | ıg/g |
| Study Visit | • | VV) | (N=X | <b>YY</b> ) |

Update Note: to read "Subjects are summarized by randomized treatment group. The EQ-5D is a measure of health related quality of life. The EQ-5D consists of a descriptive system and the EQ visual analog scale (VAS). The EQ-5D-Y is to be used for children and adolescents. The descriptive system comprises 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The EQ VAS records the subject's self-rated health on a vertical 0-100 VAS. Add VAS = visual analog scale to Abbreviations. Update SOURCE: to Listing 16.2.6.8





Table 14.3.1.1.1

Overall Summary of Treatment Emergent Adverse Events during the Double-blind Period Safety Population

| Category | Trifarotene cream<br>HE1<br>100 ug/g<br>(N=XX) | Trifarotene cream<br>HE1<br>200 ug/g<br>(N=XX) | Overall<br>Trifarotene cream<br>HE1<br>(N=XX) | Vehicle<br>(N=XX) | Overall<br>(N=XX) |
|---|---|---|---|---|---|
| | (11701) | (1.70.) | (11 701) | (, | (11704) |
| Subjects with at least 1 TEAE | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Subjects with an SAE | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Maximum Severity of TEAE [1] | | | | | |
| Mild | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Moderate | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Severe | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Relationship of TEAE [2] | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Related | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Not Related | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Subjects with a TEAE Leading to Discontinuation of Study Drug | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Subjects with an AE leading to Death | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

Abbreviations: AE = adverse event; CRF = case report form; MedDRA = Medical Dictionary for Regulatory Activities; SAE = serious adverse event; TEAE = treatment emergent adverse event.

Note: Percentages are n/Number of subjects in the Safety Population within actual treatment group and overall\*100. AEs were coded using MedDRA version 21.1. A TEAE is any AE with an onset at the time of or following the start of treatment with study drug through the Follow-up Visit or Early Termination Visit, whichever occurs first. This will include any AE starting prior to the start of treatment but increasing in severity or relationship at the time of, or following, the start of treatment with study drug through the Follow-up Visit or Early Termination Visit, whichever occurs first.

SOURCE: Listing 16.2.7.1

<sup>[1]</sup> Subjects are counted only once at the worst severity. If a severity designation is missing, it will be considered as severe.

<sup>[2]</sup> Subjects are counted only once at the strongest possible relationship. If a relationship designation is missing, the AE will be considered as related. This relationship is categorized for summarization as follows: Related = Related and Possibly Related; Not Related = Not Related and Unlikely Related.





# Table 14.3.1.1.2 Overall Summary of Treatment Emergent Adverse Events during the OLE OLE Safety Population

## Same shell as Table 14.3.1.1.1

Programming note: Only include one set of columns for Trifarotene cream HE1 200 ug/g.

Update Note: to read "Note: Percentages are n/Number of subjects in the OLE Safety population within treatment group\*100. All subjects received Trifarotene cream HE1 200 ug/g in the OLE." Add OLE = open label extension to Abbreviations.





Table 14.3.1.2.1
Incidence of Treatment Emergent Adverse Events during the Double-blind Period by System Organ Class and Preferred Term Safety Population

| System Organ Class<br>Preferred Term | Trifarotene cream HE1<br>100 ug/g<br>(N=XX) | Trifarotene cream HE1<br>200 ug/g<br>(N=XX) | Overall<br>Trifarotene cream HE1<br>(N=XX) | Vehicle<br>(N=XX) | Overall<br>(N=XX) |
|---|---|---|---|---|---|
| Subjects with at least 1 TEAE | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| System Organ Class 1 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Preferred Term 1 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Preferred Term 2 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Preferred Term 3 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| System Organ Class 2 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Preferred Term 1 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Preferred Term 2 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Preferred Term 3 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

Abbreviations: AE = adverse event; MedDRA = Medical Dictionary for Regulatory Activities; PT = preferred term; SOC = system organ class; TEAE = treatment emergent adverse event

Note: Percentages are n/Number of subjects in the Safety Population within actual treatment group and overall\*100. AEs were coded using MedDRA version 21.1. A TEAE is any AE with an onset at the time of or following the start of treatment with study drug through the Follow-up Visit or Early Termination Visit, whichever occurs first. This will include any AE starting prior to the start of treatment but increasing in severity or relationship at the time of, or following, the start of treatment with study drug through the Follow-up Visit or Early Termination Visit, whichever occurs first. Subjects are counted once for each system organ class (SOC) and once for each preferred term (PT). AEs are displayed by descending frequency of SOC, then PT within SOC, and then alphabetically by PT. SOURCE: Listing 16.2.7.1

# Table 14.3.1.2.2 Incidence of Treatment Emergent Adverse Events during the OLE by System Organ Class and Preferred Term OLE Safety Population

## Same shell as 14.3.1.2.1

Programming note: Only include one set of columns for Trifarotene cream HE1 200 ug/g.

Update Note: to read "Note: Percentages are n/Number of subjects in the OLE Safety population within treatment group\*100. All subjects received Trifarotene cream HE1 200 ug/g in the OLE." Add OLE = open label extension to Abbreviations.





Table 14.3.1.3.1
Incidence of Treatment Emergent Adverse Events during the Double-blind Period by System Organ Class, Preferred Term, and Maximum Severity Safety Population

| System Organ Class<br>Preferred Term<br>Severity | Trifarotene cream HE1<br>100 ug/g<br>(N=XX) | Trifarotene cream HE1<br>200 ug/g<br>(N=XX) | Overall<br>Trifarotene cream HE1<br>(N=XX) | Vehicle<br>(N=XX) | Overall<br>(N=XX) |
|---|---|---|---|---|---|
| Severity | (IN-AA) | (N-AA) | (IN-AA) | (N-XX) | (IV-AA) |
| Subjects with at least 1 TEAE | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Mild | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Moderate | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Severe | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| System Organ Class 1 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Mild | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Moderate | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Severe | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Preferred Term 1 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Mild | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Moderate | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Severe | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Preferred Term 2 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Mild | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Moderate | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Severe | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

Abbreviations: AE = adverse event; MedDRA = Medical Dictionary for Regulatory Activities; PT = preferred term; SOC = system organ class; TEAE = treatment emergent adverse event.

Note: Percentages are n/Number of subjects in the Safety Population within actual treatment group and overall\*100. AEs were coded using MedDRA version 21.1. A TEAE is any AE with an onset at the time of or following the start of treatment with study drug through the Follow-up Visit or Early Termination Visit, whichever occurs first. This will include any AE starting prior to the start of treatment but increasing in severity or relationship at the time of, or following, the start of treatment with study drug through the Follow-up Visit or Early Termination Visit, whichever occurs first. Subjects are counted once for each system organ class (SOC) and once for each preferred term (PT) at the maximum severity. The severity shown is the greatest severity reported for a particular subject (Severe > Moderate > Mild). AEs with a missing severity were counted as Severe. AEs are displayed by descending frequency of SOC, then PT within SOC, and then alphabetically by PT. SOURCE: Listing 16.2.7.1





Table 14.3.1.3.2
Incidence of Treatment Emergent Adverse Events during the OLE by System Organ Class, Preferred Term, and Maximum Severity
OLE Safety Population

# Same shell as 14.3.1.3.1

Programming note: Only include one set of columns for Trifarotene cream HE1 200 ug/g.

Update Note: to read "Note: Percentages are n/Number of subjects in the OLE Safety population within treatment group\*100. All subjects received Trifarotene cream HE1 200 ug/g in the OLE." Add OLE = open label extension to Abbreviations.





Table 14.3.1.4.1
Incidence of Treatment Emergent Adverse Events during the Double-blind Period by System Organ Class, Preferred Term, and Relationship to Study Drug Safety Population

| System Organ Class | Trifarotene cream HE1 | Trifarotene cream HE1 | Overall | | |
|---|---|---|---|---|---|
| Preferred Term | 100 ug/g | 200 ug/g | Trifarotene cream HE1 | Vehicle | Overall |
| Relationship [1] | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) |
| Subjects with at least 1 TEAE | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Related | XX (XX.X%) | XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%) |
| Not Related | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| System Organ Class 1 | VV /VV V0/ \ | VV /VV V0/ \ | VV /VV V0/ \ | VV (VV V0/ ) | VV (VV V0/ ) |
| System Organ Class 1 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Related | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Not Related | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Preferred Term 1 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Related | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Not Related | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Preferred Term 2 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Related | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Not Related | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

Abbreviations: AE = adverse event; MedDRA = Medical Dictionary for Regulatory Activities; PT = preferred term; SOC = system organ class; TEAE = treatment emergent adverse event.

Note: Percentages are n/Number of subjects in the Safety Population within actual treatment group and overall\*100. AEs were coded using MedDRA version 21.1. A TEAE is any AE with an onset at the time of or following the start of treatment with study drug through the Follow-up Visit or Early Termination Visit, whichever occurs first. This will include any AE starting prior to the start of treatment but increasing in severity or relationship at the time of, or following, the start of treatment with study drug through the Follow-up Visit or Early Termination Visit, whichever occurs first. Subjects are counted once for each system organ class (SOC) and once for each preferred term (PT) at the greatest relationship category. The relationship shown is the greatest relationship reported for a particular subject (Related > Not Related). AEs with a missing relationship were counted as Related. AEs are displayed by descending frequency of SOC, then PT within SOC, and then alphabetically by PT.

[1] Related = Related and Possibly Related; Not Related = Not Related and Unlikely Related.

SOURCE: Listing 16.2.7.1





Table 14.3.1.4.2
Incidence of Treatment Emergent Adverse Events during the OLE by System Organ Class, Preferred Term, and Relationship to Study Drug
OLE Safety Population

## Same shell as 14.3.1.4.1

Programming note: Only include one set of columns for Trifarotene cream HE1 200 ug/g.

Update Note: to read "Note: Percentages are n/Number of subjects in the OLE Safety population within treatment group\*100. All subjects received Trifarotene cream HE1 200 ug/g in the OLE." Add OLE = open label extension to Abbreviations.



Table 14.3.2.1.1
Incidence of Adverse Events Leading to Withdrawal during the Double-blind Period by SOC, PT, and Treatment Safety Population

### Same shell as Table 14.3.1.2.1

Programming note: Update first row text to "Subjects with at least 1 TEAE Leading to Withdrawal."

Table 14.3.2.1.2
Incidence of Adverse Events Leading to Withdrawal during the OLE by SOC, PT, and Treatment OLE Safety Population

## Same shell as Table 14.3.1.2.2

Programming note: Update first row text to "Subjects with at least 1 TEAE Leading to Withdrawal."

Table 14.3.2.2.1
Incidence of Serious Adverse Events during the Double-blind Period by SOC, PT, and Treatment Safety Population

## Same shell as Table 14.3.1.2.1

Programming note: Update first row text to "Subjects with at least 1 SAE." Add SAE = serious adverse event to abbreviations.

Table 14.3.2.2.2
Incidence of Serious Adverse Events during the OLE by SOC, PT, and Treatment OLE Safety Population

# Same shell as Table 14.3.1.2.2

Programming note: Update first row text to "Subjects with at least 1 SAE." Add SAE = serious adverse event to abbreviations.





# Table 14.3.3.1.1 Listing of Adverse Events Leading to Withdrawal during the Double-blind Period Safety Population

## Randomized Treatment: XXXXXXXXXXXXXXXXX

| Subject | TE 4 E 0 [4] | System Organ Class/<br>Preferred Term/ | Start Date/Time (Study Day)/ | | Outcome | Serious?/ | Action Taken/<br>Other Action Taken? |
|---|---|---|---|---|---|---|---|
| ID | TEAE? [1] | Verbatim Term | End Date/Time (Study Day) | Relationship to Study Drug | | Criteria Met | |
| xxxxx | xxx | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYYY/HH:MM (X)/<br>DDMMMYYYY/HH:MM (X) | XXXXXXXXX/<br>XXXXXXXXXX | xxxxxxxx | XX | XXXXXXXX/<br>XXXXXXXXX |
| xxxxx | XX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYYY/HH:MM (X)/<br>DDMONYYYY/HH:MM (X) | XXXXXXXXX/<br>XXXXXXXXXX | xxxxxxxx | XX | XXXXXXXXX/<br>XXXXXXXXX |
| | XXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYYY/HH:MM (X)/<br>Ongoing | XXXXXXXXX/<br>XXXXXXXXXX | XXXXXXXXX/ | XXX/<br>XXXXXXXXX | XXXXXXXXX/<br>XXXXXXXXX |

Abbreviations: AE = adverse event; MedDRA = Medical Dictionary for Regulatory Activities; TEAE = treatment emergent adverse event.

Note: Study day is calculated relative to the date of first dose of study drug. AEs were coded using MedDRA version 21.1.

[1] A TEAE is any AE with an onset at the time of or following the start of treatment with study drug through the Follow-up Visit or Early Termination Visit, whichever occurs first. This will include any AE starting prior to the start of treatment but increasing in severity or relationship at the time of, or following, the start of treatment with study drug through the Follow-up Visit or Early Termination Visit, whichever occurs first.

Programming note: If time missing, display "- -:- -". If Serious? is Yes, concatenate all serious criteria marked as Yes with a semicolon. If Other Action Taken? Is Yes, concatenate Medication Required, Relevant Procedure, Procedure Specify, Other, or Other Specify with a colon as applicable. If no events meet the criteria for display, present "No events are reported." SOC & PT text should be in proper case in table.





Table 14.3.3.1.2
Listing of Adverse Events Leading to Withdrawal during the OLE
OLE Safety Population

### Same shell as Table 14.3.3.1.1

**Programming note:** Add OLE = open label extension to Abbreviations.

Table 14.3.3.2.1 Listing of Serious Adverse Events during the Double-blind Period Safety Population

Same shell as Table 14.3.3.1.1

Table 14.3.3.2.2
Listing of Serious Adverse Events during the OLE
OLE Safety Population

Same shell as Table 14.3.3.1.1

**Programming note:** Add OLE = open label extension to Abbreviations.

Table 14.3.3.3.1 Listing of Deaths during the Double-blind Period Safety Population

Same shell as Table 14.3.3.1.1

Table 14.3.3.3.1 Listing of Deaths during the OLE OLE Safety Population

Same shell as Table 14.3.3.1.1

**Programming note:** Add OLE = open label extension to Abbreviations.





# Table 14.3.4.1 Listing of Abnormal Laboratory Data Safety Population and OLE Safety Population

# Randomized Treatment: XXXXXXXXXXX

| Subject ID | Parameter Category | Parameter (unit) | Study<br>Visit | Date/Time of<br>Assessment<br>(Study Day) | Standard<br>Results | Standard<br>Reference<br>Range<br>[1] | Standard<br>Reference<br>Range<br>Flag |
|---|---|---|---|---|---|---|---|
| XXXXX | Chemistry | Albumin (unit) | xxxxx | DDMMMYYYY/<br>HH:MM (X) | XX | XX – YY | |
| | | | XXXXXX | DDMMMYYYY/<br>HH:MM (X) | XX | XX – YY | XXX |
| | | | XXXXXX | DDMMMYYYY/<br>HH:MM (X) | XX | XX – YY | |
| | | | XXXXXX | ( ) | ND | | |
| | | | XXXXXX | DDMMMYYYY/<br>HH:MM (X) | XX | XX – YY | |

Abbreviations: AL = abnormal-low; AH = abnormal-high; ND = not done.

Note: Study day is calculated relative to the date of first dose of study drug. Assessments marked as Not Done are not presented.

[1] Reference range is used to identify potentially clinically significant laboratory values.

**Programming note:** include all parameter categories and parameters.





Table 14.3.5.1.1.1 Laboratory Data: Change from Baseline in Clinical Chemistry Parameters by Study Visit Safety Population

Parameter: XXXXXXX (unit)

| Study Visit | 100 | Trifarotene cream HE1<br>100 ug/g<br>(N=XX) | | Trifarotene cream HE1<br>200 ug/g<br>(N=XX) | | erall<br>cream HE1<br>XX) |
|---|---|---|---|---|---|---|
| Statistic | Observed | CFB | Observed | CFB | Observed | CFB |
| Baseline [1] | | | | | | |
| n<br>Mean (SD)<br>Median<br>Min, Max | XX<br>XX.X (XX.XX)<br>XX.X<br>XX, XX | | XX<br>XX.X (XX.XX)<br>XX.X<br>XX, XX | | XX<br>XX.X (XX.XX)<br>XX.X<br>XX, XX | |
| Day 30 | | | | | | |
| n<br>Mean (SD)<br>Median<br>Min, Max | XX<br>XX.X (XX.XX)<br>XX.X<br>XX, XX | XX<br>XX.X (XX.XX)<br>XX.X<br>XX, XX | XX<br>XX.X (XX.XX)<br>XX.X<br>XX, XX | XX<br>XX.X (XX.XX)<br>XX.X<br>XX, XX | XX<br>XX.X (XX.XX)<br>XX.X<br>XX, XX | XX<br>XX.X (XX.XX)<br>XX.X<br>XX, XX |
| Day 90 | | | | | | |
| n<br>Mean (SD)<br>Median<br>Min, Max | XX<br>XX.X (XX.XX)<br>XX.X<br>XX, XX | XX<br>XX.X (XX.XX)<br>XX.X<br>XX, XX | XX<br>XX.X (XX.XX)<br>XX.X<br>XX, XX | XX<br>XX.X (XX.XX)<br>XX.X<br>XX, XX | XX<br>XX.X (XX.XX)<br>XX.X<br>XX, XX | XX<br>XX.X (XX.XX)<br>XX.X<br>XX, XX |

Repeat for all clinical chemistry parameters.

Abbreviation: CFB = change from baseline; SD = standard deviation. Note: Subjects are summarized by actual treatment group and overall.

[1] Baseline is defined as the last non-missing assessment recorded prior to the first dose of treatment in the Double-blind Period.

SOURCE: Listing 16.2.8.1

Programming note: Repeat table for Vehicle and Overall columns.





Table 14.3.5.1.1.2
Laboratory Data: Change from Baseline in Clinical Chemistry Parameters by Study Visit
OLE Safety Population

# Same shell as Table 14.3.5.1.1.1

**Programming note:** Only include one set of columns for Trifarotene cream HE1 200 ug/g. Update Note: to read "Subjects are summarized by treatment group. All subjects received Trifarotene cream HE1 200 ug/g in the OLE." Visits will be Baseline, Day 120, and Day 180. Add OLE = open label extension to Abbreviations.





# Table 14.3.5.1.2.1 Laboratory Data: Shift from Baseline in Clinical Chemistry Parameters by Study Visit Safety Population

Parameter: XXXXXXX

| | | Baselin | e [1] | |
|---|---|---|---|---|
| | Trifarotene cream HE1 100 ug/g (N=XX) | | | |
| Study Visit | Low | Normal | High | Missing |
| Category | n (%) | n (%) | n (%) | n (%) |
| Day 30 | | | | |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Normal | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Missing | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Day 90 | | | | |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Normal | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Missing | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

Continue for other parameters. Sort alphabetically by parameter.

Note: Note: Percentages are n/Number of subjects in the Safety Population within actual treatment group and overall\*100.

[1] Baseline is defined as the last non-missing assessment recorded prior to the first dose of treatment in the Double-blind Period.

SOURCE: Listing 16.2.8.1

Programming note: Repeat table for Trifarotene cream HE1 200 ug/g, Overall Trifarotene cream HE1, Vehicle, and Overall treatment groups.

Table 14.3.5.1.2.2
Laboratory Data: Shift from Baseline in Clinical Chemistry Parameters by Study Visit
OLE Safety Population

## Same shell as Table 14.3.5.1.2.1

Programming note: Only include Trifarotene cream HE1 200 ug/g. Update Note: to read "Subjects are summarized by treatment group. All subjects received Trifarotene cream HE1 200 ug/g in the OLE." Visits will be Baseline, Day 120, and Day 180. Add OLE = open label extension to Abbreviations.





Table 14.3.5.2.1.1

Laboratory Data: Change from Baseline in Hematology Parameters by Study Visit

Safety Population

### Same shell as Table 14.3.5.1.1.1

Programming note: Update SOURCE: to Listing 16.2.8.2

Table 14.3.5.2.1.2
Laboratory Data: Change from Baseline in Hematology Parameters by Study Visit
OLE Safety Population

### Same shell as Table 14.3.5.1.1.1

**Programming note:** Only include one set of columns for Trifarotene cream HE1 200 ug/g. Update Note: to read "Subjects are summarized by treatment group. All subjects received Trifarotene cream HE1 200 ug/g in the OLE." Visits will be Baseline, Day 120, and Day 180. Add OLE = open label extension to Abbreviations. Update SOURCE: to Listing 16.2.8.2

Table 14.3.5.2.2.1
Laboratory Data: Shift from Baseline in Hematology Parameters by Study Visit
Safety Population

## Same shell as Table 14.3.5.1.2.1

**Programming note:** Update SOURCE: to Listing 16.2.8.2

Table 14.3.5.2.2.2
Laboratory Data: Shift from Baseline in Hematology Parameters by Study Visit
OLE Safety Population

### Same shell as Table 14.3.5.1.2.1

**Programming note:** Only include one set of columns for Trifarotene cream HE1 200 ug/g. Update Note: to read "Subjects are summarized by treatment group. All subjects received Trifarotene cream HE1 200 ug/g in the OLE." Visits will be Baseline, Day 120, and Day 180. Add OLE = open label extension to Abbreviations. Update SOURCE: to Listing 16.2.8.2





Table 14.3.5.3.1.1
Laboratory Data: Change from Baseline in Coagulation Parameters by Study Visit
Safety Population

### Same shell as Table 14.3.5.1.1.1

Programming note: Update SOURCE: to Listing 16.2.8.3

Table 14.3.5.3.1.2
Laboratory Data: Change from Baseline in Coagulation Parameters by Study Visit
OLE Safety Population

### Same shell as Table 14.3.5.1.1.1

**Programming note:** Only include one set of columns for Trifarotene cream HE1 200 ug/g. Update Note: to read "Subjects are summarized by treatment group. All subjects received Trifarotene cream HE1 200 ug/g in the OLE." Visits will be Baseline, Day 120, and Day 180. Add OLE = open label extension to Abbreviations. Update SOURCE: to Listing 16.2.8.3

Table 14.3.5.3.2.1
Laboratory Data: Shift from Baseline in Coagulation Parameters by Study Visit
Safety Population

## Same shell as Table 14.3.5.1.2.1

**Programming note:** Update SOURCE: to Listing 16.2.8.3

Table 14.3.5.3.2.2
Laboratory Data: Shift from Baseline in Coagulation Parameters by Study Visit
OLE Safety Population

### Same shell as Table 14.3.5.1.2.1

**Programming note:** Only include one set of columns for Trifarotene cream HE1 200 ug/g. Update Note: to read "Subjects are summarized by treatment group. All subjects received Trifarotene cream HE1 200 ug/g in the OLE." Visits will be Baseline, Day 120, and Day 180. Add OLE = open label extension to Abbreviations. Update SOURCE: to Listing 16.2.8.3





Table 14.3.5.4.1.1 Laboratory Data: Change from Baseline in Quantitative Urinalysis Parameters by Study Visit Safety Population

### Same shell as Table 14.3.5.1.1.1

Programming note: Update SOURCE: to Listing 16.2.8.4

Table 14.3.5.4.1.2
Laboratory Data: Change from Baseline in Quantitative Urinalysis Parameters by Study Visit
OLE Safety Population

## Same shell as Table 14.3.5.1.1.1

**Programming note:** Only include one set of columns for Trifarotene cream HE1 200 ug/g. Update Note: to read "Subjects are summarized by treatment group. All subjects received Trifarotene cream HE1 200 ug/g in the OLE." Visits will be Baseline, Day 120, and Day 180. Add OLE = open label extension to Abbreviations. Update SOURCE: to Listing 16.2.8.4

Table 14.3.5.4.2.1
Laboratory Data: Shift from Baseline in Quantitative Urinalysis Parameters by Study Visit Safety Population

## Same shell as Table 14.3.5.1.2.1

Programming note: Update SOURCE: to Listing 16.2.8.4

Table 14.3.5.4.2.2 Laboratory Data: Shift from Baseline in Quantitative Urinalysis Parameters by Study Visit OLE Safety Population

### Same shell as Table 14.3.5.1.2.1

**Programming note:** Only include one set of columns for Trifarotene cream HE1 200 ug/g. Update Note: to read "Subjects are summarized by treatment group. All subjects received Trifarotene cream HE1 200 ug/g in the OLE." Visits will be Baseline, Day 120, and Day 180. Add OLE = open label extension to Abbreviations. Update SOURCE: to Listing 16.2.8.4





Table 14.3.5.4.3.1 Laboratory Data: Summary of Qualitative Urinalysis Parameters by Study Visit Safety Population

Parameter: XXXXXXX (unit)

| | Trifarotene cream HE1 | Trifarotene cream HE1 | Overall | | |
|---|---|---|---|---|---|
| Study Visit | 100 ug/g | 200 ug/g<br>(N=XX) | Trifarotene cream HE1<br>(N=XX) | Vehicle<br>(N=XX) | Overall<br>(N=XX) |
| Category | (N=XX) | | | | |
| Baseline [1] | | | | | |
| Category 1 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Category 2 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Category 3 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Day 30 | | | | | |
| Category 1 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Category 2 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Category 3 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 5 , | , | , | ( | , | , |
| Day 90 | | | | | |
| Category 1 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Category 2 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Category 3 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

Note: Percentages are n/Number of subjects in the ITT population within randomized treatment group and overall\*100.

[1] Baseline is defined as the last non-missing assessment recorded prior to the first dose of treatment in the Double-blind Period.

SOURCE: Listing 16.2.8.4

Table 14.3.5.4.3.2 Laboratory Data: Summary of Qualitative Urinalysis Parameters by Study Visit OLE Safety Population

## Same shell as Table 14.3.5.4.3.1

**Programming note:** Only include one set of columns for Trifarotene cream HE1 200 ug/g. Update Note: to read "Subjects are summarized by treatment group. All subjects received Trifarotene cream HE1 200 ug/g in the OLE." Visits will be Baseline, Day 120, and Day 180. Add OLE = open label extension to Abbreviations.





Table 14.3.6.1.1 Summary of Vital Signs by Study Visit Safety Population

## Same shell as Table 14.3.5.1.1.1

Programming note: Visits include Baseline [1], Days 14, 30, 60, and 90. Parameters include weight (kg), BMI (kg/m²), systolic blood pressure (mmHg), and diastolic blood pressure (mmHg). Include derivation of BMI in Note: Body Mass Index (BMI) = weight (kg) / [height (m)]². Update SOURCE: to Listings 16.2.9.1

Table 14.3.6.1.2 Summary of Vital Signs by Study Visit OLE Safety Population

## Same shell as Table 14.3.5.1.1.1

Programming note: Only include one set of columns for Trifarotene cream HE1 200 ug/g. Update Note: to read "Subjects are summarized by treatment group. All subjects received Trifarotene cream HE1 200 ug/g in the OLE." Visits include Baseline [1], Days 120, 180, and 194. Parameters include weight (kg), BMI (kg/m²), systolic blood pressure (mmHg), and diastolic blood pressure (mmHg). Include derivation of BMI in Note: Body Mass Index (BMI) = weight (kg) / [height (m)]². Add OLE = open label extension to Abbreviations. Update SOURCE: to Listings 16.2.9.1





# Table 14.3.6.2.1 Summary of 12-Lead Electrocardiogram by Study Visit Safety Population

## Same shell as Table 14.3.5.1.1.1

Programming note: Visits include Baseline [1], Days 30 and 90. Parameters include heart rate (bpm), PR interval (ms), QRS interval (ms), uncorrected QT interval (ms), and QTcF (ms). Update SOURCE: to Listings 16.2.9.2

Table 14.3.6.2.2 Summary of 12-Lead Electrocardiogram by Study Visit OLE Safety Population

## Same shell as Table 14.3.5.1.1.1

Programming note: Only include one set of columns for Trifarotene cream HE1 200 ug/g. Update Note: to read "Subjects are summarized by treatment group. All subjects received Trifarotene cream HE1 200 ug/g in the OLE." Visits include Baseline [1], Days 120 and 180. Parameters include heart rate (bpm), PR interval (ms), QRS interval (ms), uncorrected QT interval (ms), and QTcF (ms). Add OLE = open label extension to Abbreviations. Update SOURCE: to Listings 16.2.9.2





# Table 14.3.6.2.3 Summary of 12-Lead Electrocardiogram Interpretation by Study Visit Safety Population

| Study Visit<br>Category | Trifarotene cream HE1<br>100 ug/g<br>(N=XX) | Trifarotene cream HE1<br>200 ug/g<br>(N=XX) | Overall<br>Trifarotene cream HE1<br>(N=XX) | Vehicle<br>(N=XX) | Overall<br>(N=XX) |
|---|---|---|---|---|---|
| Baseline [1]<br>Normal<br>Abnormal | XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%) |
| Day 30<br>Normal<br>Abnormal | XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%) |
| Day 90<br>Normal<br>Abnormal | XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%) |

Note: Percentages are n/Number of subjects in the Safety population within actual treatment group and overall\*100.

[1] Baseline is defined as the last non-missing assessment recorded prior to the first dose of treatment in the Double-blind Period.

SOURCE: Listing 16.2.9.2

# Table 14.3.6.2.4 Summary of 12-Lead Electrocardiogram Interpretation by Study Visit OLE Safety Population

## Same shell as Table 14.3.6.2.3

**Programming note:** Only include one set of columns for Trifarotene cream HE1 200 ug/g. Update Note: to read "Subjects are summarized by treatment group. All subjects received Trifarotene cream HE1 200 ug/g in the OLE." Visits include Baseline [1], Days 120 and 180.





# Table 14.3.6.3.1 Summary of Local Tolerability Assessments by Study Visit Safety Population

| Body Area | Trifarotene cream HE1 | ne cream HE1 Trifarotene cream HE1 | | | |
|---|---|---|---|---|---|
| Assessment | 100 ug/g | 200 ug/g | Trifarotene cream HE1 | Vehicle | Overall |
| Score | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) |
| Chest/Abdomen | | | | | |
| Erythema | | | | | |
| None | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Mild | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Moderate | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Severe | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Stinging/Burning | | | | | |
| None | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Mild | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Moderate | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Severe | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Pruritus | | | | | |
| None | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Mild | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Moderate | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Severe | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

Note: Percentages are n/Number of subjects in the Safety population within actual treatment group and overall\*100.

[1] Baseline is defined as the last non-missing assessment recorded prior to the first dose of treatment in the Double-blind Period.

SOURCE: Listing 16.2.9.3

Programming note: Continue for Back, Arms, and Legs. Visits will be Baseline [1], Day 14, Day 30, Day 60, and Day 90.

Table 14.3.6.3.2 Summary of Local Tolerability Assessments by Study Visit OLE Safety Population

### Same shell as Table 14.3.6.3.1

Programming note: Continue for Back, Arms, and Legs. Visits will be Baseline [1], Day 104, Day 120, and Day 150. Update Note: to read "Note: Percentages are n/Number of subjects in the OLE Safety population within treatment group\*100. All subjects received Trifarotene cream HE1 200 ug/g in the OLE." Add OLE = open label extension to Abbreviations.





# Table 14.3.6.4.1 Summary of Physical Examination Results by Study Visit Safety Population

| Result<br>Clinically<br>Significant? | Trifarotene cream HE1<br>100 ug/g<br>(N=XX) | Trifarotene cream HE1<br>200 ug/g<br>(N=XX) | Overall<br>Trifarotene cream HE1<br>(N=XX) | Vehicle<br>(N=XX) | Overall<br>(N=XX) |
|---|---|---|---|---|---|
| Body System 1 | | | | | |
| Not Done | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Normal | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Abnormal | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Yes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| No | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Body System 2 | | | | | |
| Not Done | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Normal | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Abnormal | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Yes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| No | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

Note: Percentages are n/Number of subjects in the Safety population within actual treatment group and overall\*100.

[1] Baseline is defined as the last non-missing assessment recorded prior to the first dose of treatment in the Double-blind Period.

SOURCE: Listing 16.3.9.4

Programming note: Continue for all body systems. Visits will be Baseline [1] and Day 90.

Table 14.3.6.4.2 Summary of Physical Examination Results by Study Visit OLE Safety Population

## Same shell as Table 14.3.6.4.1

Programming note: Visits will be Day 180 and Day 194. Update Note: to read "Note: Percentages are n/Number of subjects in the OLE Safety population within treatment group\*100.

All subjects received Trifarotene cream HE1 200 ug/g in the OLE." Add OLE = open label extension to Abbreviations.





Table 14.3.6.5.1
Summary of Concomitant Medications during the Double-blind Period by ATC Class Level 4 and Preferred Term Safety Population

### Same shell as Table 14.1.4

Programming note: Update Note: to read "Note: Percentages are n/Number of subjects in the Safety population within actual treatment group and overall\*100. Medications were coded using WHO-DDE version March 2019. Concomitant medications are any medications continuing or starting after the first dose of study drug through the end of study. Medications are displayed by descending frequency of ATC Level 4 classification, by PT within ATC, and then alphabetically by PT, based on the overall column. Subjects were counted only once for each ATC and PT. Include an additional column for Overall Trifarotene cream HE1.

Table 14.3.6.5.2
Summary of Concomitant Medications during the OLE by ATC Class Level 4 and Preferred Term Safety Population

### Same shell as Table 14.1.4

Programming note: Update Note: to read "Note: Percentages are n/Number of subjects in the OLE Safety population within treatment group\*100. All subjects received Trifarotene cream HE1 200 ug/g in the OLE. Medications were coded using WHO-DDE version March 2019. Concomitant medications are any medications continuing or starting after the first dose of study drug through the end of study. Medications are displayed by descending frequency of ATC Level 4 classification, by PT within ATC, and then alphabetically by PT, based on the overall column. Subjects were counted only once for each ATC and PT. Include an additional column for Overall Trifarotene cream HE1.




Table 14.4.1.1 Summary of Pharmacokinetic Concentrations by Study Visit PK Population

| | Trifarotene cream HE1 | Trifarotene cream HE1 |
|--------------------------|-----------------------|-----------------------|
| Study Visit | 100 ug/g | 200 ug/g |
| Statistic | (N=XX) | (N=XX) |
| Day 1, Pre-Dose | | |
| n | XX | XX |
| Mean (SD) | XX.X (XX.X) | XX.X (XX.X) |
| Geomètric Mean | XX.X ′ | xx.x ´ |
| Median | XX.X | XX.X |
| Min, Max | XX, XX | XX, XX |
| %CV | XX.X | XX.X |
| Day 1, 1 hour Post-Dose | | |
| n | XX | XX |
| Mean (SD) | XX.X (XX.X) | XX.X (XX.X) |
| Geometric Mean | XX.X | XX.X |
| Median | XX.X | XX.X |
| Min, Max | XX, XX | XX, XX |
| %CV | XX.X | XX.X |
| Day 1, 2 Hours Post-Dose | | |
| n | XX | XX |
| Mean (SD) | XX.X (XX.X) | XX.X (XX.X) |
| Geometric Mean | XX.X | XX.X |
| Median | XX.X | XX.X |
| Min, Max | XX, XX | XX, XX |
| %CV | XX.X | XX.X |
| | · <del></del> | |

Abbreviation: BLQ = below limit of quantification; PK = pharmacokinetic; SD = standard deviation.

Note: Values below the lower limit of quantification (<BLQ) have been set to zero in the calculation of the summary statistics.

SOURCE: Listing 16.2.5.4.1, 16.2.5.4.2, 16.2.4.3

Programming note: Time points will be pre-dose, 1, 2, 4, 8, 12, and 24 hours post dose on Day 1 and Day 30.





### Table 14.4.1.2 Summary of Pharmacokinetic Parameters PK Population

| | Trifarotene cream HE1 | Trifarotene cream HE1 |
|---|---|---|
| Study Visit | 100 ug/g | 200 ug/g |
| Statistic | (N=XX) | (N=XX) |
| ALLO (resolved *her) | | |
| $AUC_{(0-t)}$ (ng/mL*hr) | VOV | <b>V</b> 0/ |
| n (OD) | XX | XX |
| Mean (SD) | XX.X (XX.X) | XX.X (XX.X) |
| Geometric Mean | XX.X | XX.X |
| Median | XX.X | XX.X |
| Min, Max | XX, XX | XX, XX |
| %CV | XX.X | XX.X |
| C <sub>max</sub> (ng/mL) n Mean (SD) Geometric Mean Median Min, Max %CV | XX<br>XX.X (XX.X)<br>XX.X<br>XX.X<br>XX, XX<br>XX.X | XX<br>XX.X (XX.X)<br>XX.X<br>XX.X<br>XX, XX<br>XX.X |
| Median | XX.X | XX.X |
| IVICUIAII | XX, XX | |

Abbreviation: AUC = area under the plasma concentration-time curve; BLQ = below limit of quantification; Cmax = peak plasma concentration; CV = coefficient of variation;  $\lambda_z$  = apparent terminal phase rate constant; PK = pharmacokinetic; SD = standard deviation; t1/2= first order termination half-life; Tmax = time of Cmax. SOURCE: Listing 16.2.5.4.4

**Programming note:** Continue for AUC<sub>0-inf</sub>,  $t_{1/2}$ ,  $\lambda_z$  if data permit. If not, do not include in abbreviations.





## 14.3. Planned Listing Shells

Listing 16.2.1 Subject Disposition All Subjects

Randomized Treatment: XXXXXXXXX

| | | | Doub | ole-blind Period | | | OLE | |
|---|---|---|---|---|---|---|---|---|
| Subject<br>ID | Date Informed<br>Consent Signed | Subject<br>Status | Date of<br>Completion/<br>Discontinuation<br>(Study Day) | Reason for Early<br>Termination | Was the Blind<br>Broken<br>For This<br>Subject? | Subject<br>Status | Date of<br>Completion/<br>Discontinuation<br>(Study Day) | Reason for Early<br>Termination |
| XXXXXX | DDMMMYYYY | xxxxx | DDMMMYYYY<br>(XX) | | | xxxxxx | DDMMMYYYY<br>(XX) | |
| XXXXXX | DDMMMYYYY | XXXXXX | DDMMMYYYY<br>(XX) | | | XXXXXX | DDMMMYYYY<br>(XX) | |
| XXXXXX | DDMMMYYYY | XXXXXX | DDMMMYYYY<br>(XX) | XXXXXXXX: XXXXXX | | XXXXXX | DDMMMYYYY<br>(XX) | XXXXXXXX: XXXXXX |
| XXXXXX | DDMMMYYYY | XXXXXX | DDMMMYYYY (X) | XXXXXX | | XXXXXX | DDMMMYYYY (X) | XXXXXX |
| XXXXXX | DDMMMYYYY | XXXXXX | DDMMMYYYY<br>(XX) | xxxxxxxxxxx | XXX;<br>XXXXXX;<br>XXXXX | XXXXXX | DDMMMYYYY<br>(XX) | XXXXXXXXXXXXX |

Abbreviation: OLE = open label extension.

Note: Subjects were randomized to either Trifarotene cream HE1 100 ug/g, Trifarotene cream HE1 200 ug/g, or vehicle in the double-blind period. All subjects received Trifarotene cream HE1 200 ug/g in the open label extension period. Study day is calculated relative to the date of first dose of study drug.

Programming Note: Subject status will be completed continuing, completed not continuing, or early termination. If reason for early termination is AE, Physician Decision, Protocol Violation, or Other, concatenate the specify text as follows: "Other: XXXXXXXXX". If reason for early termination is lost to follow-up, concatenate with date of last contact and comments as follows: "Lost to follow-up; date of last contact: DDMMMYYYY; XXXXX". If reason for early termination is death, concatenate with comment, cause of death and date of death as follows: "Lost to follow-up; XXXXX; date of death: DDMMMYYYY; comment: XXXX".





### Listing 16.2.2.1 Inclusion and Exclusion Criteria All Subjects

Randomized Treatment: XXXXXXX

| | Assessment Date | | Inclusion Criteria | | Exclusion Criteria |
|---|---|---|---|---|---|
| Subject ID | (Study Day) | Met All Inclusion Criteria? | Number(s) Not Met [1] | Met Any Exclusion Criteria? | Number(s) Met [2] |
| xxxxx | DDMMMYYYY (XX) | Yes | | No | |
| xxxxx | DDMMMYYYY (XX) | Yes | | No | |
| XXXXX | DDMMMYYYY (XX) | Yes | | No | |
| XXXXX | DDMMMYYYY (XX) | No | XX | No | |
| XXXXX | DDMMMYYYY (XX) | Yes | | No | |
| XXXXX | DDMMMYYYY (XX) | Yes | | Yes | XX; XX |

Note: Subjects were randomized to either Trifarotene cream HE1 100 ug/g, Trifarotene cream HE1 200 ug/g, or vehicle in the double-blind period. All subjects received Trifarotene cream HE1 200 ug/g in the open label extension period. Study day is calculated relative to the date of first dose of study drug.

**Programming note:** If more than 1 inclusion or exclusion criterion number exists, concatenate with a comma as shown above. Decode any relevant criteria in the footnotes as shown in the example. If no criteria are present for a column, remove the [1] and/or [2] from the column header.





Listing 16.2.2.2 Screen Failures All Subjects

| Subject ID | Date of Screen Failure<br>(Study Day) | Reason for Screen Failure | Other Reason for Screen Failure |
|---|---|---|---|
| XXXXXX | DDMMMYYYY (XX) | xxxxxx | xxxxxxxxxxxx |
| xxxxx | DDMMMYYYY (XX) | xxxxxx | |
| xxxxx | DDMMMYYYY (XX) | xxxxxx | |
| xxxxx | DDMMMYYYY (XX) | xxxxxx | xxxxxxxxxxx |
| xxxxx | DDMMMYYYY (XX) | xxxxxx | |
| xxxxx | DDMMMYYYY (XX) | xxxxxx | |

Note: Subjects were randomized to either Trifarotene cream HE1 100 ug/g, Trifarotene cream HE1 200 ug/g, or vehicle in the double-blind period. All subjects received Trifarotene cream HE1 200 ug/g in the open label extension period. Study day is calculated relative to the date of first dose of study drug.





### Listing 16.2.2.3 Protocol Deviations All Subjects

Randomized Treatment: XXXXXXXXXXX

| Subject<br>ID | Date Identified<br>(Study Day) | Event Date<br>(Study Day) | Study<br>Visit | Event Type | Violation<br>Level | Description | Action/Resolution | Reportable to IRB? | Excluded from PP Population? |
|---|---|---|---|---|---|---|---|---|---|
| xxxxx | DDMMMYYYYE<br>(XX) | DDMMMYYYY<br>(XX) | 'XXXXX | (XXXXXXXXXXX | MAJOR | xxxxxx | xxxxxx | XXX;<br>DDMMMYYYY;<br>XXXXX | XXX |
| | DDMMMYYYYE<br>(XX) | DDMMMYYYY<br>(XX) | XXXXX | (XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | MINOR | XXXXXXXXXXXXX | XXXXXXXXXXXXX | | XXX |
| xxxxx | DDMMMYYYYI<br>(XX) | DDMMMYYYY<br>(XX) | ′XXXXX | (XXXXXXXXXXXX | MINOR | xxxxxxxxxxxxxxx | xxxxxxxxxxxxxxx | | XX |
| xxxxx | DDMMMYYYYI<br>(X) | DDMMMYYYY<br>(X) | ′XXXXX | (XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | MAJOR | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | (XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | < | xx |

Abbreviation: IRB = institutional review board; PP = per protocol.

Note: Subjects were randomized to either Trifarotene cream HE1 100 ug/g, Trifarotene cream HE1 200 ug/g, or vehicle in the double-blind period. All subjects received Trifarotene cream HE1 200 ug/g in the open label extension period. Study day is calculated relative to the date of first dose of study drug.

**Programming note:** the structure of this listing may change depending on the information in the protocol deviations file. If Reportable to IRB is yes, concatenate IRB Submission Date and IRB Submission Comments fields with a semicolon.





### Listing 16.2.3 Analysis Populations All Subjects

| Subject | | Randomiza | ntion | Actual | | | Anal | ysis Populat | ions | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | ITT/ | mITT/<br>OLE | PP/<br>OLE | Safety/<br>OLE | | |
| | | | | | OLE ITT | mITT | PP | Safety | PK | Primary Reason(s) for |
| ID | Date | Number | Treatment | Treatment | [1] | [2] | [3] | [4] | [5] | Exclusion |
| xxxxxx | DDMMMYYYY | xxxx | xxxxxxxxxx | XXXXXXXXXXX | Yes | Yes | No | Yes | No | PP: Subject had a significant protocol violation. |
| XXXXXX | DDMMMYYYY | XXXX | xxxxxxxxx | xxxxxxxxx | Yes | Yes | Yes | Yes | Yes | |
| XXXXXX | DDMMMYYYY | xxxx | xxxxxxxxx | xxxxxxxx | No | Yes | No | Yes | No | Safety: Subject did not receive at least one application of study drug. |

Abbreviations: ITT = intent-to-treat: mITT = modified intent-to-treat: OLE = open label extension: PK= pharmacokinetic: PP = per protocol.

Note: Subjects were randomized to either Trifarotene cream HE1 100 ug/g, Trifarotene cream HE1 200 ug/g, or vehicle in the double-blind period. All subjects received Trifarotene cream HE1 200 ug/g in the open label extension period.

**Programming note:** Concatenate all reasons for exclusion with a colon.

<sup>[1]</sup> The ITT population includes all randomized subjects. The OLE ITT population includes all subjects who complete the 90-day Double-blind Treatment Period and sign the OLE informed consent.

<sup>[2]</sup> The mITT includes all subjects in the Safety population with at least 1 post baseline assessment of efficacy in the Double-blind Period. The OLE mITT population includes all subjects in the OLE Safety population with at least 1 assessment of efficacy after Visit 6.

<sup>[3]</sup> The PP Population includes subjects in the mITT population who met all inclusion criteria and no exclusion criteria, were compliant with study drug application, and who had no significant protocol deviations. The OLE PP population includes all subjects in the OLE mITT population who met all inclusion criteria and no exclusion criteria, were compliant with study drug application from baseline through EOT, and who had no significant protocol deviations throughout the study.

<sup>[4]</sup> The Safety Population includes all subjects who are randomized to treatment and receive at least 1 application of study drug in the Double-blind Period. The OLE Safety population includes all subjects who complete the 90-day Double-blind Treatment Period and receive at least 1 application of study drug in the OLE.

<sup>[5]</sup> The PK Population includes all subjects in the Safety population who have at least 1 plasma sample with quantifiable concentration.





### Listing 16.2.4.1 Subject Demographics All Subjects

| Subject<br>ID | Date of<br>Birth | Age<br>(years) | QOL<br>Questionnaires<br>Used | Sex | Child-<br>Bearing<br>Potential? | Ethnicity | Race | Weight<br>(kg) | Height<br>(cm) | BMI<br>(mg/m²) [1] |
|---|---|---|---|---|---|---|---|---|---|---|
| xxxxxx | DDMMMYYY | XX | XXXX | XXXX | No | xxxxxx | xxxxxx | XX.X | XX.X | XX.X |
| xxxxxx | DDMMMYYY | XX | XXXXXX | xxxxx | No | XXXXXXX | XXXXXX | XX.X | XX.X | XX.X |
| XXXXXX | DDMMMYYY | XX | XXXXXX | xxxxx | Yes | XXXXXXX | XXXXXX | XX.X | XX.X | XX.X |
| XXXXXX | DDMMMYYY | XX | XXXX | XXXX | No | XXXXXXX | XXXXX | XX.X | XX.X | XX.X |
| XXXXXX | DDMMMYYY | XX | XXXXXX | xxxxx | No | XXXXXXX | XXXXXX | XX.X | XX.X | XX.X |
| XXXXXX | DDMMMYYY | XX | XXXX | XXXX | Yes | XXXXXX | XXXXXX | XX.X | XX.X | XX.X |

Abbreviations: BMI = body mass index; QOL =quality of life.

Note: Subjects were randomized to either Trifarotene cream HE1 100 ug/g, Trifarotene cream HE1 200 ug/g, or vehicle in the double-blind period. All subjects received Trifarotene cream HE1 200 ug/g in the open label extension period. Height and weight are values obtained at screening.

[1] BMI = weight (kg) / [height (m)]<sup>2</sup>.





### Listing 16.2.4.2 Informed Consent and Reconsent All Subjects

Randomized Treatment: XXXXXXXXXXX

| Subject<br>ID | Screened<br>Previously? | Previous<br>Subject<br>Number | Protocol Version of Initial Consent/Assent | Date Informed<br>Consent/Assent<br>Signed | Consent to<br>PK Sub-<br>study? | Signed<br>Photographic<br>ICF? | Re-consent<br>to Later<br>Protocol<br>Version 2.0? | Date<br>Reconsent | Date of<br>Assent | Date OLE<br>Informed<br>Consent/Assent<br>Signed |
|---|---|---|---|---|---|---|---|---|---|---|
| XXXXXX | No | | X.X | DDMMMYYY | No | No | Yes | DDMMMYYY | DDMMMYYY | DDMMMYYY |
| XXXXXX | No | | X.X | DDMMMYYY | No | No | Yes | DDMMMYYY | DDMMMYYY | DDMMMYYY |
| XXXXXX | Yes | xxxxxx | X.X | DDMMMYYY | Yes | Yes | Yes | DDMMMYYY | DDMMMYYY | DDMMMYYY |
| XXXXXX | No | | X.X | DDMMMYYY | No | No | Yes | DDMMMYYY | DDMMMYYY | DDMMMYYY |
| xxxxx | No | | X.X | DDMMMYYY | No | No | Yes | DDMMMYYY | DDMMMYYY | DDMMMYYY |
| xxxxx | Yes | xxxxxx | X.X | DDMMMYYY | Yes | Yes | Yes | DDMMMYYY | DDMMMYYY | DDMMMYYY |

Abbreviations: ICF = informed consent form; OLE =open label extension; PK = pharmacokinetic.

Note: Subjects were randomized to either Trifarotene cream HE1 100 ug/g, Trifarotene cream HE1 200 ug/g, or vehicle in the double-blind period. All subjects received Trifarotene cream HE1 200 ug/g in the open label extension period.





Listing 16.2.4.3 Medical History All Subjects

| _ | System Organ Class/ | Object Deby (Objects Dept) |
|---|---|---|
| Subject ID | Preferred Term/<br>Verbatim Term | Start Date (Study Day)/<br>End Date (Study Day)/ |
| Subject ID | verbaum reim | End Date (Study Day) |
| XXXXXX | XXXXXXXXXXXXXXX/ | DDMMMYYYY (X)/ |
| | XXXXXXXXXXXXX/ | DDMMMYYYY (X) |
| | XXXXXXXXXXX | · / |
| | XXXXXXXXXXXXXXX/ | MMMYYYY/ |
| | XXXXXXXXXXXXX/ | Ongoing |
| | XXXXXXXXXXX | • • |
| | XXXXXXXXXXXXXX/ | DDMMMYYYY (X)/ |
| | XXXXXXXXXXXXX/ | Ongoing |
| | XXXXXXXXXXX | |
| XXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYYY (X)/ |
| | XXXXXXXXXXXXXXX/ | DDMMMYYYY (X) |
| | XXXXXXXXXXXXX | |

Abbreviation: MedDRA = Medical Dictionary for Regulatory Activities.

Note: Subjects were randomized to either Trifarotene cream HE1 100 ug/g, Trifarotene cream HE1 200 ug/g, or vehicle in the double-blind period. All subjects received Trifarotene cream HE1 200 ug/g in the open label extension period. Study day is calculated relative to the date of first dose of study drug. Medical history was coded using MedDRA version 21.1. Only subjects with any medical history recorded are listed.

Programming note: SOC & PT text should be in title case in table.





# Listing 16.2.5.1 Initial Study Drug Application All Subjects

| Subject ID | Was Study Drug<br>Applied? | Date of Application (Study Day) | Time of Administration | Tube Weight Before<br>Drug Application (grams) | Tube Weight After<br>Drug Application (grams) | Amount Used (grams) |
|---|---|---|---|---|---|---|
| XXXXXX | xxx | DDMMMYYYY<br>(X) | HH:MM (X) | XXX | XXX | XXX |
| xxxxx | XX; XXXXX | | | | | |
| XXXXXX | XXX | DDMMMYYYY<br>(X) | HH:MM (X) | XXX | XXX | XXX |

Note: Subjects were randomized to either Trifarotene cream HE1 100 ug/g, Trifarotene cream HE1 200 ug/g, or vehicle in the double-blind period. All subjects received Trifarotene cream HE1 200 ug/g in the open label extension period. Study day is calculated relative to the date of first dose of study drug.

**Programming Note:** If drug was not applied, concatenate reason in cell with a semicolon.





### Listing 16.2.5.2 Drug Accountability (Dispensed and Returned) All Subjects

Randomized Treatment: XXXXXXXXXXXXXXXXX

| Subject<br>ID | Study<br>Visit | Was Study Drug<br>Dispensed at this<br>Visit? | Dispensation<br>Date<br>(Study Day) | Tube Weight<br>of Tubes<br>Dispensed<br>(grams) | Kit ID<br>Dispensed | Was Study<br>Drug<br>Returned at<br>this Visit? | Return Date<br>(Study Day) | Number<br>of Tubes<br>Returned | Number<br>of Tubes<br>Returned<br>Unused | Tube<br>Weight<br>of Tubes<br>Returned<br>(grams) | Kits<br>Returned |
|---|---|---|---|---|---|---|---|---|---|---|---|
| XXXXXX | XXXXXX | xxx | DDMMMYYYY<br>(X) | XXX | XXX | XXX | DDMMMYYYY<br>(X) | XXX | XXX | XXX | XXX |
| xxxxxx | XXXXXX | XX; XXXXX | | | | XX; XXXXX | | | | | |
| XXXXXX | XXXXXX | XXX | DDMMMYYYY<br>(X) | XXX | XXX | XXX | DDMMMYYYY<br>(X) | XXX | XXX | XXX | XXX |

Note: Subjects were randomized to either Trifarotene cream HE1 100 ug/g, Trifarotene cream HE1 200 ug/g, or vehicle in the double-blind period. All subjects received Trifarotene cream HE1 200 ug/g in the open label extension period. Study day is calculated relative to the date of first dose of study drug.

Programming Note: If drug was not dispensed/returned at a visit, concatenate reason in cell with a semicolon.





Listing 16.2.5.3 Subject Diary All Subjects

Randomized Treatment: XXXXXXXXXXXXXXXXX

| Subject<br>ID | Study<br>Visit | Was Diary Data<br>Collected at this<br>Visit? | Dose<br>Number | Date of Dose<br>(Study Day) | Day of the<br>Week | Time Drug<br>Taken | Areas of Skin<br>Treated | Areas Not<br>Treated | Reasons | Cream<br>Reaction |
|---|---|---|---|---|---|---|---|---|---|---|
| xxxxxx | XXXXXX | XXX | XX | DDMMMYYYY<br>(X) | XXXXXXX | HH:MM | xxxxxxx | xxxxxxx | xxxxxxx | xxxxxxx |
| | | | | () | | | | XXXXXXX | XXXXXXX | XXXXXXX |
| XXXXXX | xxxxx | XX; XXXXX | | | | | | | | |
| XXXXXX | XXXXXX | XXX | XX | DDMMMYYYY | XXXXXX | HH:MM | XXXXXXX | XXXXXXX | xxxxxxx | xxxxxxx |
| | | | | (X) | | | | XXXXXXXX | XXXXXXXX | XXXXXXXX |
| | | | | | | | | XXXXXXXX | XXXXXXXX | XXX |

Note: Subjects were randomized to either Trifarotene cream HE1 100 ug/g, Trifarotene cream HE1 200 ug/g, or vehicle in the double-blind period. All subjects received Trifarotene cream HE1 200 ug/g in the open label extension period. Study day is calculated relative to the date of first dose of study drug.

**Programming Note:** If diary data was not collected at this visit, concatenate reason in cell with a semicolon. Include all body areas not treated. If body area not treated or reason is other, concatenate specify field in cell with a semicolon.





# Listing 16.2.5.4.1 Pharmacokinetic Sample Collection PK Population

### Randomized Treatment: XXXXXXXXXXXXXXXXX

| Subject ID | Was the Sample Collected? | Reason | Date Collected<br>(Study Day) |
|---|---|---|---|
| xxxxxx | XXXXXXX<br>XXXXXXX<br>XXXXXXX | XXXXXXX<br>XXXXXXX<br>XXXXXXX | DDMMMYYYY (X)<br>DDMMMYYYY (X)<br>DDMMMYYYY (X) |
| | XXXXXXX | XXXXXX | DDMMMYYYY (X) |
| XXXXXX | xxxxxx | xxxxxx | DDMMMYYYY (X) |

Abbreviation: PK = pharmacokinetic.

Note: Subjects were randomized to either Trifarotene cream HE1 100 ug/g, Trifarotene cream HE1 200 ug/g, or vehicle in the double-blind period. All subjects received Trifarotene cream HE1 200 ug/g in the open label extension period. Study day is calculated relative to the date of first dose of study drug.





# Listing 16.2.5.4.2 Pharmacokinetic Sample Collection (Substudy) PK Population

| Subject ID | Initial Study Drug<br>Application? | Date Collected<br>(Study Day) | Time | Timepoints | Sample Collected? | Date/Time Collected<br>(Study Day) |
|---|---|---|---|---|---|---|
| xxxxxx | XXX | DDMMMYYYY (X) | HH:MM | XXXXXXX | XXX | DDMMMYYYY/HH:MM (X) |
| | XXX | DDMMMYYYY (X) | HH:MM | XXXXXXX | XXX | DDMMMYYYY/HH:MM (X) |
| | XX | DDMMMYYYY (X) | HH:MM | XXXXXXX | XXX | DDMMMYYYY/HH:MM (X) |
| | XX | DDMMMYYYY (X) | HH:MM | XXXXXXX | XXX | DDMMMYYYY/HH:MM (X) |
| XXXXXX | XX | DDMMMYYYY (X) | HH:MM | xxxxxx | xxx | DDMMMYYYY/HH:MM (X) |

Abbreviation: PK = pharmacokinetic.

Note: Subjects were randomized to either Trifarotene cream HE1 100 ug/g, Trifarotene cream HE1 200 ug/g, or vehicle in the double-blind period. All subjects received Trifarotene cream HE1 200 ug/g in the open label extension period. Study day is calculated relative to the date of first dose of study drug.

**Programming Note:** If sample was not collected, concatenate reason in cell with a semicolon.





# Listing 16.2.5.4.3 Pharmacokinetic Concentrations PK Population

### 

| | | Time In-Clinic Dose | | | Date/Time Sample<br>Collected | Concentration |
|---|---|---|---|---|---|---|
| Subject ID | Study Visit | Taken | Time Point | Was Sample Collected? | (Study Day) | (unit) |
| XXXXXX | xxxxxx | HH:MM | xxxxxx | Yes | DDMMMYYYY/HH:MM<br>(X) | X.XX |
| | XXXXXXX | HH:MM | XXXXXXX | Yes | DDMMMYYYY/HH:MM | X.XX |
| | xxxxxx | HH:MM | XXXXXX | Yes | (X)<br>DDMMMYYYY/HH:MM<br>(X) | X.XX |
| | XXXXXXX | HH:MM | XXXXXX | No; XXXXXXXX | . , | |
| XXXXXX | xxxxxx | нн:мм | XXXXXXX | Yes | DDMMMYYYY/HH:MM<br>(X) | X.XX |

Abbreviation: BLQ = below the limit of quantification; PK = pharmacokinetic.

Note: Subjects were randomized to either Trifarotene cream HE1 100 ug/g, Trifarotene cream HE1 200 ug/g, or vehicle in the double-blind period. All subjects received Trifarotene cream HE1 200 ug/g in the open label extension period. Study day is calculated relative to the date of first dose of study drug. Any results that are BLQ (i.e., <0.xx) are displayed as BLQ in the listing.





# Listing 16.2.5.4.4 Pharmacokinetic Calculated Parameters PK Population

Randomized Treatment: XXXXXXXXX

| Subject ID | AUC <sub>0-t</sub><br>(unit) | C <sub>max</sub><br>(unit) | T <sub>max</sub><br>(unit) | AUC <sub>0-inf</sub><br>(unit) | t <sub>1/2</sub><br>(unit) | λ <sub>z</sub><br>(unit) |
|---|---|---|---|---|---|---|
| XXXXX | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX |
| XXXXX | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX |

Abbreviation: AUC = area under the plasma concentration-time curve; Cmax = peak plasma concentration; CV = coefficient of variation;  $\lambda_z$  = apparent terminal phase rate constant. PK = pharmacokinetic; SD = standard deviation; t1/2= first order termination half-life; Tmax = time of Cmax.

Note: Subjects were randomized to either Trifarotene cream HE1 100 ug/g, Trifarotene cream HE1 200 ug/g, or vehicle in the double-blind period. All subjects received Trifarotene cream HE1 200 ug/g in the open label extension period. Study day is calculated relative to the date of first dose of study drug. 0-t represents time from 0 to the time of the last quantifiable plasma concentration.

**Programming note**: the number of decimal places depends on the raw data. The above parameters are expected, however the final parameters provided by the pharmacokineticist will be listed.





### Listing 16.2.6.1 Investigator's Global Assessment (IGA) All Subjects

### 

| Subject<br>D | Was<br>Assessment<br>Performed? | Study Visit | Assessment Date<br>(Study Day) | Body Area [1] | Result | Baseline [2] | CFB [3] | % CFB [4] | Successful<br>Resolution of<br>LI? |
|---|---|---|---|---|---|---|---|---|---|
| xxxxx | XXX | XXXXXX | DDMMMYYYY | xxxxxx | Х | Х | Х | Х | XXX |
| | | | (XX) | XXXXXX | X | X | Χ | X | XX |
| xxxxx | XXX | xxxxxx | DDMMMYYYY<br>(XX) | | X | X | X | Χ | XXX |
| | | | , | | XX | XX | XX | XX | XX |
| | | | | | XX | XX | XX | XX | XXX |
| | | | | | XX | XX | XX | XX | XXX |

Abbreviations: CFB = change from baseline; IGA = Investigator's Global Assessment; LI = Lamellar Ichthyosis.

Note: Subjects were randomized to either Trifarotene cream HE1 100 ug/g, Trifarotene cream HE1 200 ug/g, or vehicle in the double-blind period. All subjects received Trifarotene cream HE1 200 ug/g in the open label extension period. Study day is calculated relative to the date of first dose of study drug. The 5-point (0 - 4) IGA is a measure of disease severity which considers both scaling and roughness. Higher IGA scores represent more severe disease. Successful resolution is defined as clear/almost clear overall and at least a 2-grade change from Baseline on the 5-point (0 - 4) IGA scale.

- [1] Body area only for subjects enrolled under protocol version 1.0.
- [2] Baseline is defined as the last non-missing assessment recorded prior to the first dose of treatment in the Double-blind Period.
- [3] CFB is calculated as Result Baseline.
- [4] % CFB is calculated as Change from baseline / Result at baseline \* 100.

Programming note: If assessment was not performed, concatenate reason with a semicolon. CFB, % CFB and Successful Resolution of LI columns will not be populated for Baseline rows.





### Listing 16.2.6.2 Visual Index for Ichthyosis (VIIS) All Subjects

| Subject ID | Was Assessment Performed? | Study Visit | Assessment Date (Study Day) | Body Area | Scaling Score | Baseline [2] | CFB [3] | % CFB [4] |
|---|---|---|---|---|---|---|---|---|
| xxxxxx | XXX | XXXXXX | DDMMMYYYY<br>(XX) | Chest/Abdomen | X | X | X | X |
| | | | , | Back | Χ | Χ | X | X |
| | | | | Arms | X | X | Χ | Χ |
| | | | | Legs | XX | XX | XX | XX |
| | | | | Total | XX | XX | XX | XX |

XXXXXX XX; XXXXX

Abbreviations: CFB = change from baseline; VIIS = .Visual Index for Ichthyosis.

Note: Subjects were randomized to either Trifarotene cream HE1 100 ug/g, Trifarotene cream HE1 200 ug/g, or vehicle in the double-blind period. All subjects received Trifarotene cream HE1 200 ug/g in the open label extension period. Study day is calculated relative to the date of first dose of study drug. The VIIS is scored on a 5-point (0 - 4) scale by body area (chest/abdomen, back, legs, and arms). Higher VIIS scores represent worse scaling.

- [1] Baseline is defined as the last non-missing assessment recorded prior to the first dose of treatment in the Double-blind Period.
- [2] CFB is calculated as Result Baseline.
- [3] % CFB is calculated as Change from baseline / Result at baseline \* 100.





### Listing 16.2.6.3 Roughness Assessment All Subjects

#### 

| Was Assessment Performed? | Study Visit | Assessment Date<br>(Study Day) | Overall Score for<br>Roughness | Baseline [2] | CFB [3] | % CFB [4] | 2-grade<br>CFB? |
|---|---|---|---|---|---|---|---|
| xxx | xxxxxx | DDMMMYYYY<br>(XX) | X | Х | X | X | XXX |
| | | (701) | X | X | Χ | X | XX |
| XXX | xxxxx | DDMMMYYYY<br>(XX) | Х | X | X | X | XXX |
| | | ( / | XX | XX | XX | XX | XX |
| | | | XX | XX | XX | XX | XXX |
| | | | XX | XX | XX | XX | XXX |
| | Performed? XXX | Performed? Study Visit XXX XXXXXX | Performed? Study Visit (Study Day) XXX XXXXX DDMMMYYYY (XX) | Performed? Study Visit (Study Day) Roughness XXX XXXXXX DDMMMYYYY X (XX) X XXXXXX DDMMMYYYY X (XX) XX XXX XXXXX DDMMMYYYY X (XX) XX XX | Performed? Study Visit (Study Day) Roughness Baseline [2] XXX XXXXXXX DDMMMYYYY X X XXX XXXXXXX DDMMMYYYY X X XXX XXXXXXX DDMMMYYYYY X X XXX XXX XX XX XXX XX XX XX XXX XX XX XX | Performed? Study Visit (Study Day) Roughness Baseline [2] CFB [3] XXX XXXXXXX DDMMMYYYY X X X XXX XX X X X XXX XXXXXXX DDMMMYYYY X X X XXX XX XX XX XX XXX XX XX XX XXX XX XX XX XXX XX XX XX | Performed? Study Visit (Study Day) Roughness Baseline [2] CFB [3] % CFB [4] XXX XXXXXXX DDMMMYYYY X X X X XXX XX X X X X XXX XXXXXXX DDMMMYYYY X X X X XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX |

Abbreviations: CFB = change from baseline.

Note: Subjects were randomized to either Trifarotene cream HE1 100 ug/g, Trifarotene cream HE1 200 ug/g, or vehicle in the double-blind period. All subjects received Trifarotene cream HE1 200 ug/g in the open label extension period. Study day is calculated relative to the date of first dose of study drug. The individual score for roughness measures the amount of roughness of the skin overall and is scored on a 5-point (0 - 4) scale. Higher scores indicate more severe roughness.

- [1] Baseline is defined as the last non-missing assessment recorded prior to the first dose of treatment in the Double-blind Period.
- [2] CFB is calculated as Result Baseline.
- [3] % CFB is calculated as Change from baseline / Result at baseline \* 100.





# Listing 16.2.6.4 Palm/Sole Assessment All Subjects

#### 

| Subject ID | Was Assessment Performed? | Study Visit | Assessment Date (Study Day) | Body Area | Assessment | Baseline [2] | CFB [3] | % CFB [4] |
|---|---|---|---|---|---|---|---|---|
| xxxxxx | XXX | xxxxxx | DDMMMYYYY | Palms | X | X | X | X |
| | | | (XX) | Soles | X | Х | X | X |
| xxxxx | xxx | xxxxx | DDMMMYYYY | Palms | XX | XX | XX | XX |
| | | | (XX) | Soles | XX | XX | XX | XX |
| XXXXXX | XX; XXXXX | | | | | | | |

Abbreviations: CFB = change from baseline.

Note: Subjects were randomized to either Trifarotene cream HE1 100 ug/g, Trifarotene cream HE1 200 ug/g, or vehicle in the double-blind period. All subjects received Trifarotene cream HE1 200 ug/g in the open label extension period. Study day is calculated relative to the date of first dose of study drug. Thickening of the skin on the palms and soles will be measured on a 5-point (0 - 4) scale. Higher scores indicate more severe thickening.

- [1] Baseline is defined as the last non-missing assessment recorded prior to the first dose of treatment in the Double-blind Period.
- [2] CFB is calculated as Result Baseline.
- [3] % CFB is calculated as Change from baseline / Result at baseline \* 100.





# Listing 16.2.6.5.1 Quality of Life per Dermatology Life Quality Index (DLQI) All Subjects

| Subject ID | Was Assessment<br>Performed? | Study Visit | Assessment Date (Study Day) | Item | Score | Baseline [2] | CFB [3] | % CFE<br>[4] |
|---|---|---|---|---|---|---|---|---|
| xxxxx | XXX | xxxxxx | DDMMMYYYY<br>(XX) | Over the last week, how itchy, sore, painful or stinging has your skin been? | X | X | X | X |
| | | | () | Over the last week, how embarrassed or self conscious have you been because of your skin? | X | X | X | X |
| | | | | 10. Over the last week, how much of a problem has the treatment for your skin been, for example by making your home | XX | XX | xx | xx |
| | | | | messy, or by taking up time? Total Score | XX | XX | XX | XX |

XXXXXX XX; XXXXX

Abbreviations: CFB = change from baseline; DLQI = Quality of Life per Dermatology Life Quality Index.

Note: Subjects were randomized to either Trifarotene cream HE1 100 ug/g, Trifarotene cream HE1 200 ug/g, or vehicle in the double-blind period. All subjects received Trifarotene cream HE1 200 ug/g in the open label extension period. Study day is calculated relative to the date of first dose of study drug. DLQI total score is derived as the sum of the 10 individual item scores, with a range of 0 to 30. Higher scores indicate poorer quality of life.

- [1] Baseline is defined as the last non-missing assessment recorded prior to the first dose of treatment in the Double-blind Period.
- [2] CFB is calculated as Result Baseline.
- [3] % CFB is calculated as Change from baseline / Result at baseline \* 100.

Programming note: If assessment was not performed, concatenate reason with a semicolon. CFB and % CFB columns will not be populated for Baseline rows.

Listing 16.2.6.5.2

Quality of Life per Children's Dermatology Life Quality Index (cDLQI)

All Subjects

#### Same shell as Listing 16.2.6.5.1

**Programming note:** If update to cDLQI throughout footnotes and abbreviations.

AD-ST-33.05 Effective date: 22-Jan-2018





### Listing 16.2.6.6 Fissuring Assessment All Subjects

Randomized Treatment: XXXXXXXXXXXXXXXXX

| Subject ID | Was Assessment Performed? | Study Visit | Assessment Date (Study Day) | Fissures Present on Palms or Soles? | Body Area | Number of<br>Fissures | Fissure Pain Level |
|---|---|---|---|---|---|---|---|
| xxxxxx | xxx | XXXXXX | DDMMMYYYY | XXX | Palms | XX | xxxxx |
| | | | (XX) | | Soles | XX | XXXXX |
| XXXXXX | XXX | xxxxxx | DDMMMYYYY | xxx | Palms | XX | XXXXXXX |
| | | | (XX) | | Soles | XX | XXXX |
| XXXXX | XX; XXXXX | | | | | | |

Note: Subjects were randomized to either Trifarotene cream HE1 100 ug/g, Trifarotene cream HE1 200 ug/g, or vehicle in the double-blind period. All subjects received Trifarotene cream HE1 200 ug/g in the open label extension period. Study day is calculated relative to the date of first dose of study drug.

Programming note: If assessment was not performed, concatenate reason with a semicolon.





Listing 16.2.6.7 Ectropion Score All Subjects

#### 

| Subject ID | Was Assessment Performed? | Study Visit | Assessment Date<br>(Study Day) | Item | Score | Baseline [2] | CFB [3] | % CFB [4] |
|---|---|---|---|---|---|---|---|---|
| XXXXXX | xxx | xxxxx | DDMMMYYYY<br>(XX) | Lateral apposition | XX | XX | XX | XX |
| | | | , | Medial apposition | XX | XX | XX | XX |
| | | | | Scleral show | XX | XX | XX | XX |
| | | | | Conjunctival show | XX | XX | XX | XX |
| | | | | Excess tear film | XX | XX | XX | XX |
| | | | | Redness of the eye | XX | XX | XX | XX |
| | | | | Round canthus | XX | XX | XX | XX |
| | | | | Punctum lacrimate | XX | XX | XX | XX |
| | | | | Total Score | XX | XX | XX | XX |

Abbreviations: CFB = change from baseline.

Note: Subjects were randomized to either Trifarotene cream HE1 100 ug/g, Trifarotene cream HE1 200 ug/g, or vehicle in the double-blind period. All subjects received Trifarotene cream HE1 200 ug/g in the open label extension period. Study day is calculated relative to the date of first dose of study drug. Ectropion total score is derived as the sum of the 8 individual item scores (lateral apposition, medial apposition, scleral show, conjunctival show, excess tear film, redness of the eye, round canthus, punctum lacrimale), with a range of 0 to 8. Each individual item is scored 0 (nonaffected/no/invisible), 0.5 (<= 1 mm/emerging), or 1 (affected/yes/visible). Higher scores indicates worse ectropion.

- [1] Baseline is defined as the last non-missing assessment recorded prior to the first dose of treatment in the Double-blind Period.
- [2] CFB is calculated as Result Baseline.
- [3] % CFB is calculated as Change from baseline / Result at baseline \* 100.





Listing 16.2.6.8 EQ-5D All Subjects

#### 

| | Was Assessment | | Assessment Date | | | | | |
|---|---|---|---|---|---|---|---|---|
| Subject ID | Performed? | Study Visit | (Study Day) | Item | Score | Baseline [2] | CFB [3] | % CFB [4] |
| XXXXXX | XXX | XXXXXX | DDMMMYYYY<br>(XX) | Mobility | XX | XX | XX | XX |
| | | | , | Self-care | XX | XX | XX | XX |
| | | | | Usual Activities | XX | XX | XX | XX |
| | | | | Pain/Discomfort | XX | XX | XX | XX |
| | | | | Anxiety Depression | XX | XX | XX | XX |
| | | | | Your Health Today | XX | XX | XX | XX |
| xxxxx | XX; XXXXX | | | | | | | |

Abbreviations: CFB = change from baseline; VAS = visual analog scale.

Note: Subjects were randomized to either Trifarotene cream HE1 100 ug/g, Trifarotene cream HE1 200 ug/g, or vehicle in the double-blind period. All subjects received Trifarotene cream HE1 200 ug/g in the open label extension period. Study day is calculated relative to the date of first dose of study drug. The EQ-5D is a measure of health related quality of life. The EQ-5D consists of a descriptive system and the EQ visual analog scale (VAS). The EQ-5D-5L is intended for use in adult subjects. The descriptive system comprises 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The EQ VAS records the subject's self-rated health on a vertical 0-100 VAS.

- [1] Baseline is defined as the last non-missing assessment recorded prior to the first dose of treatment in the Double-blind Period.
- [2] CFB is calculated as Result Baseline.
- [3] % CFB is calculated as Change from baseline / Result at baseline \* 100.





Listing 16.2.7.1 Adverse Events All Subjects

#### Randomized Treatment: XXXXXXXXXXXXXXXXX

| Subject<br>ID | TEAE? [1] | System Organ Class/<br>Preferred Term/<br> Verbatim Term | Start Date/Time (Study Day)/<br>End Date/Time (Study Day) | | Outcome | Serious?/<br>Criteria Met | Action Taken/<br>Other Action Taken? |
|---|---|---|---|---|---|---|---|
| XXXXX | xxx | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYYY/HH:MM (X)/<br>DDMMMYYYY/HH:MM (X) | XXXXXXXX/<br>XXXXXXXXXX | xxxxxxxx | XX | XXXXXXXXX/<br>XXXXXXXXX |
| XXXXX | XX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYYY/HH:MM (X)/<br>DDMONYYYY/HH:MM (X) | XXXXXXXXX/<br>XXXXXXXXXX | xxxxxxxx | xx | XXXXXXXXX/<br>XXXXXXXXX |
| | XXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYYY/HH:MM (X)/<br>Ongoing | XXXXXXXXX/<br>XXXXXXXXXX | XXXXXXXXX/ | XXX/<br>XXXXXXXXX | XXXXXXXXX/<br>XXXXXXXXX |

Abbreviations: AE = adverse event; MedDRA = Medical Dictionary for Regulatory Activities; TEAE = treatment emergent adverse event.

Note: Subjects were randomized to either Trifarotene cream HE1 100 ug/g, Trifarotene cream HE1 200 ug/g, or vehicle in the double-blind period. All subjects received Trifarotene cream HE1 200 ug/g in the open label extension period. Study day is calculated relative to the date of first dose of study drug. AEs were coded using MedDRA version 21.1.
[1] A TEAE is any AE with an onset at the time of or following the start of treatment with study drug through the Follow-up Visit or Early Termination Visit, whichever occurs first. This will include any AE starting prior to the start of treatment but increasing in severity or relationship at the time of, or following, the start of treatment with study drug through the Follow-up Visit or Early Termination Visit, whichever occurs first.

Programming note: If time missing, display "- -:- -". If Serious? is Yes, concatenate all serious criteria marked as Yes with a semicolon. If no events meet the criteria for display, present "No events are reported." SOC & PT text should be in proper case in table.





### Listing 16.2.8.1 Laboratory Data: Clinical Chemistry All Subjects

#### Randomized Treatment: XXXXXXXXXXX

| Subject ID | Parameter<br>(unit) | Study<br>Visit | Date/Time of<br>Assessment<br>(Study Day) | Standard<br>Results | Standard<br>Reference<br>Range<br>[1] | Standard<br>Reference Range<br>Flag | CFB<br>[2] | %CFB<br>[3] | Accession<br>Number | Comments |
|---|---|---|---|---|---|---|---|---|---|---|
| XXXXX | Albumin (unit) | XXXXXX | DDMMMYYYY/ | XX | XX – YY | | | | XXXXXX | |
| | | 100000 | HH:MM (X) | | | 1007 | 1001 | | ,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,, | |
| | | XXXXXX | DDMMMYYYY/<br>HH:MM (X) | XX | XX – YY | XXX | XXX | XXX | XXXXXXX | |
| | | XXXXXX | DDMMMYYYY/<br>HH:MM (X) | XX | XX – YY | | XXX | XXX | XXXXXX | |
| | | XXXXXX | | ND | | | | | | XXXXXXX |
| | | XXXXXX | DDMMMYYYY/<br>HH:MM (X) | XX | XX – YY | | XXX | XXX | XXXXXXX | |

Abbreviations: AE = adverse event; AL = abnormal-low; AH = abnormal-high; CFB = change from baseline; CS = clinically significant; NCS = not clinically significant; ND = not done

Note: Subjects were randomized to either Trifarotene cream HE1 100 ug/g, Trifarotene cream HE1 200 ug/g, or vehicle in the double-blind period. All subjects received Trifarotene cream HE1 200 ug/g in the open label extension period. Study day is calculated relative to the date of first dose of study drug.

- [1] Reference range is used to identify potentially clinically significant laboratory values.
- [2] Baseline is defined as the last non-missing assessment recorded prior to the first dose of treatment in the Double-blind Period.
- [2] CFB is calculated as Result Baseline.
- [3] % CFB is calculated as Change from baseline / Result at baseline \* 100.

**Programming note:** update abbreviations to reflect actual data. If test was not done, set results to ND. For reference range flag, concatenate AL or AH with clinical significant like "XX-YY" (e.g., AL-CS). CFB and %CFB columns will be blank for Baseline. Include all parameters.





Listing 16.2.8.2 Laboratory Data: Hematology All Subjects

Same shell as Listing 16.2.8.1

Listing 16.2.8.3 Laboratory Data: Coagulation All Subjects

Same shell as Listing 16.2.8.1

Listing 16.2.8.4 Laboratory Data: Urinalysis All Subjects

Same shell as Listing 16.2.8.1

Listing 16.2.8.5 Laboratory Data: Serology All Subjects

Same shell as Listing 16.2.8.1





## Listing 16.2.8.6 Laboratory Data: Pregnancy Tests All Subjects

Randomized Treatment: XXXXXXXXXXXX

| Subject ID | Sample Type | Was Sample for Urine/Serum Pregnancy Test Collected? | Date of<br>Collection<br>(Study Day) | Result |
|---|---|---|---|---|
| XXXXX | xxxxxx | XXX | DDMMMYYYY<br>(X) | xxxxxxx |
| XXXXX | XXXXXX | XXX | DDMMMYYYY<br>(X) | xxxxxxx |
| XXXXX | XXXXXX | XX; XXXXX | | |

Note: Subjects were randomized to either Trifarotene cream HE1 100 ug/g, Trifarotene cream HE1 200 ug/g, or vehicle in the double-blind period. All subjects received Trifarotene cream HE1 200 ug/g in the open label extension period. Study day is calculated relative to the date of first dose of study drug.

Programming note: If sample not collected, concatenate reason in cell with a semicolon.





Listing 16.2.9.1 Vital Signs All Subjects

#### Randomized Treatment: XXXXXXXXXXX

| Subject ID | Parameter (unit) | Study<br>Visit | Date/Time Collected<br>(Study Day) | Result | CFB [2] | %CFB [3] |
|---|---|---|---|---|---|---|
| XXXXX | Pulse (bpm) | xxxxxx | DDMMMYYYY/<br>HH:MM (X) | XX | | |
| | | XXXXXX | DDMMMYYYY/<br>HH:MM (X) | XX | XXX | XXX |
| | | xxxxx | DDMMMYÝÝY/<br>HH:MM (X) | XX | XXX | XXX |
| XXXXX | XXXXXX | XXXXXX | DDMMMYYYY/<br>HH:MM (X) | XX | XXX | XXX |

Abbreviations: CFB = change from baseline.

Note: Subjects were randomized to either Trifarotene cream HE1 100 ug/g, Trifarotene cream HE1 200 ug/g, or vehicle in the double-blind period. All subjects received Trifarotene cream HE1 200 ug/g in the open label extension period. Study day is calculated relative to the date of first dose of study drug.

[1] Baseline is defined as the last non-missing assessment recorded prior to the first dose of treatment in the Double-blind Period.

[2] CFB is calculated as Result – Baseline.

[3] % CFB is calculated as Change from baseline / Result at baseline \* 100.

Programming note: CFB and %CFB columns will be blank for Baseline. Include all parameters.





### Listing 16.2.9.2 12-Lead Electrocardiogram All Subjects

Randomized Treatment: XXXXXXXXXXX

| Subject ID | Parameter (unit) | Study<br>Visit | Timepoint | Was ECG Performed at this Time point? | Date/Time Collected<br>(Study Day) | Result | CFB [2] | %CFB [3] |
|---|---|---|---|---|---|---|---|---|
| XXXXX | Pulse (bpm) | xxxxx | xxxxx | XX | DDMMMYYYY/<br>HH:MM (X) | XX | | |
| | | XXXXXX | XXXXXX | XX | DDMMMYYYY/<br>HH:MM (X) | XX | XXX | XXX |
| | | XXXXXX | XXXXXX | XX | DDMMMYYYY/<br>HH:MM (X) | XX | XXX | XXX |
| XXXXX | XXXXXX | XXXXXX | XXXXXX | XX | DDMMMYYYY/<br>HH:MM (X) | XX | XXX | XXX |

Abbreviations: CFB = change from baseline; ECG= electrocardiogram.

Note: Subjects were randomized to either Trifarotene cream HE1 100 ug/g, Trifarotene cream HE1 200 ug/g, or vehicle in the double-blind period. All subjects received Trifarotene cream HE1 200 ug/g in the open label extension period. Study day is calculated relative to the date of first dose of study drug.

[1] Baseline is defined as the last non-missing assessment recorded prior to the first dose of treatment in the Double-blind Period.

[2] CFB is calculated as Result – Baseline.

Programming note: If ECG was not performed, concatenate reason in cell with a semicolon.

<sup>[3] %</sup> CFB is calculated as Change from baseline / Result at baseline \* 100.





### Listing 16.2.9.3 Local Tolerability Assessments All Subjects

### Randomized Treatment: XXXXXXXXXXXXXXXX

| Subject ID | Was Assessment Collected? | Study Visit | Date Assessment Collected (Study Day) | Body Area | Assessment | Score |
|---|---|---|---|---|---|---|
| xxxxx | XXX | XXXXXXX | DDMMMYYYY<br>(X) | Face/Neck | Erythema | xxxxx |
| | | | ` ' | | Stinging/Burning | XXXXX |
| | | | | xxxxx | Pruritus<br>XXXXXXXX | XXXXX |
| | | | | XXXXX | XXXXXXXX | XXXXX |

Note: Subjects were randomized to either Trifarotene cream HE1 100 ug/g, Trifarotene cream HE1 200 ug/g, or vehicle in the double-blind period. All subjects received Trifarotene cream HE1 200 ug/g in the open label extension period. Study day is calculated relative to the date of first dose of study drug.

Programming note: If assessment was not collected, concatenate reason in cell with a semicolon.





### Listing 16.2.9.4 Physical Examination All Subjects

| Subject<br>ID | Was Exam<br>Performed? | Study<br>Visit | Exam Date<br>(Study Day) | Body System | Result | Abnormal<br>Findings | Clinically<br>Significant? |
|---|---|---|---|---|---|---|---|
| טו | Periormed? | VISIL | (Study Day) | Body System | Result | rindings | Significant |
| XXXXXX | XXX | XXXXXX | DDMMMYYYY<br>(-X) | General Appearance | Normal | | |
| | | | , , | Integumentary<br>Head, Ears, Eyes,<br>Nose, Throat | Abnormal<br>Normal | XXXXXXX | No |

Note: Subjects were randomized to either Trifarotene cream HE1 100 ug/g, Trifarotene cream HE1 200 ug/g, or vehicle in the double-blind period. All subjects received Trifarotene cream HE1 200 ug/g in the open label extension period. Study day is calculated relative to the date of first dose of study drug.

Programming note: if physical examination was not performed, concatenate reason with a semicolon.





# Listing 16.2.9.5 Prior and Concomitant Medications All Subjects

Randomized Treatment: XXXXXXXXXXXXXXXXX

| | Prior/<br>Concomitant | | ATC Class (Level 4)/ Preferred Term (ATC Level 5)/ | Start Date/Time (Study Day)/ | | Route/ |
|---|---|---|---|---|---|---|
| Subject ID | [1] | Indication | Verbatim Term | End Date/Time (Study Day) | Dose (unit) | Frequency |
| XXXXXX I | Prior | XXXXXXX | XXXXXXXXXXXXXXX/<br>XXXXXXXXXXXXXX/<br>XXXXXXX | DDMMMYYYY/hh:mm (X)/<br>DDMMMYYYY/hh:mm (X) | XXX (XXX) | XXXXXXXX/<br>XXXXXXX |
| | Both | XXXXXXX | XXXXXXXXX/<br>XXXXXXXXXXXXXXX/<br>XXXXXXXXXX | MMMYYYY/: (X)/<br>Ongoing | XXX (XXX) | XXXXXXX/<br>XXXXXXX |
| | Concomitant | XXXXXXX | XXXXXXXXX/<br>XXXXXXXXXXXXXXX/<br>XXXXXXXXXX | DDMMMYYYY/hh:mm (X)/<br>DDMMMYYYY/hh:mm (XX) | XXX (XXX) | XXXXXXX/<br>XXXXXXX |

Abbreviations: ATC = anatomic therapeutic chemical; NA = not applicable; WHO-DDE = World Health Organization-Drug Dictionary Enhanced. Note: Subjects were randomized to either Trifarotene cream HE1 100 ug/g, Trifarotene cream HE1 200 ug/g, or vehicle in the double-blind period. All subjects received Trifarotene cream HE1 200 ug/g in the open label extension period. Study day is calculated relative to the date of first dose of study drug. Medications were coded using WHO-DDE version March 2019.

[1] "Prior" medications are all medications that were started before the first dose of study medication. "Concomitant" medications are medications continuing or starting after the first dose through the end of study. "Both" indicates medication that was started before the first dose and continued during the study.

**Programming note:** If Dose unit, Route or Frequency is Other, display other specify text only (i.e., do not display "Other: XXXXXX" but just "XXXXXX"). Sort by subject, start date/time, end date/time, ATC level 4 & PT. ATC & PT text should be in title case in table, as shown in the shell. Ensure proper WHO-DDE version is printed in footnote.





Listing 16.2.9.6 Photography All Subjects

Randomized Treatment: XXXXXXXXXXXXXXXXX

| Subject ID | Was Photography Collected? | Collection Date<br>(Study Day) |
|------------|----------------------------|--------------------------------|
| xxxxx | XXX | DDMMMYYYY (XX) |
| xxxxx | XXX | DDMMMYYYY (XX) |
| xxxxxx | xxx | DDMMMYYYY (XX) |
| XXXXXX | xxx | DDMMMYYYY (XX) |
| XXXXXX | xx | |
| xxxxx | XXX | DDMMMYYYY (XX) |

Note: Subjects were randomized to either Trifarotene cream HE1 100 ug/g, Trifarotene cream HE1 200 ug/g, or vehicle in the double-blind period. All subjects received Trifarotene cream HE1 200 ug/g in the open label extension period. Study day is calculated relative to the date of first dose of study drug.





### Listing 16.2.9.7 Trial Continuation All Subjects

Randomized Treatment: XXXXXXXXXXXXXXXX

| | • | Next Visit? | Drug Administration? | Continuing to OLE? |
|--------|--------|-------------|----------------------|--------------------|
| XXXXXX | XXXXXX | XXX | XXX | XXX |
| XXXXXX | XXXXXX | XXX | XXX | XXX |
| XXXXXX | XXXXXX | XXX | XXX | XXX |
| XXXXXX | XXXXXX | XXX | XXX | XXX |
| XXXXXX | XXXXXX | XX | XX | XX |
| xxxxx | XXXXXX | XXX | XXX | XXX |

Abbreviation: OLE = open label extension.

Note: Subjects were randomized to either Trifarotene cream HE1 100 ug/g, Trifarotene cream HE1 200 ug/g, or vehicle in the double-blind period. All subjects received Trifarotene cream HE1 200 ug/g in the open label extension period.





### Listing 16.2.9.8 Telephone Contact All Subjects

Randomized Treatment: XXXXXXXXXXXXXXXX

| Subject ID | Study Visit | Contacted to Assess New AEs/SAEs? | Contact Date<br>(Study Day) | Report Any New or Worsening<br>AEs/SAEs? | Report Any New Concomitant Medications? |
|---|---|---|---|---|---|
| XXXXXX | xxxxxx | XXX | DDMMMYYYY (XX) | XXX | xxx |
| XXXXX | XXXXXX | XXX | DDMMMYYYY (XX) | XXX | XXX |
| XXXXX | XXXXXX | XXX | DDMMMYYYY (XX) | XXX | XXX |
| XXXXXX | XXXXXX | XXX | DDMMMYYYY (XX) | XXX | XXX |
| XXXXXX | XXXXXX | XX; XXXXX | | | |
| XXXXXX | XXXXXX | XXX | DDMMMYYYY (XX) | XXX | XXX |

Abbreviation: AE = adverse event; OLE = open label extension; SAE = serious adverse event.

Note: Subjects were randomized to either Trifarotene cream HE1 100 ug/g, Trifarotene cream HE1 200 ug/g, or vehicle in the double-blind period. All subjects received Trifarotene cream HE1 200 ug/g in the open label extension period. Study day is calculated relative to the date of first dose of study drug.

Listing 16.2.9.9 COVID-19 Impact Log All Subjects

Programming Note: The structure of this listing will be determined prior to database lock, when the log is finalized.





## 14.4. Planned Figure Shells



# **Appendix 1: Premier Research Library of Abbreviations**

| Abbreviation | Definition |
|--------------|---------------------------------|
| AE | adverse event |
| AESI | adverse events special interest |
| AIC | Akaike information criterion |
| ANCOVA | analysis of covariance |
| ATC | anatomical therapeutic chemical |
| BLQ | beneath limit of quantification |
| BMI | body mass index |
| BP | Blood pressure |
| bpm | Beats per minute |
| CFB | Change from baseline |
| CFR | code of federal regulations |
| CI | confidence intervals |
| CRF | case report form |
| CRO | contract research organization |
| CS | clinically significant |
| CSR | clinical study report |
| DBP | diastolic blood pressure |
| DEA | drug enforcement administration |
| DIA | drug information association |
| DOB | date of birth |



| Abbreviation | Definition |
|--------------|----------------------------------------------|
| EC | ethics committee |
| ECG | electrocardiogram |
| EMA | European medicines agency |
| EOS | End of study |
| ET | Early termination |
| FAS | Full analysis set |
| FDA | food and drug administration |
| FOCP | Females of childbearing potential |
| FPC | Follow-up phone call |
| HR | heart rate |
| IC or ICF | informed consent or informed consent form |
| ICH | international council for harmonization |
| ID | identification |
| IND | investigational new drug |
| IRB | institutional review board |
| LS | Least squares |
| MAR | Missing at random |
| MedDRA | medical dictionary for regulatory activities |
| mg | milligram |
| MI | Multiple imputation |
| MI | Metacognitive index |



| Abbreviation | Definition |
|--------------|------------------------------------------|
| MMRM | mixed effect model repeat measurement |
| MNAR | Missing not at random |
| ms | millisecond |
| N | number |
| NA | not applicable |
| NCS | non-clinically significant |
| OLE | Open-label extension |
| PD | protocol deviation |
| PE | physical examination |
| PK | pharmacokinetic |
| PKAP | pharmacokinetic analysis plan |
| POC | Point of care |
| PP | per-protocol |
| QD | Once daily |
| QOL | quality of life |
| REML | Restricted maximum likelihood |
| RR | respiratory rate or relative rate |
| SAE | serious adverse event |
| SAP | statistical analysis plan |
| SAS® | a software system used for data analysis |
| SBP | systolic blood pressure |





| Abbreviation | Definition |
|--------------|----------------------------------------------------|
| SD | standard deviation |
| SDQ | Symptoms of Depression Questionnaire |
| SF | screen failure |
| SM | Study medication |
| SOC | system organ class |
| SOP | standard operating procedure |
| TEAE | treatment-emergent adverse event |
| USA | United States of America |
| UTC | universal coordinated time |
| WHO | world health organization |
| WHO-DDE | world health organization drug dictionary enhanced |